

#### 1. RCT Details

This section provides a high-level overview of the RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 Title

CArdiovascular safety and Renal Microvascular outcomE study with LINAgliptin (CARMELINA trial)

#### 1.2 <u>Intended aim(s)</u>

The primary hypothesis was that treatment with linagliptin would be non-inferior with a hazard ratio of < 1.3 compared with placebo as assessed by the time to first occurrence of any of the 3P-MACE (primary endpoint) events.

### 1.3 Primary endpoint for replication and RCT finding

First occurrence of CV death, non-fatal myocardial infarction, or non-fatal stroke.

#### 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

Power- 0.90. Assuming a HR of 1.0, to demonstrate non-inferiority of linagliptin versus placebo within the pre-specified non-inferiority margin of 1.3 at a one-sided  $\alpha$ -level of 2.5%.

## 1.5 Primary trial estimate targeted for replication

HR = 1.02 (95% CI 0.89-1.17) comparing linagliptin to placebo (Rosenstock et al.)

#### 2. Person responsible for implementation of replication in Aetion

Ajinkya Pawar, Ph.D. implemented the study design in the Aetion Evidence Platform. S/he is not responsible for the validity of the design and analytic choices. All implementation steps are recorded and the implementation history is archived in the platform.

## 3. Data Source(s)

United/Optum, MarketScan, Medicare

### 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.

#### **Design Diagram – CARMELINA TRIAL REPLICATION**



#### 5. Cohort Identification

#### 5.1 Cohort Summary

This study will involve a new user, parallel group, cohort study design comparing linagliptin to the 2nd generation sulfonylurea (SU) antidiabetic class as a proxy for placebo. 2<sup>nd</sup> generation SUs are not known to have an impact on the outcome of interest. In addition, SUs were the most frequent background treatment in CARMELINA (after metformin), and DPP4i and SUs are preferentially prescribed to similarly older patients in real world (Patorno et al., 2019). The patients will be required to have continuous enrollment during the baseline period of 180 days before initiation of linagliptin or a comparator drug (cohort entry date). Follow-up for the outcome (3P-MACE), begins the day after drug initiation. As in the trial, patients are allowed to take other antidiabetic medications during study follow-up.

### 5.2 Important steps for cohort formation

#### 5.2.1 Eligible cohort entry dates

Market availability of linagliptin in the U.S. started on May 2, 2011.

- For Marketscan: May 2, 2011-Dec 31, 2017 (end of data availability).
- For Medicare: Jan 1, 2012-Dec 31, 2017 (start- end of data availability).
- For Optum: May 2, 2011-March 31, 2019 (end of data availability).

### 5.2.2 Specify <u>inclusion/exclusion</u> criteria for cohort entry and define the index date

Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

#### 5.3 Flowchart of the study cohort assembly

| Opt | um | Marke | etscan | Medi | care* |
|---|---|---|---|---|---|
| Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients |

| All patients in the database | | 74,864,884 | | 191,990,035 | | 23,466,175 |
|---|---|---|---|---|---|---|
| Patients who used exposure or a reference between <b>02 May 2011</b> to Dec 2017 (for Marketscan)/March 2019 (for Optum) and 01 January 2012-December 2017 for Medicare | -73,493,670 | 1,371,214 | -<br>190,287,730 | 1,702,305 | -19,944,169 | 3,522,006 |
| Patients who have continuous 6 months registration in the database | -185,581 | 1,185,633 | -171,524 | 1,530,781 | -972,275 | 2,549,731 |
| Patients without prior use of reference | -877,495 | 308,138 | -1,180,188 | 350,593 | -1,838,491 | 711,240 |
| Patients without prior use of exposure | -68,637 | 239,501 | -59,423 | 291,170 | -133,733 | 577,507 |
| Excluded because patient qualified in >1 exposure category | -275 | 239,226 | -211 | 290,959 | -370 | 577,137 |
| Patients who did not have missing age information | -12 | 239,214 | 0 | 290,959 | 0 | 577,137 |
| Patients who did not have missing gender information | -19 | 239,195 | 0 | 290,959 | 0 | 577,137 |
| Excluded based on Inclusion 1- DM Type 2 | -18,341 | 220,854 | -37,618 | 253,341 | -10,507 | 566,630 |
| Excluded based on Inclusion 5- Age >= 18 | -19 | 220,835 | -76 | 253,265 | 0 | 566,630 |
| Excluded based on Inclusion 6- Body Mass Index (BMI) =< 45 kg/m2 at visit 1 (as a proxy, excluding patients with morbid obesity) | -9,096 | 211,739 | -8,032 | 245,233 | -13,155 | 553,475 |
| Excluded based on Inclusion 8 - High risk of CV events | -64,122 | 147,617 | -98,434 | 146,799 | -67,114 | 486,361 |
| Excluded based on Exclusion 1- Type 1 DM with ICD10 CODES | -2,983 | 144,634 | -3,481 | 143,318 | -12,175 | 474,186 |
| Excluded based on Exclusion 2- Treatment (≥ 7 days) with GLP-1 RA, other DPP-4i or SGLT-2i | -7,712 | 136,922 | -9,388 | 133,930 | -23,347 | 450,839 |
| Excluded based on Exclusion 3- Liver disease | -2,648 | 134,274 | -1,931 | 131,999 | -8,953 | 441,886 |
| Excluded based on Exclusion 4- CKD Stage 5 (proxy for eGFR <15 ml/min/1.73 m2)/Dialysis | -707 | 133,567 | -470 | 131,529 | -3,368 | 438,518 |
| Excluded based on Exclusion 5- Any history of or planned bariatric surgery | 0 | 133,567 | 0 | 131,529 | 0 | 438,518 |
| Excluded based on Exclusion 6- Previous cardiac procedure (CABG or PTCA or Stent) $\leq$ 2 months | -436 | 133,131 | -569 | 130,960 | -1101 | 437,417 |
| Excluded based on Exclusion 8- Alcohol abuse/Drug abuse and Exclusion 10- Pregnancy | -1047 | 132,081 | -501 | 130,459 | -2,267 | 435,149 |
| Excluded based on Exclusion 11 part 1- life expectancy less than 5 years [using combined comorbidity index as a proxy (365 days) | -2,263 | 129,818 | -1,125 | 129,334 | -12,200 | 422,949 |
| Excluded based on Exclusion 11 part 2- History of Malignant Neoplasm (within last 3 years) | -4,153 | 125,665 | -4,128 | 125,206 | -14,241 | 408,708 |
| Excluded based on Exclusion 12- ACS/unstable angina ( $\leq 2$ months prior) | -374 | 125,291 | -332 | 124,874 | -788 | 407,920 |
| Excluded based on Exclusion 13- Stroke or TIA (≤ 3 months prior) | -2,292 | 122,999 | -1,981 | 122,893 | -7,081 | 400,839 |
| Final cohort | | 122,999 | | 122,893 | | 400,839 |

Effectiveness research with Real World Data to support FDA's regulatory decision making

- \* Medicare database includes only patients ≥65 years of age with at least one diagnosis for diabetes, heart failure, or stroke.
- \*\* Exclusion 8 and Exclusion 10 collapsed for adherence to CMS suppression guidelines.

#### 6. Variables

#### 6.1 Exposure-related variables:

#### Study drug:

The study exposure of interest is initiation of linagliptin. Initiation will be defined by no use of lingatliptin or a comparator in the prior 6 months before treatment initiation (washout period).

#### Comparator agents:

- Initiators of linagliptin will be compared to initiators of
  - o 2nd generation sulfonylureas

Because linagliptin and comparators are frequently used as second or third line treatments of T2DM, we expect it to be unlikely that linagliptin and comparators are initiated in patients with substantially different baseline risk for proposed outcomes.

### 6.2 Preliminary covariates:

- Age
- Sex
- Combined Comorbidity Index (CCI), measured over the baseline covariate assessment period, defined as 180 days prior to and including index date

Covariates listed above represent only a small subset of covariates that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (**Appendix B**). These covariates are based on those used by Patorno et al. (2019).

### 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Effectiveness outcomes of interest (definitions provided in **Appendix A**):

- <u>Primary outcome</u>: 3-point major adverse cardiovascular events (MACE), i.e., non-fatal myocardial infarction, non-fatal stroke, or CV mortality
- Secondary outcomes: Individual MACE components:
  - o Hospital admission for MI (for purposes of this individual component, fatal MI is included)
  - o Hospital admission for stroke (for purposes of this individual component, fatal stroke is included)
  - All-cause mortality/CV mortality:
    - All-cause inpatient mortality identified using discharge status codes will be used as a proxy for "CV mortality" in commercial databases
    - Information on CV mortality through data linkage with the National Death Index (NDI) will only become available at a later date for Medicare and will be used in secondary analyses.

Control outcomes of interest (control outcomes only serve to assess aspects of study validity but are not further interpreted):

1. End Stage Renal Disease (we expect to see no association; Rosenstock et al., 2019)

#### **Control outcome definitions**

| Outcome | Definition | Comments |
|---|---|---|
| Control Outcomes | | |
| End Stage Renal Disease<br>(ESRD) | ESRD with dialysis, defined as: An ICD9 diagnosis (inpatient or outpatient) for ESRD: o 585.5x, Chronic kidney disease, Stage V (for ESRD with no mention of dialysis) o 585.6x, End stage renal disease (for ESRD with dialysis) AND an ICD9 procedural codes for dialysis (=index date): o 39.95, Hemodialysis o 54.98, Peritoneal dialysis AND an additional procedural code for dialysis or physician provider code indicating dialysis procedure or ESRD-related activity within two time windows 31-60 and 61-90 days from index date. For patients who die prior to 61 days (31 days), the second (second and first) confirmation requirement(s) can be dropped. This ensures the inclusion of patients with true ESRD outcomes who die early (high early mortality) as well as early withdrawals from dialysis (which lead to high fatality within days or weeks). | Note- The corresponding ICD-10 codes will be used also |

Additional procedural codes for dialysis or physician provider codes indicating dialysis procedure or ESRD-related activity include:

- ICD9 procedural codes:
  - o 39.95, Hemodialysis
  - o 54.98, Peritoneal dialysis
- ICD9 diagnostic codes:
  - o 585.6x, End stage renal disease (for ESRD with dialysis)
  - o V56.0x, encounter for dialysis NOS
  - o V56.8x, encounter for peritoneal dialysis

#### - CPT4 codes:

- o 90957, 90960, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 4 or more face-to-face physician visits per month
- o 90958, 90961, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 2-3 face-to-face physician visits per month
- o 90959, 90962, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 1 face-to-face physician visit per month
- o 90920, 90921, ESRD related services per full month; for patients 12-19 and twenty years of age and over
- o 90924, 90925, ESRD related services (less than full month), per day; for patients 12-19 and twenty years of age and over
- o 90935, Hemodialysis procedure with single physician evaluation
- o 90937, Hemodialysis procedure requiring repeated evaluation(s) with or without substantial revision of dialysis prescription
- o 90945, Dialysis procedure other than hemodialysis (eg, peritoneal dialysis, hemofiltration, or other continuous renal replacement therapies), with single physician evaluation
- o 90947, Dialysis procedure other than hemodialysis (eg, peritoneal dialysis, hemofiltration, or other continuous renal replacement therapies) requiring repeated physician evaluations, with or without substantial revision of dialysis prescription
- o 90965, 90966, ESRD related services for home dialysis per full month, for patients 12-19 and 20 years of age and older
- o 90969, 90970, ESRD related services for dialysis less than a full month of service, per day; for patients 12-19 and 20 years of age and older
- o 90989, Dialysis training, patient, including helper where applicable, any mode, completed course
- o 90993, Dialysis training, patient, including helper where applicable, any mode, course not completed, per training session
- o 90999, Unlisted dialysis procedure, inpatient or outpatient
- o 99512, Home visit for hemodialysis

#### - HCPCS codes:

- o G0257, Unscheduled or emergency dialysis treatment for ESRD patient in a hospital outpatient dept. that is not certified as an ESRD facility
- o G0314, G0317, ESRD related services during the course of treatment, for patients 12-19 and 20 yrs of age an over to include monitoring for the adequacy of nutrition, etc. w/4 or more physician visit per month o G0315, G0318, ESRD related services during the course of treatment, for patients 12-19 and 20yrs of age and over to include monitoring for the adequacy of nutrition, etc. w/2 or 3 physician visit per month

- o G0316, G0319, ESRD related services during the course of treatment, for patients 12-19 and 20 yrs of age and over to include monitoring for the adequacy of nutrition, etc. w/1 physician visit per month
- o G0322, G0323, ESRD related services for home dialysis patients per full month: for patients 12-19 and 20 yrs of age and over to include monitoring for adequacy of nutrition and etc.
- o G0326, G0327, ESRD related services for home dialysis (less than full month), per day; for patients 12-19 and 20 yrs of age and over
- o S9335, Home therapy, hemodialysis; administrative services, professional pharmacy services, care coordination, and all necessary supplies and equipment (drugs and nursing services coded separately), per diem
- S9339, Home therapy, peritoneal dialysis, administrative services, care coordination and all necessary supplies and equipment, per diem

OR

Kidney transplant, defined as either 1 inpatient or 1 outpatient code Codes include:

- ICD9 prox codes:
  - o 55.6x, Transplant of kidney (Exclude 55.61)
- CPT4 codes:
  - o 50360, Renal allotransplantation, implantation, graft, w/o donor & recipient nephrectomy
- 50365, Renal allotransplantation, implantation, graft, w/ donor & recipient nephrectomy

### 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analyses will be conducted with treatment defined as the index drug on the day of cohort entry. Because adherence in the real world databases is expected to be much worse than in the trial, the AT analysis is the primary analysis, as it targets the relative hazard of outcomes on treatment.

For the AT analyses, the follow-up will start the day after initiation of linagliptin and comparator and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- Nursing home admission

- Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (linagliptin and comparator) plus a defined grace period (i.e., 30 days after the end of the last prescription's days' supply in main analyses).
- The date of augmentation or switching from an exposure to a comparator or any other agent in the comparator class and vice versa (e.g. switching from glimepiride to glipizide would be a censoring event);
  - o A dosage change on the index treatment does not fulfill this criterion
  - An added treatment that is not part of the exposure or comparator group does not fulfill this criterion (e.g. if a linagliptin user adds insulin, he or she does not get censored at the time of insulin augmentation)

For the ITT analyses, the censoring based on the augmentation/switching and treatment discontinuation will be replaced with a maximum allowed follow-up time of 365 days.

### 7. Initial Feasibility Analysis

#### Aetion report links:

Optum: https://bwh-dope.aetion.com/#/projects/details/702/results/30636/result/0
Marketscan: https://bwh-dope.aetion.com/#/projects/details/701/results/30634/result/0
Medicare: https://bwh-dope.aetion.com/#/projects/details/703/results/30635/result/0

Date conducted: rerun on January 28, 2019

Complete Aetion feasibility analysis using age, sex, and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed nor will incidence rates stratified by treatment group.

- Report patient characteristics by treatment group
- Report summary parameters of the overall study population
- Report median follow-up time by treatment group
- Report reasons for censoring in the overall study population

#### 8. Initial Power Assessment

#### Aetion report links:

Optum: https://bwh-dope.aetion.com/#/projects/details/702/results/30639/result/1

Marketscan: https://bwh-dope.aetion.com/#/projects/details/701/results/30637/result/1

Medicare: https://bwh-dope.aetion.com/#/projects/details/703/results/30638/result/1

Date conducted: rerun on January 28, 2019

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 3 covariates: age, sex, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

• Stop analyses until feasibility and power are reviewed by primary investigators and FDA. Reviewers evaluate the results of the analyses described above in Sections 7 and 8, including numbers of patients, patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power. These parameters are re-evaluated and reported in the subsequent sections, after incorporating feedback and refining the protocol.

| Reviewed by PI: | Jessica M. Franklin | Date reviewed: | 10/26/18 |
|-------------------------|---------------------|----------------|----------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 12/19/18 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

### 9. Balance Assessment after PS matching

## Aetion report name:

Optum: https://bwh-dope.aetion.com/projects/details/702/results/44872/result/0
Marketscan: https://bwh-dope.aetion.com/projects/details/701/results/44873/result/0
Medicare: https://bwh-dope.aetion.com/projects/details/703/results/45415/result/0

Date conducted: 11/18/2019 (Medicare 11/30/2019)

After review of initial feasibility and power analyses, complete creation of the remaining covariates (see Table 1 below for list of covariates). Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates (excluding laboratory values, which are missing in some patients).

• Provide plot of PS distributions stratified by treatment group.

Note- Please refer to **Appendix B**.

• Report covariate balance after matching.

Note- For Table 1, please refer to Appendix B.

• Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy Outcome | 0 (0.00%) | 0 (0.00%) | 0 (0.00%) |
| Death | 1,704 (1.67%) | 929 (1.82%) | 775 (1.52%) |
| Start of an additional exposure | 4,752 (4.67%) | 746 (1.47%) | 4,006 (7.87%) |
| End of index exposure | 58,792 (57.74%) | 29,602 (58.14%) | 29,190 (57.33%) |
| Specified date reached | 18,168 (17.84%) | 9,825 (19.30%) | 8,343 (16.39%) |
| End of patient enrollment | 9,190 (9.02%) | 4,583 (9.00%) | 4,607 (9.05%) |
| Switch to other SUs (for censoring) + nursing home admission | 9,224 (9.06%) | 5,230 (10.27%) | 3,994 (7.84%) |

• Report follow-up time by treatment group.

| | Median Follow-Up Time (Days) [IQR] | | |
|---|---|---|---|
| Patient Group | Optum | Marketscan | Medicare |
| Overall Patient Population | 118 [58-286] | 128 [63-304] | 137 [65-323] |
| Referent | 122 [65-304] | 148 [86-344] | 148 [86-344] |
| Exposure | 118 [58-269] | 127 [58-303] | 127 [58-303] |

• Report overall risk of the primary outcome.

| | Optum | Marketscan | Medicare |
|-------------------------|-------|------------|----------|
| Risk per 1,000 patients | 16.55 | 18.7 | 42.47 |

#### **10. Final Power Assessment**

Date conducted: 12/01/2019

• Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8. If the study is to be implemented in more than one database, copy and paste excel sheet to report power for each database separately and for the pooled analysis that uses data from all databases together. Power calculations are based on the formulas from Chow et al. (2008).

#### Pooled

| Non-inferiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | |
| Reference | 50,915 |
| Exposed | 50,915 |
| Risk per 1,000 patients | 25.91 |
| Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 |
| Non-inferiority margin | 1.3 |
| Number of events expected | 2638.4153 |
| Power | 0.999999116 |

#### o Optum

| 8,880 |
|-------------|
| 8,880 |
| 16.55 |
| 1 |
| 0.05 |
| 1.3 |
| 293.928 |
| 0.613734405 |

## Marketscan

| Non-inferiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | |
| Reference | 8,716 |
| Exposed | 8,716 |
| Risk per 1,000 patients | 18.7 |
| Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 |
| Non-inferiority margin | 1.3 |
| Number of events expected | 325.9784 |
| Power | 0.658551313 |

## o Medicare

Effectiveness research with Real World Data to support FDA's regulatory decision making: Protocol Template

| Non-inferiority Analysis | |
|----------------------------|------------|
| Number of patients matched | |
| Reference | 33,319 |
| Exposed | 33,319 |
| Risk per 1,000 patients | 42.47 |
| Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 |
| Non-inferiority margin | 1.3 |
| Number of events expected | 2830.11586 |
| Power | 0.9999974 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board. Reviewers evaluate the results of the analyses described above in Sections 9 and 10, including numbers of patients, balance in patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 12/9/19 |
|-------------------------|------------------|----------------|----------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 12/20/19 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

### 11. Study Confidence and Concerns

Deadline for voting on study confidence and listing concerns: 12/20/19

- If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.
- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the success of the RWD study in the <a href="Google Form">Google Form</a>. This form also provides space for reviewers to list any concerns that they feel may

contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the individual respondent.

### 12. Register study protocol on clinicalTrials.gov

#### Date conducted:

• Register the study on <u>clinicalTrials.gov</u> and upload this document.

### 13. Comparative Analyses

Aetion report name:

Date conducted:

#### 13.1 For **primary analysis**:

• In the PS-matched cohort from Section 9, calculate the HR for each outcome for linagliptin versus referent patients using a Cox proportional hazards model.

### 13.2 For secondary analyses:

• In the pre-matched cohort, perform asymmetrical trimming to remove patients with PS values below the 2.5<sup>th</sup> percentile of treated patients and above the 97.5<sup>th</sup> percentile of untreated patients. In the trimmed cohort, calculate the HR for canagliflozin versus referent patients using a Cox proportional hazards model, adjusting for deciles of the PS.

#### 14. Requested Results

### 14.1 Results from primary and secondary analyses:

Effectiveness research with Real World Data to support FDA's regulatory decision making: Protocol Template

Separately for each endpoint:

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Primary analysis | | | | | |
| Analysis 2 | | | | | |

HR, Hazard Ratio; CI, Confidence Interval.

#### 15. References

Chow S, Shao J, Wang H. 2008. Sample Size Calculations in Clinical Research. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. page 177

Patorno E, Pawar A, Franklin JM, et al. Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study. Circulation. 2019; in press. (https://www.ahajournals.org/doi/pdf/10.1161/CIRCULATIONAHA.118.039177)

Rosenstock J, Perkovic V, Johansen OE, Cooper ME, Kahn SE, Marx N, Alexander JH, Pencina M, Toto RD, Wanner C, Zinman B, Woerle HJ, Baanstra D, Pfarr E, Schnaidt S, Meinicke T, George JT, von Eynatten M, McGuire DK, CARMELINA Investigators. Effect of Linagliptin vs Placebo on Major Cardiovascular Events in Adults With Type 2 Diabetes and High Cardiovascular and Renal Risk: The CARMELINA Randomized Clinical Trial. *JAMA*. 2019; 321(1):69-79.

| # | CARMELINA trial definitions | Implementation in routine care | References/Rationale | Color coding |
|---|---|---|---|---|
| | 5a- Successful NI v | rith label change | Please see the following Google Drive for further details or any missing information:<br>https://drive.google.com/open?id=1WD618wrywYiEaXzfLTcuK-VCcnb6b-gV | Criteria |
| | EXPOSURE vs. ( | COMPARISON | ICD-10 codes are not listed in this document because of excel cell size limitations and excessive number of ICD-10 codes. Full ICD-10 code lists will be available in the above Google Drive Folder (link above). ICD-9 to ICD-10 code conversions were completed using a SAS macro that implements forward/backward mapping based on the CMS ICD-9 to ICD-10 mapping: <a href="https://www.nber.org/data/icd9-icd-10-cm-and-pcs-crosswalk-general-equivalence-mapping.html">https://www.nber.org/data/icd9-icd-10-cm-and-pcs-crosswalk-general-equivalence-mapping.html</a> | Adequate mapping in claims |
| | Linagliptin 5mg/day vs. placebo | linagliptin vs. 2nd generation sulfonylureas | | Intermediate mapping in claims |
| | PRIMARY C | DUTCOME | | Poor mapping or cannot be measured in claims |
| | The primary outcome is the time to the first occurrence of CV death, non-fatal myocardial infarction (MI) or non-fatal stroke—the so-called 3-point major adverse CV events (3P-MACE) composite outcome. | Measured 1 days after drug initiation in diagnosis position specified below and inpatient care setting: Inpatient mortality/MI/Stroke — For MI Any diagnosis position in inpatient care setting ICD-9 Dx 410.X (acute myocardial infarction) excluding 410.x2 (subsequent episode of care) For stroke Primary diagnosis position in inpatient care setting ICD-9 discharge diagnosis: 430.xx Subarachnoid hemorrhage (SAH) 431.xx Intracerebral hemorrhage (ICH) 433.x1 Dcclusion and stenosis of precerebral arteries with cerebral infarction 434.xx (excluding 434.x0) Occlusion and stenosis of cerebral arteries with cerebral infarction 436.x Acute, but ill-defined cerebrovascular events Mortality-See Mortality Sheet. | For MI: →PPV 94% in Medicare claims data [Kiyota Y, Schneeweiss S, Glynn RJ, Cannuscio CC, Avorn J, Solomon DH. Accuracy of Medicare claims-based diagnosis of acute myocardial infarction: estimating positive predictive value on the basis of review of hospital records. American heart journal 2004;148:99-104.] →PPV 88.4% in commercially-insured population [Wahl PM, Rodgers K, Schneeweiss S, et al. Validation of claims-based diagnostic and procedure codes for cardiovascular and gastrointestinal serious adverse events in a commercially-insured population. Pharmacoepidemiology and Drug Safety 2010;19:596-603.] For stroke: PPV of 85% or higher for ischemic stroke PPV ranging from 80% to 98% for hemorrhagic stroke PPV ranging from 80% to 98% for hemorrhagic stroke PPV ranging from 80% to 98% for hemorrhagic stroke identifying cerebrovascular accident or transient ischemic attack using administrative data. Pharmacoepidemiology and Drug Safety 2012;21 Suppl 1:100-28.] →[Tirschwell DL, Longstreth WT, Jr. Validating administrative data in stroke research. Stroke, a journal of cerebral circulation 2002;33:2465-70.] →[Roumie CL, Mitchel E, Gideon PS, Varas-Lorenzo C, Castellsague J, Griffin MR. Validation of ICD-9 codes with a high positive predictive value for incident strokes resulting in hospitalization using Medicaid health data. Pharmacoepidemiology and drug safety 2008;17:20-6.] | Can't be measured in claims but not important for the analysis |
| | INCLUSION | CRITERIA | | |
| | Documented diagnosis of T2DM before visit 1 (screening). | lem:Measured 180 days prior to drug initiation any diagnosis position in inpatient or outpatient care settings: Patients with a diagnosis of T2DM (ICD-9 Dx code of 250.x0 or 250.x2; ICD-10 Dx code of E11.x) in the 6 months prior to drug initiation | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA 118.039177 | |
| | <ol> <li>Male or female patients who are drug-naïve or pre-treated with any antidiabetic background<br/>therapy, excluding treatment with GLP-1 receptor agonists, DPP-4 inhibitors or SGLT-2 inhibitors if ≥<br/>7 consecutive days.</li> </ol> | This is basically everyone except for those with treatment with GLP-1 receptor agonists, DPP-4 inhibitors or SGLT-2 inhibitors if ≥7 consecutive days. One of the exclusion criteria below is exclusion based on ≥7 consecutive days use of GLP-1 receptor agonists, DPP-4 inhibitors or SGLT-2 inhibitors, so ignoring this inclusion criteria. | | |
| | 3) Ssheetle antidiabetic background medication (unchanged daily dose) for at least 8 weeks prior to randomization. If insulin is part of the background therapy, the average daily insulin dose should not have been changed by more than 10% within the 8 weeks prior to randomization compared with the daily insulin dose at randomization. 4) HbA1c of 26.5% and 510.0% at visit 1 (screening). | | - | |
| | 4) HbA1c ot≥6.5% and ≤10.0% at visit 1 (screening). 5) Age≥18 years at visit 1 (screening). For Japan only: Age ≥ 20 years at Visit 1. | N/A Measured 180 days prior to drug initiation Age ≥18 years | - | |

| | | Measured 180 days prior to drug initiation any diagnosis position in inpatient or outpatient care | |
|---|---|---|---|
| | | setting: Excluding patients with | |
| | | ICD-9 Diagnosis Code (any position) is any of: { "278.01" } | |
| - | Body Mass Index (BMI) £ 45 kg/m2 at visit 1 (screening). Signed and dated written informed consent by date of visit 1 (screening) in accordance with GCP. | 278.01 - MORBID OBESITY | |
| | and local legislation prior to any study related procedure. | N/A | - |
| | 8) High risk of CV events (I and/or II): | | |
| ' | Abbuminuria (UACR $\geq$ 30 mg/g creatinine or $\geq$ 30 µg/min [microgram albumin per minute] or $\geq$ 30 mg/24 h [milligram albumin per 24 hours] in two out of three unrelated spot urine or timed samples in the last 24 months prior to randomization)* | | |
| | AND previous macrovascular disease, defined as either one or more: | Manager of from the stand of all couldness data as a standard of discouldness of the standard | |
| <u></u> | Confirmed history of MI (> 2 months prior to Visit 1) | Measured from the start of all available data to on the date of drug initiation with diagnosis/procedure position and care setting as noted below: | |
| la | Confirmed history of Mil (> 2 months prior to visit 1) | leshamis ha ant disagra in any diagnasis nacities and investigat ay outputiont care setting ICD 0 | |
| | Advanced coronary artery disease, defined by any one of the following: | Ischemic heart disease in any diagnosis position and inpatient or outpatient care setting: ICD-9 410.xx-414.xx | |
| | <ul> <li>≥50% narrowing of the luminal diameter in 2 or more major coronary arteries by coronary<br/>angiography, MRI angiography or CT angiography;</li> </ul> | OR | |
| | Definition of major coronary arteries: LAD (Left Anterior Descending). CX (Circumflex) or RCA (right coronary artery) | | |
| lb | Left main stem coronary artery with ≥50% narrowing of the luminal diameter by coronary | Previous cardiac procedure (CABG or PTCA or Stent) in any procedure position and care setting defined below: | |
| " | angiography, MRI angiography or CT angiography; • Prior percutaneous or surgical revascularization of ≥ 2 major coronary arteries at least 2 months | PTCA: | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus |
| | prior to Visit 1 (screening); | Inpatient CPT-4: 92973, 92982, 92984, 92995, 92996, 92920 – 92921, 92924 – 92925, 92937, 92938, 92941, 92943, 92944 | other non-gliflozin antidiabetic drugs: population based cohort study." BMJ |
| | <ul> <li>The combination of prior percutaneous or surgical revascularization of 1 major coronary artery at<br/>least 2 months prior to visit 1 (screening), and ≥ 50% narrowing of the luminal diameter by coronary</li> </ul> | OR – | 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 |
| | angiography, MRI angiography or CT angiography of at least 1 additional major coronary artery. | Inpatient or outpatient ICD-9 procedure: 00.66, 36.01, 36.02, 36.03, 36.05, 36.09 | Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness |
| $\vdash$ | | Stenting:<br>Inpatient CPT-4: 92980, 92981, 92928 – 92929, 92933 - 92934 | and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: |
| | High-risk single-vessel coronary artery disease, defined as the presence of≥50% | OR – | 10.1161/CIRCULATIONAHA.118.039177 |
| | narrowing of the luminal diameter of one major coronary artery by coronary angiography, MRI | Inpatient or outpatient ICD-9 procedure: 36.06, 36.07 | |
| | angiography or CT angiography in patients not revascularized: AND at least one of the following: | CABG: | |
| | A positive non invasive stress test, confirmed by either: | Inpatient CPT-4: 33510 – 33536, 33545, 33572. OR – | |
| Ic | o a positive ECG exercise tolerance test in patients without left bundle branch block, Wolff-Parkinson White syndrome, left ventricular hypertrophy with repolarization abnormality, or paced ventricular | Inpatient or outpatient ICD-9 procedure: 36.1x, 36.2x | |
| | rhythm, atrial fibrillation in case of abnormal ST-T segments; o a positive stress echocardiogram showing induced regional systolic wall motion abnormalities; | Transmyocardial revascularization: Inpatient or Outpatient CPT-4: 33140, 33141 OR - Inpatient or | |
| | o a positive stress echocardiogram showing induced regional systolic wall motion abnormalities;<br>o a positive nuclear myocardial perfusion imaging stress test showing stress-induced reversible | outpatient ICD-9 procedure: 36.31-36.34 | |
| | perfusion abnormality; o a positive cardiac stress perfusion MRI showing a stress induced perfusion defect; | | |
| | <ul> <li>Patient discharged from hospital with a documented diagnosis of unstable angina pectoris between</li> </ul> | | |
| | 2 and 12 months prior to visit 1 (screening). | | |
| | | | We including anytime prior to drug initiation here, but then any patients with any |
| Id | | Measured from the start of all available data to on the date of drug initiation in any diagnosis position and procedure position in inpatient or outpatient care setting: | stroke within last 3 months are excluded due to the last exclusion criteria. |
| 1 | History of lash and a substitute of 2 and the substitute of 3 | Any stroke ICD-9 Dx: 430.xx, 431.xx, 433.xx, 434.xx, 436.xx | |
| | History of ischemic or haemorrhagic stroke (>3 months prior to visit 1) | | |
| | | | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus |
| | | Measured from the start of all available data to on the date of drug initiation in any diagnosis | other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 |
| le | | position and procedure position in inpatient or outpatient care setting: | |
| " | Presence of carotid artery disease (symptomatic or not) documented by either: o imaging techniques with at least one lesion estimated to be ≥50% | Carotid artery disease ICD-9 433.10: Occlusion and stenosis of carotid artery without mention of cerebral infarction. | Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness |
| | narrowing of the luminal diameter; | ICD-10-CM I65.29 Occlusion and stenosis of unspecified carotid artery | and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: |
| | o prior percutaneous or surgical carotid revascularization. | | 10.1161/CIRCULATIONAHA.118.039177 |

| _ | | | |
|---|---|---|---|
| | Presence of peripheral artery disease documented by either: o previous limb angioplasty, stenting or bypass surgery; o previous limb or foot amputation due to macrocirculatory insufficiency; o angiographic evidence of peripheral artery stenosis 250% narrowing of the luminal diameter in at least one limb (definition of peripheral artery; senosis 250% narrowing and the luminal diameter in at least one limb (definition of peripheral artery; common iliac artery, internal iliac artery, external iliac artery, femoral artery, popliteal artery). | Measured from the start of all available data to on the date of drug initiation in any diagnosis position and procedure position in inpatient or outpatient care setting Carotid bypass: ICD9 procedure: 39.28 ICD10 procedure: 39.28 | |
| 11. | Evidence of impaired renal function with predefined UACR, with or without CV co-morbidities, defined as follows (and/or criteria): - Impaired renal function (as defined by MDRD formula) with an eGFR: 15-<45 mL/min/1.73 m2 at visit 1 (screening) with any UACR. - Impaired renal function (as defined by MDRD formula) with an eGFR ≥ 45-75 mL/min/1.73 m2 at visit 1 (screening) with an UACR > 200 mg/g creatinine or | Measured 180 days prior to drug initiation in any diagnosis position in inpatient or outpatient filters: CKD stage 3 and stage 4 585.3x-585.4x | CKD stage 1: GFR >90 CKD stage 2: GFR 60 to 89 CKD stage 3a: GFR 45 to 59 CKD stage 3b: GFR 30 to 44 CKD stage 4: GFR 15 to 29 CKD stage 5: GFR <15 |
| | > 200 µg/min (microgram albumin per minute) or > 200 mg/24 h [milligram albumin per 24 hours] demonstrated in two out of three unrelated spot urine or timed samples in the last 24 months prior to randomization. EXCLUSION | N/A CRITERIA | · |
| _ | EXCLUSION | | |
| | 1) Type 1 diabetes mellitus. | Measured 180 days prior to drug initiation in any diagnosis position in inpatient or outpatient care setting: $DM \text{ type } 1-At \text{least 1 inpatient or outpatient ICD-9 Dx code of 250.x1 or 250.x3 or ICD-10 Dx code of E10.x in the 12 months prior to drug initiation. 6-months prior D = \frac{1}{2} \frac{1}$ | |
| | 2) Treatment (≥ 7 consecutive days) with GLP-1 receptor agonists, other DPP-4 inhibitors or SGLT-2 inhibitors prior to informed consent. Note: This also includes clinical trials where these antidiabetic drugs have been provided to the patient. | Measured 180 days prior to drug initiation as a dispensing for one of the following: Treatment (≥7 days) with GLP-1 receptor agonists (lixisenatide, dulaglutide, albiglutide, liraglutide, exenatide), other DPP-4 inhibitors (alogliptin, sitagliptin, saxagliptin) or SGLT-2 inhibitors (canagliflozin, dapagliflozin, empagliflozin) prior to CED | |
| | <ol> <li>Active liver disease or impaired hepatic function, defined by serum levels of either ALT (SGPT), AST<br/>(SGOT), or alkaline phosphatase (AP)≥3 x upper limit of normal (ULN) as determined at Visit 1.</li> </ol> | Measured 180 days prior to drug initiation in any diagnosis/procedure position in inpatient or outpatient care setting: Liver disease-ICD-9 diagnosis: 070.xx, 570.xx-573.xx 456.0x-456.2x, 576.8x, 782.4x, 789.5x ICD-9 procedure codes: 39.1x, 42.91 | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety [EMPRISE] Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
| | GFFR <15 ml/min/1.73 m2 (severe renal impairment or ESRD, MDRD formula), as determined during screening at Visit 1 and/or the need for maintenance dialysis. | Measured 180 days prior to drug initiation: CKD stage 5 in any diagnosis/procedure position in inpatient or outpatient care setting-585.5x OR Dialysis in any diagnosis/procedure position and inpatient care setting: Codes are in the sheet 'Dialysis' Sheet | |

| 5) Any previous (or planned within next 12 months) bariatric surgery (open or laparoscopic) or intervention (gastric sleeve). | Measured 180 days prior to drug initiation in any procedure position in inpatient or outpatient care setting: Any history CPT-Code-Abbreviation Procedure 43644 -LRYBG -Laparoscopic Roux-en-Ygastric bypass (Roux limb 150 cm or less) 43645 -LRYGBX- Laparoscopic gastric bypass with small intestine reconstruction to limit absorption 43770 -LAGB- Laparoscopic adjustable gastric band 43846 -ORYGB- Open Roux-en-Ygastric bypass (Roux limb 150 cm or less) 43847 -ORYGBX- Open gastric bypass with small intestine reconstruction to limit absorption | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
|---|---|---|
| 6) Pre-planned coronary artery re-vascularization (PCI, CABG) or any previous PCI and/or CABG ≤ 2 months prior informed consent | Measured 60 days prior to drug initiation in any diagnosis position and procedure position in care settings indicated below: (\$2 months) PTCA: Inpatient CPT-4: 92973, 92982, 92984, 92995, 92996, 92920 –92921, 92924 –92925, 92937, 92938, 92941, 92943, 92944 OR – Inpatient or outpatient: ICD-9 procedure: 00.66, 36.01, 36.02, 36.03, 36.05, 36.09 Stenting: Inpatient CPT-4: 92980, 92981, 92928 –92929, 92933 -92934 OR – Inpatient or outpatient ICD-9 procedure: 36.06, 36.07 CABG: Inpatient CPT-4: 33510 – 33536, 33545, 33572. OR – Inpatient or outpatient ICD-9 procedure: 36.1x, 36.2x | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
| 7) Known hypersensitivity or allergy to the investigational products or its excipients. | N/A | - |
| <ol> <li>Any previous or current alcohol or drug abuse that would interfere with trial participation in the<br/>opinion of the investigator.</li> </ol> | Measured 180 days prior to drug initiation in any diagnosis position in inpatient or outpatient care setting: Alcohol abuse or dependence 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x Drug abuse or dependence 292.xx, 304.xx, 305.2x-305.9x, 648.3x | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gilflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
| 9) Participation in another trial with an investigational drug ongoing or within 2 months prior to visit 1 (screening)*. | N/A | - |
| 9) Participation in another trial with an investigational drug ongoing or within 2 months prior to visit 1 (screening)*. | Measured 180 days prior to drug initiation in any diagnosis/procedure position in inpatient or outpatient care setting: Please see Pregnancy codes sheet. | |
| 11) Patients considered unreliable by the investigator concerning the requirements for follow-up during the study and/or compliance with study drug administration, have a life expectancy less than 5 years for non-CV causes, or have cancer other than non-melanoma skin cancer within last 3 years, or has any other condition than mentioned which in the opinion of the investigator, would not allow safe participation in the study. | Measured over 365 days prior to drug initiation: CCl >= 10 OR Measured 1095 days prior to drug initiation in any diagnosis position in inpatient and outpatient care setting: History of malignant neoplasm ICD-9: 140.xx-208.xx (except 173.xx, non-melanoma skin cancer)-in prior 3 years | "Gagne, Josh J et. al. ""A combined comorbidity score predicted mortality in elderly patients better than existing scores."" J Clin Epidemiol. 2011 Jul;64(7):749-59. doi: 10.1016/j.jclinepi.2010.10.004. Sun, Jenny W et. al. ""Validation of the Combined Comorbidity Index of Charlson and Elixhauser to Predict 30-Day Mortality Across ICD-9 and ICD-10."" Med Care. 2018 Sep;56(9):812. doi: 10.1097/MLR.000000000000954." |
| 12) Acute coronary syndrome (ACS), diagnosed ≤ 2 months prior to visit 1 (screening). | Measured 60 days prior to drug initiation in any diagnosis position in inpatient and outpatient care setting: ACS/unstable angina 411.xx | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |

| 13) Stroke or ∏A≤3 mo | Measured 90 days prior to drug initiation in any diagnosis position in inpatient and outpatient care setting: Any stroke ICD-9 Dx: 430.xx, 431.xx, 433.xx, 434.xx, 436.xx TIA 435. yx | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
|---|---|---|
|---|---|---|

| Trial ID | |
|---|---|
| Trial Name (with web links) | CARMELINA |
| <u>NCT</u> | NCT01897532 |
| <u>Trial category</u> | 5a- Successful NI with label change |
| Therapeutic Area | Endocrinology |
| RCT Category | Secondary indication |
| <b>Brand Name</b> | |
| <b>Generic Name</b> | Linagliptin |
| Sponsor | Boehringer Ingelheim |
| <u>Year</u> | 2019 |
| Measurable endpoint | Composite of Cardiovascular Death, Non-fatal Myocardial Infarction, or Non-fatal Stroke |
| <u>Exposure</u> | Linagliptin |
| <u>Comparator</u> | Placebo |
| <u>Population</u> | |
| Trial finding | 1.02 (95% CI 0.89-1.17) |
| No. of Patients | 6979 |
| Non-inferiority margin | 1.3 |
| Assay Sens. Endpoint | |
| Assay Sens. Finding | |
| <u>Power</u> | Power- 0.90. Assuming a HR of 1.0, to demonstrate non-inferiority of linagliptin versus placebo within the pre-specified non-inferiority margin of 1.3 at a one-sided $\alpha$ -level of 2.5%. |
| Blinding | |
| Statistical Method | |

### Mortality-Dependent on data source.

1. All-cause mortality / inpatient mortality Identified using the vital status file-

#### Medicare

Identified using the discharge status codes-

#### Optum-

- 20 = EXPIRED
- 21 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 22 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 23 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 24 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 25 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 26 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 27 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 28 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 29 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 40 = EXPIRED AT HOME (HOSPICE)
- 41 = EXPIRED IN A MEDICAL FACILITY (HOSPICE)
- 42 = EXPIRED PLACE UNKNOWN (HOSPICE)

#### Truven-

- 20 Died
- 22 Died
- 23 Died
- 24 Died
- 25 Died
- 26 Died
- 27 Died
- 28 Died
- 29 Died
- 40 Other died status or Expired at home (Hospice claims only) (depends on year)
- 41 Other died status or Expired in medical facility (Hospice claims only) (depends on year)

- 42 Other died status or Expired place unknown (Hospice claims only) (depends on year)
- 21 Died or Disch./Transf. to court/law enforcement (depends on year)

### 2. CV mortality

Information on CV mortality through data linkage with the National Death Index (NDI) will be available for Medicare at a later date. We will conduct secondary analyses using CV mortality at that time.

| Antidiabetic class | Specific agent | Notes |
|---|---|---|
| | Canagliflozin | Approved 3/29/2013 |
| SGLT2-inhibitors | Dapagliflozin | |
| SGL 12-inhibitors | Empagliflozin | |
| | Ertugliflozin | Approved Dec 21, 2017 |
| | Glimepiride | |
| 2 <sup>nd</sup> generation sulfonylureas | Glipizide | |
| | Glyburide | |
| | Alogliptin | |
| DPP-4 inhibitors | Linagliptin | |
| DPP-4 Innibitors | Saxagliptin | |
| | Sitagliptin | |
| | Exenatide | |
| | Liraglutide | |
| GLP-1 receptor agonist (GLP1-RA) | Albiglutide | Approved April 15, 2014 and discontinued July 26, 2017 |
| | Dulaglutide | Approved Sep 18, 2014 |
| | Lixisenatide | Approved July 28, 2016 |
| | Semaglutide | Approved Dec 5, 2017 |
| | Insulin Aspart | |
| | Insulin Aspart/Insulin Aspart | |
| | Protamine | |
| | Insulin Degludec | |
| | Insulin Detemir | |
| | Insulin Glargine | |
| | Insulin Glulisine | |
| Insulin | Insulin human isophane (NPH) | |
| | Insulin human regular (search with NPH, don't want bf-pk) | |
| | Insulin human regular/ Insulin human isophane (NPH) | |
| | Insulin Lispro | |

| | Insulin Lispro/Insulin Lispro<br>Protamine |
|---|---|
| Clitaranas | Pioglitazone |
| Glitazones | Rosiglitazone |
| Maglitinidas | Nateglinide |
| Meglitinides | Repaglinide |
| A1.1 1 11 1 | Acarbose |
| Alpha-glucosidase inhibitors | Miglitol |
| Pramlintide | Pramlintide |
| | Acetohexamide |
| 1 <sup>st</sup> generation sulfonylureas | Chlorpropamide |
| | Tolazamide |
| | Tolbutamide |

## Pregnancy Dx codes 650 NORMAL DELIVERY 660 OBSTRUCTED LABOR 661 ABNORMALITY OF FORCES OF LABOR 662 LONG LABOR 663 UMBILICAL CORD COMPLICATIONS DURING LABOR AND DELIVERY 664 TRAUMA TO PERINEUM AND VULVA DURING DELIVERY 665 OTHER OBSTETRICAL TRAUMA 667 RETAINED PLACENTA OR MEMBRANES WITHOUT HEMORRHAGE 668 COMPLICATIONS OF THE ADMINISTRATION OF ANESTHETIC OR OTHER SEDATION IN LABOR AND **DELIVERY** 669.94 UNSPECIFIED COMPLICATION OF LABOR AND DELIVERY POSTPARTUM CONDITION OR COMPLICATION V24 POSTPARTUM CARE AND EXAMINATION V24.0 POSTPARTUM CARE AND EXAMINATION IMMEDIATELY AFTER DELIVERY V24.1 POSTPARTUM CARE AND EXAMINATION OF LACTATING MOTHER V24.2 ROUTINE POSTPARTUM FOLLOW V27 OUTCOME OF DELIVERY V27.0 MOTHER WITH SINGLE LIVEBORN V27.1 MOTHER WITH SINGLE STILLBORN V27.2 MOTHER WITH TWINS BOTH LIVEBORN V27.3 MOTHER WITH TWINS ONE LIVEBORN AND ONE STILLBORN V27.4 MOTHER WITH TWINS BOTH STILLBORN V27.5 MOTHER WITH OTHER MULTIPLE BIRTH ALL LIVEBORN V27.6 MOTHER WITH OTHER MULTIPLE BIRTH SOME LIVEBORN V27.7 MOTHER WITH OTHER MULTIPLE BIRTH ALL STILLBORN V27.9 MOTHER WITH UNSPECIFIED OUTCOME OF DELIVERY **Procedure codes** 72.0 LOW FORCEPS OPERATION 72.1 LOW FORCEPS OPERATION WITH EPISIOTOMY 72.2 MID FORCEPS OPERATION 72.21 MID FORCEPS OPERATION WITH EPISIOTOMY 72.29 OTHER MID FORCEPS OPERATION 72.3 HIGH FORCEPS OPERATION

| 72.31 HIGH FORCEPS OPERATION WITH EPISIOTOMY |
|------------------------------------------------------------------|
| 72.39 OTHER HIGH FORCEPS OPERATION |
| 72.4 FORCEPS ROTATION OF FETAL HEAD |
| 72.5 BREECH EXTRACTION |
| 72.51 PARTIAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD |
| 72.52 OTHER PARTIAL BREECH EXTRACTION |
| 72.53 TOTAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD |
| 72.54 OTHER TOTAL BREECH EXTRACTION |
| 72.6 FORCEPS APPLICATION TO AFTERCOMING HEAD |
| 72.7 VACUUM EXTRACTION |
| 72.71 VACUUM EXTRACTION WITH EPISIOTOMY |
| 72.79 OTHER VACUUM EXTRACTION |
| 72.8 OTHER SPECIFIED INSTRUMENTAL DELIVERY |
| 72.9 UNSPECIFIED INSTRUMENTAL DELIVERY |
| 73.0 ARTIFICIAL RUPTURE OF MEMBRANES |
| 73.01 INDUCTION OF LABOR BY ARTIFICIAL RUPTURE OF MEMBRANES |
| 73.09 OTHER ARTIFICIAL RUPTURE OF MEMBRANES |
| 73.1 OTHER SURGICAL INDUCTION OF LABOR |
| 73.2 INTERNAL AND COMBINED VERSION AND EXTRACTION |
| 73.21 INTERNAL AND COMBINED VERSION WITHOUT EXTRACTION |
| 73.22 INTERNAL AND COMBINED VERSION WITH EXTRACTION |
| 73.3 FAILED FORCEPS |
| 73.4 MEDICAL INDUCTION OF LABOR |
| 73.5 MANUALLY ASSISTED DELIVERY |
| 73.51 MANUAL ROTATION OF FETAL HEAD |
| 73.59 OTHER MANUALLY ASSISTED DELIVERY |
| 73.6 EPISIOTOMY |
| 73.8 OPERATIONS ON FETUS TO FACILITATE DELIVERY |
| 73.9 OTHER OPERATIONS ASSISTING DELIVERY |
| 73.91 EXTERNAL VERSION ASSISTING DELIVERY |
| 73.92 REPLACEMENT OF PROLAPSED UMBILICAL CORD |
| 73.93 INCISION OF CERVIX TO ASSIST DELIVERY |
| 73.94 PUBIOTOMY TO ASSIST DELIVERY |
| 73.99 OTHER OPERATIONS ASSISTING DELIVERY |

74.0 CLASSICAL CESAREAN SECTION

| 74 1 | I OW CFRVICAL | CESAREAN | SECTION |
|------|---------------|----------|---------|

- 74.2 EXTRAPERITONEAL CESAREAN SECTION
- 74.3 REMOVAL OF EXTRATUBAL ECTOPIC PREGNANCY
- 74.4 CESAREAN SECTION OF OTHER SPECIFIED TYPE
- 74.9 CESAREAN SECTION OF UNSPECIFIED TYPE
- 74.91 HYSTEROTOMY TO TERMINATE PREGNANCY
- 74.99 OTHER CESAREAN SECTION OF UNSPECIFIED TYPE
- 75.4 MANUAL REMOVAL OF RETAINED PLACENTA
- 75.5 REPAIR OF CURRENT OBSTETRIC LACERATION OF UTERUS
- 75.6 REPAIR OF OTHER CURRENT OBSTETRIC LACERATION
- 75.7 MANUAL EXPLORATION OF UTERINE CAVITY, POSTPARTUM
- 75.9 OTHER OBSTETRIC OPERATIONS

#### **Dialysis**

Dialysis

Codes include:

- ICD9 prox codes:

39.95, Hemodialysis

54.98, Peritoneal dialysis

- ICD9 dx codes:

V56.0x, encounter for dialysis NOS

V56.8x, encounter for peritoneal dialysis

V45.1x, renal dialysis status

- CPT4 codes:

90957, 90960, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 4 or more face-to-face physician visits per month

90958, 90961, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 2-3 face-to-face physician visits per month

90959, 90962, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 1 face-to-face physician visit per month

90920, 90921, ESRD related services per full month; for patients 12-19 and twenty years of age and over

90924, 90925, ESRD related services (less than full month), per day; for patients 12-19 and twenty years of age and over

90935, Hemodialysis procedure with single physician evaluation

90937, Hemodialysis procedure requiring repeated evaluation(s) with or without substantial revision of dialysis prescription 90945, Dialysis procedure other than hemodialysis (eg, peritoneal dialysis, hemofiltration, or other continuous renal replacement therapies), with single physician evaluation

90947, Dialysis procedure other than hemodialysis (eg, peritoneal dialysis, hemofiltration, or other continuous renal replacement

therapies) requiring repeated physician evaluations, with or without substantial revision of dialysis prescription

90965, 90966, ESRD related services for home dialysis per full month, for patients 12-19 and 20 years of age and older

90969, 90970, ESRD related services for dialysis less than a full month of service, per day; for patients 12-19 and 20 years of age and older

90989, Dialysis training, patient, including helper where applicable, any mode, completed course

90993, Dialysis training, patient, including helper where applicable, any mode, course not completed, per training session

90999, Unlisted dialysis procedure, inpatient or outpatient

99512, Home visit for hemodialysis

- HCPCS codes:

G0257, Unscheduled or emergency dialysis treatment for ESRD patient in a hospital outpatient dept. that is not certified as an ESRD facility

G0314, G0317, ESRD related services during the course of treatment, for patients 12-19 and 20 yrs of age an over to include monitoring for the adequacy of nutrition, etc. w/4 or more physician visit per month

G0315, G0318, ESRD related services during the course of treatment, for patients 12-19 and 20yrs of age and over to include monitoring for the adequacy of nutrition, etc. w/2 or 3 physician visit per month

G0316, G0319, ESRD related services during the course of treatment, for patients 12-19 and 20 yrs of age and over to include

monitoring for the adequacy of nutrition, etc. w/1 physician visit per month

G0322, G0323, ESRD related services for home dialysis patients per full month: for patients 12-19 and 20 yrs of age and over to include monitoring for adequacy of nutrition and etc.

G0326, G0327, ESRD related services for home dialysis (less than full month), per day; for patients 12-19 and 20 yrs of age and over

S9335, Home therapy, hemodialysis; administrative services, professional pharmacy services, care coordination, and all necessary supplies and equipment (drugs and nursing services coded separately), per diem

S9339, Home therapy, peritoneal dialysis, administrative services, care coordination and all necessary supplies and equipment, per diem

# Appendix B



| | Unmatched | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Optu | m I | Markets | Scan | Medicare | | | POOLED | |
| | Reference-2nd | | Reference-2nd | | Reference-2nd | Exposure- | Reference-2nd | | |
| Variable | Generation SUs | Exposure-Linagliptin | Generation SUs | Exposure-Linagliptin | Generation SUs | Linagliptin | Generation SUs | Exposure-Linagliptin | St. Diff. |
| Number of patients | 113,991 | 8,904 | 114,025 | 8,736 | 366,136 | 33,401 | 594,152 | 51,041 | |
| Age | 50.55 (40.30) | CC 04 (44 C4) | CE 25 (44 07) | 62.75 (44.52) | 75 67 (7.25) | 75 07 (7 44) | 72.54(0.00) | 72 20 (0 00) | 0.00 |
| mean (sd) | 69.66 (10.39) | 66.94 (11.64) | 65.35 (11.87) | 63.75 (11.53) | 75.67 (7.35) | 75.97 (7.44) | 72.54 (9.00) | 72.30 (9.09) | 0.03 |
| median [IQR] | 70.00 [64.00, 77.00] | 67.00 [59.00, 76.00] | 64.00 [57.00, 74.00] | 62.00 [56.00, 71.00] | 75.00 [70.00, 81.00] 5 | .00 [70.00, 81.00] | 71.93 (9.00) | 71.38 (9.09) | 0.06 |
| Age categories | | | | | | - //1 | | | |
| 18 - 54; n (%) | 10,233 (9.0%) | 1,320 (14.8%) | 19,802 (17.4%) | 1,718 (19.7%) | 0 (0.0%) | 0 (0.0%) | 30,035 (5.1%) | 3,038 (6.0%) | -0.04<br>-0.04 |
| 55 - 64; n (%) | 20,561 (18.0%) | 2,441 (27.4%) | 40,305 (35.3%)<br>26,643 (23.4%) | 3,535 (40.5%) | 4,429 (1.2%) | 340 (1.0%)<br>15,653 (46.9%) | 65,295 (11.0%)<br>248,754 (41.9%) | 6,316 (12.4%) | 0.04 |
| 65 - 74; n (%)<br>>= 75; n (%) | 44,396 (38.9%)<br>38,801 (34.0%) | 2,639 (29.6%)<br>2,504 (28.1%) | 27,275 (23.9%) | 1,785 (20.4%)<br>1,698 (19.4%) | 177,715 (48.5%)<br>183,992 (50.3%) | 17,408 (52.1%) | 250,068 (42.1%) | 20,077 (39.3%)<br>21,610 (42.3%) | 0.00 |
| Gender | 38,801 (34.0%) | 2,304 (28.176) | 27,273 (23.376) | 1,038 (13.478) | 183,552 (30.376) | 17,408 (32.176) | 250,008 (42.178) | 21,010 (42.370) | 0.00 |
| Males; n (%) | 63,640 (55.8%) | 4,680 (52.6%) | 68,352 (59.9%) | 5,051 (57.8%) | 175,512 (47.9%) | 14,152 (42.4%) | 307,504 (51.8%) | 23,883 (46.8%) | 0.10 |
| Females; n (%) | 50,351 (44.2%) | 4,224 (47.4%) | 45,673 (40.1%) | 3,685 (42.2%) | 190,624 (52.1%) | 19,249 (57.6%) | 286,648 (48.2%) | 27,158 (53.2%) | -0.10 |
| Race | | , , , , | -,, -, | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | , , | ., . ( , | , , | , ( , | |
| White; n (%) | N/A | N/A | N/A | N/A | 288,259 (78.7%) | 23,448 (70.2%) | 288,259 (78.7%) | 23,448 (70.2%) | 0.20 |
| Black; n (%) | N/A | N/A | N/A | N/A | 40,279 (11.0%) | 4,263 (12.8%) | 40,279 (11.0%) | 4,263 (12.8%) | -0.06 |
| Asian; n (%) | N/A | N/A | N/A | N/A | 11,760 (3.2%) | 2,180 (6.5%) | 11,760 (3.2%) | 2,180 (6.5%) | -0.15 |
| Hispanic; n (%) | N/A | N/A | N/A | N/A | 13,446 (3.7%) | 1,876 (5.6%) | 13,446 (3.7%) | 1,876 (5.6%) | -0.09 |
| North American Native; n (%) | N/A | N/A | N/A | N/A | 2,376 (0.6%) | 270 (0.8%) | 2,376 (0.6%) | 270 (0.8%) | -0.02 |
| Other/Unknown; n (%) | N/A | N/A | N/A | N/A | 10,016 (2.7%) | 1,364 (4.1%) | 10,016 (2.7%) | 1,364 (4.1%) | -0.08 |
| Region (lumping missing&other category with West) | | | | | | | | | |
| Northeast; n (%) | 11,593 (10.2%) | 1,146 (12.9%) | 18,556 (16.3%) | 1,945 (22.3%) | 59,526 (16.3%) | 6,826 (20.4%) | 89,675 (15.1%) | 9,917 (19.4%) | -0.11 |
| South; n (%) | 54,025 (47.4%) | 4,626 (52.0%) | 33,925 (29.8%) | 1,644 (18.8%) | 159,156 (43.5%) | 14,335 (42.9%) | 247,106 (41.6%) | 20,605 (40.4%) | 0.02 |
| Midwest; n (%) | 22,555 (19.8%) | 1,593 (17.9%) | 45,492 (39.9%) | 4,155 (47.6%) | 89,214 (24.4%) | 5,801 (17.4%) | 157,261 (26.5%) | 11,549 (22.6%) | 0.09 |
| West; n (%) | 25,818 (22.6%) | 1,539 (17.3%) | 15,054 (13.2%) | 897 (10.3%) | 58,240 (15.9%) | 6,439 (19.3%) | 99,112 (16.7%) | 8,875 (17.4%) | -0.02 |
| Unknown+missing; n (%) | N/A | N/A | 998 (0.9%) | 95 (1.1%) | N/A | N/A | 998 (0.9%) | 95 (1.1%) | -0.02 |
| CV Covariates | | | | | | | | | |
| Ischemic heart disease; n (%) | 45,790 (40.2%) | 3,476 (39.0%) | 41,586 (36.5%) | 3,037 (34.8%) | 159,800 (43.6%) | 13,793 (41.3%) | 247,176 (41.6%) | 20,306 (39.8%) | 0.04 |
| Acute MI; n (%) | 2,328 (2.0%) | 211 (2.4%) | 2,429 (2.1%) | 164 (1.9%) | 7,206 (2.0%) | 572 (1.7%) | 11,963 (2.0%) | 947 (1.9%) | 0.01 |
| ACS/unstable angina; n (%) | 1,604 (1.4%) | 117 (1.3%) | 1,705 (1.5%) | 125 (1.4%) | 4,863 (1.3%) | 443 (1.3%) | 8,172 (1.4%) | 685 (1.3%) | 0.01 |
| Old MI; n (%) | 6,271 (5.5%) | 428 (4.8%) | 3,486 (3.1%) | 243 (2.8%) | 19,590 (5.4%) | 1,572 (4.7%) | 29,347 (4.9%) | 2,243 (4.4%) | 0.02 |
| Stable angina; n (%) | 6,380 (5.6%) | 540 (6.1%) | 4,778 (4.2%) | 382 (4.4%) | 17,135 (4.7%) | 1,710 (5.1%) | 28,293 (4.8%) | 2,632 (5.2%) | -0.02 |
| Coronary atherosclerosis and other forms of chronic ischemic heart disease; n (%) | 42,037 (36.9%) | 3,219 (36.2%) | 38,319 (33.6%) | 2,842 (32.5%) | 151,932 (41.5%) | 13,061 (39.1%) | 232,288 (39.1%) | 19,122 (37.5%) | 0.03 |
| Other atherosclerosis with ICD10; n (%) | 1,534 (1.3%) | 114 (1.3%) | 1,423 (1.2%) | 107 (1.2%) | 7,853 (2.1%) | 681 (2.0%) | 10,810 (1.8%) | 902 (1.8%) | 0.03 |
| other atheroscierosis with red to , ii (///) | 1,554 (1.576) | 114 (1.370) | 1,423 (1.270) | 107 (1.278) | 7,833 (2.170) | 081 (2.0%) | 10,810 (1.8%) | 302 (1.8%) | 0.00 |
| Previous cardiac procedure (CABG or PTCA or Stent); n (%) | 720 (0.6%) | 56 (0.6%) | 919 (0.8%) | 80 (0.9%) | 2,049 (0.6%) | 170 (0.5%) | 3,688 (0.6%) | 306 (0.6%) | 0.00 |
| History of CABG or PTCA; n (%) | 9,769 (8.6%) | 778 (8.7%) | 4,953 (4.3%) | 382 (4.4%) | 40,597 (11.1%) | 3,417 (10.2%) | 55,319 (9.3%) | 4,577 (9.0%) | 0.01 |
| Any stroke; n (%) | 5,024 (4.4%) | 347 (3.9%) | 4,490 (3.9%) | 355 (4.1%) | 20,639 (5.6%) | 1,835 (5.5%) | 30,153 (5.1%) | 2,537 (5.0%) | 0.00 |
| Ischemic stroke (w and w/o mention of cerebral | | | | | | | | | |
| infarction); n (%) | 4,945 (4.3%) | 339 (3.8%) | 4,425 (3.9%) | 349 (4.0%) | 20,378 (5.6%) | 1,815 (5.4%) | 29,748 (5.0%) | 2,503 (4.9%) | 0.00 |
| Hemorrhagic stroke; n (%) | 114 (0.1%) | 13 (0.1%) | 100 (0.1%) | 10 (0.1%) | 431 (0.1%) | 32 (0.1%) | 645 (0.1%) | 55 (0.1%) | 0.00 |
| TIA; n (%) | 847 (0.7%) | 56 (0.6%) | 801 (0.7%) | 63 (0.7%) | 3,716 (1.0%) | 337 (1.0%) | 5,364 (0.9%) | 456 (0.9%) | 0.00 |
| Other cerebrovascular disease; n (%) | 2,079 (1.8%) | 179 (2.0%) | 1,489 (1.3%) | 112 (1.3%) | 9,408 (2.6%) | 949 (2.8%) | 12,976 (2.2%) | 1,240 (2.4%) | -0.01 |
| Late effects of cerebrovascular disease; n (%) | 2,041 (1.8%) | 172 (1.9%) | 1,238 (1.1%) | 71 (0.8%) | 8,670 (2.4%) | 846 (2.5%) | 11,949 (2.0%) | 1,089 (2.1%) | -0.01 |
| Cerebrovascular procedure; n (%)<br>Heart failure (CHF); n (%) | 63 (0.1%) | 3 (0.0%) | 63 (0.1%)<br>10,022 (8.8%) | 3 (0.0%) | 192 (0.1%)<br>54,617 (14.9%) | 11 (0.0%) | 318 (0.1%)<br>78,434 (13.2%) | 17 (0.0%)<br>7,322 (14.3%) | 0.04<br>-0.03 |
| neart failure (Cnr), if (%) | 13,795 (12.1%) | 1,146 (12.9%) | 10,022 (6.6%) | 822 (9.4%) | 34,617 (14.9%) | 5,354 (16.0%) | 76,434 (13.2%) | 7,322 (14.3%) | -0.03 |
| Peripheral Vascular Disease (PVD) or PVD Surgery; n (%) | 10,030 (8.8%) | 875 (9.8%) | 6,941 (6.1%) | 559 (6.4%) | 45,805 (12.5%) | 4,977 (14.9%) | 62,776 (10.6%) | 6,411 (12.6%) | -0.06 |
| Atrial fibrillation; n (%) | 12,216 (10.7%) | 849 (9.5%) | 9,816 (8.6%) | 734 (8.4%) | 55,664 (15.2%) | 4,895 (14.7%) | 77,696 (13.1%) | 6,478 (12.7%) | 0.01 |
| Other cardiac dysrhythmia; n (%) | 13,746 (12.1%) | 1,109 (12.5%) | 9,751 (8.6%) | 803 (9.2%) | 55,599 (15.2%) | 5,545 (16.6%) | 79,096 (13.3%) | 7,457 (14.6%) | -0.04 |
| Cardiac conduction disorders; n (%) | 4,173 (3.7%) | 329 (3.7%) | 2,960 (2.6%) | 238 (2.7%) | 18,071 (4.9%) | 1,582 (4.7%) | 25,204 (4.2%) | 2,149 (4.2%) | 0.00 |
| Other CVD; n (%) | 16,453 (14.4%) | 1,283 (14.4%) | 13,648 (12.0%) | 1,135 (13.0%) | 65,860 (18.0%) | 6,376 (19.1%) | 95,961 (16.2%) | 8,794 (17.2%) | -0.03 |
| Diabetes-related complications | | | | | | | | | |
| Diabetic retinopathy; n (%) | 6,853 (6.0%) | 677 (7.6%) | 4,623 (4.1%) | 398 (4.6%) | 22,873 (6.2%) | 2,677 (8.0%) | 34,349 (5.8%) | 3,752 (7.4%) | -0.06 |
| Diabetes with other ophthalmic manifestations; n (%)<br>Retinal detachment, vitreous hemorrhage, vitrectomy; n | 793 (0.7%) | 58 (0.7%) | 3,389 (3.0%) | 255 (2.9%) | 8,854 (2.4%) | 943 (2.8%) | 13,036 (2.2%) | 1,256 (2.5%) | -0.02 |
| (%) | 459 (0.4%) | 62 (0.7%) | 356 (0.3%) | 52 (0.6%) | 1,303 (0.4%) | 165 (0.5%) | 2,118 (0.4%) | 279 (0.5%) | -0.01 |
| Retinal laser coagulation therapy; n (%) | 578 (0.5%) | 70 (0.8%) | 602 (0.5%) | 67 (0.8%) | 1,792 (0.5%) | 253 (0.8%) | 2,972 (0.5%) | 390 (0.8%) | -0.04 |
| Occurrence of Diabetic Neuropathy ; n (%) | 21,622 (19.0%) | 1,842 (20.7%) | 12,232 (10.7%) | 1,115 (12.8%) | 65,212 (17.8%) | 7,325 (21.9%) | 99,066 (16.7%) | 10,282 (20.1%) | -0.09 |

| Occurrence of diabetic nephropathy with ICD10 ; n (%) | 23,814 (20.9%) | 2,283 (25.6%) | 8,997 (7.9%) | 1,121 (12.8%) | 40,660 (11.1%) | 6,463 (19.3%) | 73,471 (12.4%) | 9,867 (19.3%) | -0.19 |
|---|---|---|---|---|---|---|---|---|---|
| Hypoglycemia ; n (%) | 2,895 (2.5%) | 227 (2.5%) | 3,373 (3.0%) | 207 (2.4%) | 10,042 (2.7%) | 1,090 (3.3%) | 16,310 (2.7%) | 1,524 (3.0%) | -0.02 |
| Hyperglycemia; n (%) | 5,084 (4.5%) | 547 (6.1%) | 3,784 (3.3%) | 344 (3.9%) | 17,473 (4.8%) | 2,169 (6.5%) | 26,341 (4.4%) | 3,060 (6.0%) | -0.07 |
| Discordance of florid alcoholotes and asid base below as a (0/) | 10.375 (0.00/) | 1.050 (11.00/) | 7.106 (6.30() | (20 /7 49/) | 20.074 (10.0%) | 4 024 (42 49/) | FC 442 (0 F8/) | F 700 (11 38/) | -0.06 |
| Disorders of fluid electrolyte and acid-base balance; n (%) Diabetic ketoacidosis; n (%) | 10,275 (9.0%)<br>356 (0.3%) | 1,058 (11.9%)<br>35 (0.4%) | 7,196 (6.3%)<br>391 (0.3%) | 620 (7.1%)<br>24 (0.3%) | 38,971 (10.6%)<br>1,273 (0.3%) | 4,031 (12.1%)<br>126 (0.4%) | 56,442 (9.5%)<br>2,020 (0.3%) | 5,709 (11.2%)<br>185 (0.4%) | -0.06 |
| Hyperosmolar hyperglycemic nonketotic syndrome | 330 (0.3%) | 33 (0.4%) | 391 (0.5%) | 24 (0.5%) | 1,273 (0.3%) | 126 (0.4%) | 2,020 (0.5%) | 165 (0.4%) | -0.02 |
| (HONK); n (%) | 590 (0.5%) | 55 (0.6%) | 452 (0.4%) | 41 (0.5%) | 1,806 (0.5%) | 217 (0.6%) | 2,848 (0.5%) | 313 (0.6%) | -0.01 |
| Diabetes with peripheral circulatory disorders with ICD- | | (, | | () | _,=== (====, | (=:==== | _,= .= (=.=,-, | 0 = 0 (0.07.7) | |
| 10 ; n (%) | 9,520 (8.4%) | 811 (9.1%) | 4,372 (3.8%) | 400 (4.6%) | 29,150 (8.0%) | 3,138 (9.4%) | 43,042 (7.2%) | 4,349 (8.5%) | -0.05 |
| Diabetic Foot; n (%) | 2,764 (2.4%) | 269 (3.0%) | 2,556 (2.2%) | 199 (2.3%) | 11,287 (3.1%) | 1,082 (3.2%) | 16,607 (2.8%) | 1,550 (3.0%) | -0.01 |
| Gangrene ; n (%) | 361 (0.3%) | 31 (0.3%) | 272 (0.2%) | 16 (0.2%) | 1,087 (0.3%) | 101 (0.3%) | 1,720 (0.3%) | 148 (0.3%) | 0.00 |
| Lower extremity amputation; n (%) | 894 (0.8%) | 96 (1.1%) | 413 (0.4%) | 38 (0.4%) | 2,771 (0.8%) | 277 (0.8%) | 4,078 (0.7%) | 411 (0.8%) | -0.01 |
| Osteomyelitis; n (%) | 772 (0.7%) | 78 (0.9%) | 681 (0.6%) | 46 (0.5%) | 2,477 (0.7%) | 211 (0.6%) | 3,930 (0.7%) | 335 (0.7%) | 0.00 |
| Skin infections; n (%) | 6,727 (5.9%) | 540 (6.1%) | 6,925 (6.1%) | 522 (6.0%) | 26,721 (7.3%) | 2,539 (7.6%) | 40,373 (6.8%) | 3,601 (7.1%) | -0.01 |
| Erectile dysfunction; n (%) | 2,715 (2.4%) | 241 (2.7%) | 2,209 (1.9%) | 216 (2.5%) | 6,905 (1.9%) | 647 (1.9%) | 11,829 (2.0%) | 1,104 (2.2%) | -0.01 |
| Diabetes with unspecified complication; n (%) | 5,499 (4.8%) | 613 (6.9%) | 3,886 (3.4%) | 389 (4.5%) | 16,369 (4.5%) | 2,081 (6.2%) | 25,754 (4.3%) | 3,083 (6.0%) | -0.08 |
| Diabetes mellitus without mention of complications; n (%) | 98,647 (86.5%) | 7,625 (85.6%) | 105,362 (92.4%) | 7,961 (91.1%) | 342,350 (93.5%) | 30,829 (92.3%) | 546,359 (92.0%) | 46,415 (90.9%) | 0.04 |
| (70) Hypertension: 1 inpatient or 2 outpatient claims within | 96,047 (60.5%) | 7,023 (83.0%) | 105,562 (92.4%) | 7,901 (91.176) | 342,330 (93.3%) | 30,629 (92.3%) | 340,339 (92.0%) | 40,413 (90.9%) | 0.04 |
| 365 days; n (%) | 98,566 (86.5%) | 7,879 (88.5%) | 82,028 (71.9%) | 6,834 (78.2%) | 336,292 (91.8%) | 31,533 (94.4%) | 516,886 (87.0%) | 46,246 (90.6%) | -0.11 |
| Hyperlipidemia ; n (%) | 81,202 (71.2%) | 6,711 (75.4%) | 64,841 (56.9%) | 5,646 (64.6%) | 275,172 (75.2%) | 26,459 (79.2%) | 421,215 (70.9%) | 38,816 (76.0%) | -0.12 |
| Edema; n (%) | 8,887 (7.8%) | 811 (9.1%) | 5,991 (5.3%) | 557 (6.4%) | 39,092 (10.7%) | 4,456 (13.3%) | 53,970 (9.1%) | 5,824 (11.4%) | -0.08 |
| Renal Dysfunction (non-diabetic) ; n (%) | 37,562 (33.0%) | 3,755 (42.2%) | 20,954 (18.4%) | 2,525 (28.9%) | 104,923 (28.7%) | 14,337 (42.9%) | 163,439 (27.5%) | 20,617 (40.4%) | -0.27 |
| Occurrence of acute renal disease; n (%) | 5,514 (4.8%) | 609 (6.8%) | 3,904 (3.4%) | 423 (4.8%) | 18,677 (5.1%) | 2,393 (7.2%) | 28,095 (4.7%) | 3,425 (6.7%) | -0.09 |
| Occurrence of chronic renal insufficiency; n (%) | 33,235 (29.2%) | 3,393 (38.1%) | 16,471 (14.4%) | 2,164 (24.8%) | 89,032 (24.3%) | 12,832 (38.4%) | 138,738 (23.4%) | 18,389 (36.0%) | -0.28 |
| Chronic kidney disease ; n (%) | 32,418 (28.4%) | 3,336 (37.5%) | 16,038 (14.1%) | 2,116 (24.2%) | 85,680 (23.4%) | 12,415 (37.2%) | 134,136 (22.6%) | 17,867 (35.0%) | -0.28 |
| CKD Stage 3-4; n (%) | 25,804 (22.6%) | 2,799 (31.4%) | 12,085 (10.6%) | 1,713 (19.6%) | 64,688 (17.7%) | 9,828 (29.4%) | 102,577 (17.3%) | 14,340 (28.1%) | -0.26 |
| Occurrence of hypertensive nephropathy; n (%) | 14,013 (12.3%) | 1,488 (16.7%) | 6,307 (5.5%) | 758 (8.7%) | 38,737 (10.6%) | 5,386 (16.1%) | 59,057 (9.9%) | 7,632 (15.0%) | -0.15 |
| Occurrence of miscellaneous renal insufficiency ; n (%) | 7,420 (6.5%) | 794 (8.9%) | 5,159 (4.5%) | 589 (6.7%) | 29,680 (8.1%) | 3,744 (11.2%) | 42,259 (7.1%) | 5,127 (10.0%) | -0.10 |
| Glaucoma or cataracts; n (%) | 22,333 (19.6%) | 1,771 (19.9%) | 17,722 (15.5%) | 1,514 (17.3%) | 91,357 (25.0%) | 9,149 (27.4%) | 131,412 (22.1%) | 12,434 (24.4%) | -0.05<br>-0.02 |
| Cellulitis or abscess of toe; n (%) Foot ulcer; n (%) | 1,682 (1.5%)<br>2,718 (2.4%) | 138 (1.5%)<br>257 (2.9%) | 1,126 (1.0%)<br>2,566 (2.3%) | 101 (1.2%)<br>194 (2.2%) | 5,368 (1.5%)<br>11,316 (3.1%) | 594 (1.8%)<br>1,073 (3.2%) | 8,176 (1.4%)<br>16,600 (2.8%) | 833 (1.6%)<br>1,524 (3.0%) | -0.02 |
| Bladder stones; n (%) | 159 (0.1%) | 16 (0.2%) | 126 (0.1%) | 17 (0.2%) | 657 (0.2%) | 66 (0.2%) | 942 (0.2%) | 99 (0.2%) | 0.00 |
| Kidney stones; n (%) | 2,539 (2.2%) | 272 (3.1%) | 2,472 (2.2%) | 260 (3.0%) | 9,310 (2.5%) | 1,017 (3.0%) | 14,321 (2.4%) | 1,549 (3.0%) | -0.04 |
| Urinary tract infections (UTIs); n (%) | 11,118 (9.8%) | 1,016 (11.4%) | 7,802 (6.8%) | 641 (7.3%) | 53,506 (14.6%) | 6,142 (18.4%) | 72,426 (12.2%) | 7,799 (15.3%) | -0.09 |
| Dipstick urinalysis; n (%) | 39,810 (34.9%) | 3,686 (41.4%) | 33,397 (29.3%) | 3,102 (35.5%) | 145,826 (39.8%) | 16,212 (48.5%) | 219,033 (36.9%) | 23,000 (45.1%) | -0.17 |
| Non-dipstick urinalysis; n (%) | 44,276 (38.8%) | 3,916 (44.0%) | 29,777 (26.1%) | 2,820 (32.3%) | 130,875 (35.7%) | 14,659 (43.9%) | 204,928 (34.5%) | 21,395 (41.9%) | -0.15 |
| Urine function test; n (%) | 2,905 (2.5%) | 212 (2.4%) | 2,885 (2.5%) | 281 (3.2%) | 12,778 (3.5%) | 1,377 (4.1%) | 18,568 (3.1%) | 1,870 (3.7%) | -0.03 |
| Cytology; n (%) | 888 (0.8%) | 90 (1.0%) | 1,110 (1.0%) | 120 (1.4%) | 3,902 (1.1%) | 439 (1.3%) | 5,900 (1.0%) | 649 (1.3%) | -0.03 |
| Cystos; n (%) | 1,367 (1.2%) | 111 (1.2%) | 1,490 (1.3%) | 151 (1.7%) | 5,876 (1.6%) | 563 (1.7%) | 8,733 (1.5%) | 825 (1.6%) | -0.01 |
| Other Covariates | | | | | | | | | |
| Liver disease; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | #VALUE! | 000 (0.0%) | #VALUE! |
| Osteoarthritis; n (%) | 18,149 (15.9%) | 1,516 (17.0%) | 13,857 (12.2%) | 1,082 (12.4%) | 85,234 (23.3%) | 8,776 (26.3%) | 117,240 (19.7%) | 11,374 (22.3%) | -0.06 |
| Other arthritis, arthropathies and musculoskeletal pain; n | | | | | | | | | |
| (%) | 40,678 (35.7%) | 3,528 (39.6%) | 36,555 (32.1%) | 2,991 (34.2%) | 165,558 (45.2%) | 16,538 (49.5%) | 242,791 (40.9%) | 23,057 (45.2%) | -0.09 |
| Dorsopathies; n (%)<br>Fractures; n (%) | 24,710 (21.7%)<br>3,692 (3.2%) | 2,038 (22.9%)<br>305 (3.4%) | 21,713 (19.0%)<br>3,370 (3.0%) | 1,834 (21.0%)<br>223 (2.6%) | 96,989 (26.5%)<br>16,248 (4.4%) | 9,505 (28.5%)<br>1,513 (4.5%) | 143,412 (24.1%)<br>23,310 (3.9%) | 13,377 (26.2%)<br>2,041 (4.0%) | -0.05<br>-0.01 |
| Falls; n (%) | 4,478 (3.9%) | 392 (4.4%) | 1,629 (1.4%) | 107 (1.2%) | 18,341 (5.0%) | 1,807 (5.4%) | 24,448 (4.1%) | 2,306 (4.5%) | -0.01 |
| Osteoporosis; n (%) | 5,505 (4.8%) | 541 (6.1%) | 3,204 (2.8%) | 263 (3.0%) | 28,297 (7.7%) | 3,994 (12.0%) | 37,006 (6.2%) | 4,798 (9.4%) | -0.02 |
| Hyperthyroidism; n (%) | 699 (0.6%) | 97 (1.1%) | 500 (0.4%) | 55 (0.6%) | 3,221 (0.9%) | 427 (1.3%) | 4,420 (0.7%) | 579 (1.1%) | -0.04 |
| Hypothyroidism ; n (%) | 17,357 (15.2%) | 1,673 (18.8%) | 11,200 (9.8%) | 1,124 (12.9%) | 54,516 (14.9%) | 5,258 (15.7%) | 83,073 (14.0%) | 8,055 (15.8%) | -0.05 |
| Other disorders of thyroid gland ; n (%) | 3,224 (2.8%) | 422 (4.7%) | 2,773 (2.4%) | 387 (4.4%) | 12,515 (3.4%) | 1,791 (5.4%) | 18,512 (3.1%) | 2,600 (5.1%) | -0.10 |
| Depression; n (%) | 9,096 (8.0%) | 805 (9.0%) | 7,304 (6.4%) | 557 (6.4%) | 38,741 (10.6%) | 3,845 (11.5%) | 55,141 (9.3%) | 5,207 (10.2%) | -0.03 |
| Anxiety; n (%) | 7,943 (7.0%) | 784 (8.8%) | 5,215 (4.6%) | 448 (5.1%) | 30,541 (8.3%) | 3,196 (9.6%) | 43,699 (7.4%) | 4,428 (8.7%) | -0.05 |
| Sleep_Disorder; n (%) | 8,147 (7.1%) | 590 (6.6%) | 11,134 (9.8%) | 870 (10.0%) | 29,743 (8.1%) | 2,723 (8.2%) | 49,024 (8.3%) | 4,183 (8.2%) | 0.00 |
| Dementia; n (%) | 5,612 (4.9%) | 540 (6.1%) | 3,565 (3.1%) | 223 (2.6%) | 32,684 (8.9%) | 3,540 (10.6%) | 41,861 (7.0%) | 4,303 (8.4%) | -0.05 |
| Delirium; n (%) | 1,424 (1.2%) | 149 (1.7%) | 1,104 (1.0%) | 72 (0.8%) | 7,315 (2.0%) | 849 (2.5%) | 9,843 (1.7%) | 1,070 (2.1%) | -0.03 |
| Psychosis; n (%) | 1,263 (1.1%) | 129 (1.4%) | 968 (0.8%) | 55 (0.6%) | 7,939 (2.2%) | 793 (2.4%) | 10,170 (1.7%) | 977 (1.9%) | -0.02 |
| Obesity; n (%) | 16,061 (14.1%) | 1,661 (18.7%) | 10,204 (8.9%) | 989 (11.3%) | 37,005 (10.1%) | 3,919 (11.7%) | 63,270 (10.6%) | 6,569 (12.9%) | -0.07 |
| Overweight; n (%) | 5,405 (4.7%) | 591 (6.6%) | 1,779 (1.6%) | 164 (1.9%) | 11,533 (3.1%) | 1,342 (4.0%) | 18,717 (3.2%) | 2,097 (4.1%) | -0.05 |
| Smoking; n (%) | 12,866 (11.3%) | 1,123 (12.6%) | 6,558 (5.8%) | 472 (5.4%) | 48,039 (13.1%) | 4,237 (12.7%) | 67,463 (11.4%) | 5,832 (11.4%) | 0.00 |
| Alcohol abuse or dependence; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | #VALUE!<br>#VALUE! | 00 (0.0%) | #VALUE! |
| Drug abuse or dependence; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%)<br>50,518 (13.8%) | 0 (0.0%) | | 00 (0.0%) | #VALUE!<br>0.00 |
| COPD; n (%) | 12,993 (11.4%) | 882 (9.9%) | 9,142 (8.0%) | 618 (7.1%) | 50,518 (13.8%) | 4,685 (14.0%) | 72,653 (12.2%) | 6,185 (12.1%) | 0.00 |

| Author (07) | 5.050 (5.20() | FCO (C 40() | 5 242 (4 50() | 425 (4.00() | 22.404.(5.40/) | 2 222 (5 70() | 22.576/5.70() | 2 240 (5 20/) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Asthma; n (%) | 5,959 (5.2%) | 569 (6.4%)<br>876 (9.8%) | 5,213 (4.6%)<br>10,424 (9.1%) | 426 (4.9%)<br>939 (10.7%) | 22,404 (6.1%) | 2,223 (6.7%) | 33,576 (5.7%) | 3,218 (6.3%)<br>4,032 (7.9%) | -0.03<br>-0.03 |
| Obstructive sleep apnea; n (%) | 9,320 (8.2%) | | | | 22,520 (6.2%) | 2,217 (6.6%) | 42,264 (7.1%) | | 0.00 |
| Pneumonia; n (%)<br>Imaging; n (%) | 3,866 (3.4%)<br>155 (0.1%) | 318 (3.6%)<br>17 (0.2%) | 3,558 (3.1%)<br>131 (0.1%) | 241 (2.8%)<br>7 (0.1%) | 16,296 (4.5%)<br>712 (0.2%) | 1,507 (4.5%)<br>54 (0.2%) | 23,720 (4.0%)<br>998 (0.2%) | 2,066 (4.0%)<br>78 (0.2%) | 0.00 |
| Diabetes Medications | 155 (0.1%) | 17 (0.2%) | 151 (0.176) | 7 (0.1%) | 712 (0.2%) | 34 (0.2%) | 996 (0.2%) | 76 (0.2%) | 0.00 |
| DM Medications - AGIs; n (%) | 359 (0.3%) | 32 (0.4%) | 308 (0.3%) | 32 (0.4%) | 1,322 (0.4%) | 202 (0.6%) | 1,989 (0.3%) | 266 (0.5%) | -0.03 |
| DM Medications - Adis, it (%) | 7,693 (6.7%) | 617 (6.9%) | 9,595 (8.4%) | 839 (9.6%) | 22,794 (6.2%) | 2,478 (7.4%) | 40,082 (6.7%) | 3,934 (7.7%) | -0.03 |
| DM Medications - Insulin; n (%) | 15,753 (13.8%) | 2,424 (27.2%) | 15,075 (13.2%) | 1,908 (21.8%) | 55,854 (15.3%) | 9,388 (28.1%) | 86,682 (14.6%) | 13,720 (26.9%) | -0.04 |
| DM Medications - Meglitinides; n (%) | 719 (0.6%) | 184 (2.1%) | 1,020 (0.9%) | 248 (2.8%) | 3,957 (1.1%) | 1,190 (3.6%) | 5,696 (1.0%) | 1,622 (3.2%) | -0.51 |
| DM Medications - Metformin; n (%) | 67,785 (59.5%) | 4,911 (55.2%) | 68,989 (60.5%) | 4,989 (57.1%) | 211,273 (57.7%) | 17,663 (52.9%) | 348,047 (58.6%) | 27,563 (54.0%) | 0.09 |
| Divi Medications - Metiorinin, ii (%) | 67,765 (59.5%) | 4,911 (33.2%) | 00,909 (00.5%) | 4,969 (37.1%) | 211,2/3 (37.7%) | 17,003 (32.9%) | 346,047 (36.0%) | 27,363 (34.0%) | 0.09 |
| Concomitant initiation or current use of SGLT2i; n (%) | 222 (0.2%) | 268 (3.0%) | 167 (0.1%) | 566 (6.5%) | 259 (0.1%) | 412 (1.2%) | #VALUE! | 1,246 (2.4%) | #VALUE! |
| Concomitant initiation or current use of AGIs; n (%) | 260 (0.2%) | 26 (0.3%) | 230 (0.2%) | 23 (0.3%) | 938 (0.3%) | 134 (0.4%) | 1,428 (0.2%) | 183 (0.4%) | -0.04 |
| concomment initiation of carrent asc or riols, in (70) | 200 (0.270) | 20 (0.570) | 250 (0.270) | 25 (0.570) | 330 (0.370) | 13 ( (0.170) | 1,120 (0.270) | 105 (0.170) | 0.01 |
| Concomitant initiation or current use of Glitazones; n (%) | 5,876 (5.2%) | 424 (4.8%) | 7,225 (6.3%) | 527 (6.0%) | 17,490 (4.8%) | 1,741 (5.2%) | 30,591 (5.1%) | 2,692 (5.3%) | -0.01 |
| Concomitant initiation or current use of Insulin; n (%) | 10,884 (9.5%) | 1,862 (20.9%) | 10,876 (9.5%) | 1,443 (16.5%) | 39,560 (10.8%) | 7,259 (21.7%) | 61,320 (10.3%) | 10,564 (20.7%) | -0.29 |
| Concomitant initiation or current use of Meglitinides; n | | | | | | | | | |
| (%) | 453 (0.4%) | 134 (1.5%) | 655 (0.6%) | 195 (2.2%) | 2,488 (0.7%) | 892 (2.7%) | 3,596 (0.6%) | 1,221 (2.4%) | -0.15 |
| Concomitant initiation or current use of Metformin; n (%) | 56,752 (49.8%) | 3,913 (43.9%) | 58,199 (51.0%) | 3,978 (45.5%) | 177,256 (48.4%) | 13,934 (41.7%) | 292,207 (49.2%) | 21,825 (42.8%) | 0.13 |
| Past use of SGLT2i; n (%) | 1 (0.0%) | 0 (0.0%) | 19 (0.0%) | 1 (0.0%) | 4 (0.0%) | 0 (0.0%) | #VALUE! | 001 (0.0%) | #VALUE! |
| Past use of AGIs ; n (%) | 99 (0.1%) | 6 (0.1%) | 78 (0.1%) | 9 (0.1%) | 384 (0.1%) | 68 (0.2%) | 561 (0.1%) | 83 (0.2%) | -0.03 |
| Past use of Glitazones ; n (%) | 1,817 (1.6%) | 193 (2.2%) | 2,371 (2.1%) | 312 (3.6%) | 5,304 (1.4%) | 737 (2.2%) | 9,492 (1.6%) | 1,242 (2.4%) | -0.06 |
| Past use of Insulin ; n (%) | 4,869 (4.3%) | 562 (6.3%) | 4,199 (3.7%) | 465 (5.3%) | 16,297 (4.5%) | 2,129 (6.4%) | 25,365 (4.3%) | 3,156 (6.2%) | -0.09 |
| Past use of Meglitinides ; n (%) | 266 (0.2%) | 50 (0.6%) | 365 (0.3%) | 53 (0.6%) | 1,469 (0.4%) | 298 (0.9%) | 2,100 (0.4%) | 401 (0.8%) | -0.05 |
| Past use of metformin ; n (%) | 11,033 (9.7%) | 998 (11.2%) | 10,790 (9.5%) | 1,011 (11.6%) | 34,017 (9.3%) | 3,729 (11.2%) | 55,840 (9.4%) | 5,738 (11.2%) | -0.06 |
| Other Medications | | | | | | | | | |
| Use of ACE inhibitors; n (%) | 52,181 (45.8%) | 3,676 (41.3%) | 50,776 (44.5%) | 3,495 (40.0%) | 163,750 (44.7%) | 12,790 (38.3%) | 266,707 (44.9%) | 19,961 (39.1%) | 0.12 |
| Use of ARBs; n (%) | 28,284 (24.8%) | 2,777 (31.2%) | 28,769 (25.2%) | 2,858 (32.7%) | 97,329 (26.6%) | 11,969 (35.8%) | 154,382 (26.0%) | 17,604 (34.5%) | -0.19 |
| Use of Loop Diuretics ; n (%) | 20,910 (18.3%) | 1,833 (20.6%) | 19,444 (17.1%) | 1,688 (19.3%) | 88,445 (24.2%) | 9,010 (27.0%) | 128,799 (21.7%) | 12,531 (24.6%) | -0.07 |
| Use of other diuretics; n (%) | 4,374 (3.8%) | 435 (4.9%) | 4,519 (4.0%) | 441 (5.0%) | 16,078 (4.4%) | 1,632 (4.9%) | 24,971 (4.2%) | 2,508 (4.9%) | -0.03 |
| Use of nitrates-United; n (%) | 10,414 (9.1%) | 772 (8.7%) | 11,043 (9.7%) | 747 (8.6%) | 42,214 (11.5%) | 3,874 (11.6%) | 63,671 (10.7%) | 5,393 (10.6%) | 0.00 |
| Use of other hypertension drugs; n (%) | 10,825 (9.5%) | 920 (10.3%) | 9,771 (8.6%) | 794 (9.1%) | 37,611 (10.3%) | 3,867 (11.6%) | 58,207 (9.8%) | 5,581 (10.9%) | -0.04 |
| Use of digoxin; n (%) | 3,374 (3.0%) | 219 (2.5%) | 3,676 (3.2%) | 272 (3.1%) | 16,616 (4.5%) | 1,350 (4.0%) | 23,666 (4.0%) | 1,841 (3.6%) | 0.02 |
| Use of Anti-arrhythmics; n (%) | 2,343 (2.1%) | 176 (2.0%) | 2,629 (2.3%) | 216 (2.5%) | 10,532 (2.9%) | 1,055 (3.2%) | 15,504 (2.6%) | 1,447 (2.8%) | -0.01<br>-0.10 |
| Use of COPD/asthma meds; n (%) | 16,005 (14.0%) | 1,608 (18.1%) | 16,846 (14.8%) | 1,465 (16.8%) | 61,145 (16.7%) | 7,008 (21.0%) | 93,996 (15.8%) | 10,081 (19.8%) | -0.10 |
| Use of statins; n (%) Use of other lipid-lowering drugs; n (%) | 77,398 (67.9%)<br>12,848 (11.3%) | 6,449 (72.4%)<br>1,223 (13.7%) | 74,851 (65.6%)<br>16,602 (14.6%) | 6,099 (69.8%)<br>1,528 (17.5%) | 249,773 (68.2%)<br>42,913 (11.7%) | 24,666 (73.8%)<br>4,879 (14.6%) | 402,022 (67.7%)<br>72,363 (12.2%) | 37,214 (72.9%)<br>7,630 (14.9%) | -0.11 |
| Use of antiplatelet agents; n (%) | 19,863 (17.4%) | 1,752 (19.7%) | 23,347 (20.5%) | 1,865 (21.3%) | 70,313 (19.2%) | 7,213 (21.6%) | 113,523 (19.1%) | 10,830 (21.2%) | -0.05 |
| Use of oral anticoagulants (Dabigatran, Rivaroxaban, | 19,003 (17.4%) | 1,/32 (19./%) | 23,347 (20.3%) | 1,003 (21.5%) | 70,515 (19.2%) | 7,213 (21.0%) | 113,323 (19.1%) | 10,030 (21.2%) | -0.05 |
| Apixaban, Warfarin); n (%) | 10,082 (8.8%) | 749 (8.4%) | 9,718 (8.5%) | 793 (9.1%) | 44,487 (12.2%) | 4,020 (12.0%) | 64,287 (10.8%) | 5,562 (10.9%) | 0.00 |
| Use of heparin and other low-molecular weight heparins; | 10,002 (0.070) | 743 (0.470) | 3,710 (0.370) | 755 (5.170) | 44,407 (12.270) | 4,020 (12.070) | 04,207 (10.070) | 3,302 (10.370) | 0.00 |
| n (%) | 469 (0.4%) | 50 (0.6%) | 23 (0.0%) | 1 (0.0%) | 1,950 (0.5%) | 157 (0.5%) | 2,442 (0.4%) | 208 (0.4%) | 0.00 |
| Use of NSAIDs; n (%) | 15,070 (13.2%) | 1,274 (14.3%) | 15,571 (13.7%) | 1,294 (14.8%) | 52,701 (14.4%) | 5,618 (16.8%) | 83,342 (14.0%) | 8,186 (16.0%) | -0.06 |
| Use of oral corticosteroids; n (%) | 18,755 (16.5%) | 1,600 (18.0%) | 18,563 (16.3%) | 1,501 (17.2%) | 70,096 (19.1%) | 6,887 (20.6%) | 107,414 (18.1%) | 9,988 (19.6%) | -0.04 |
| Use of bisphosphonate (United); n (%) | 2,806 (2.5%) | 227 (2.5%) | 1,930 (1.7%) | 137 (1.6%) | 11,978 (3.3%) | 1,663 (5.0%) | 16,714 (2.8%) | 2,027 (4.0%) | -0.07 |
| Use of opioids; n (%) | 28,735 (25.2%) | 2,259 (25.4%) | 30,829 (27.0%) | 2,294 (26.3%) | 100,433 (27.4%) | 9,027 (27.0%) | 159,997 (26.9%) | 13,580 (26.6%) | 0.01 |
| Use of antidepressants; n (%) | 25,596 (22.5%) | 2,240 (25.2%) | 25,079 (22.0%) | 2,142 (24.5%) | 92,511 (25.3%) | 9,505 (28.5%) | 143,186 (24.1%) | 13,887 (27.2%) | -0.07 |
| Use of antipsychotics; n (%) | 2,655 (2.3%) | 305 (3.4%) | 2,436 (2.1%) | 213 (2.4%) | 12,838 (3.5%) | 1,506 (4.5%) | 17,929 (3.0%) | 2,024 (4.0%) | -0.05 |
| Use of anticonvulsants; n (%) | 17,961 (15.8%) | 1,682 (18.9%) | 14,538 (12.7%) | 1,316 (15.1%) | 63,740 (17.4%) | 7,030 (21.0%) | 96,239 (16.2%) | 10,028 (19.6%) | -0.09 |
| Use of lithium; n (%) | 160 (0.1%) | 9 (0.1%) | 188 (0.2%) | 15 (0.2%) | 453 (0.1%) | 40 (0.1%) | 801 (0.1%) | 064 (0.1%) | 0.00 |
| Use of Benzos; n (%) | 10,450 (9.2%) | 1,032 (11.6%) | 13,201 (11.6%) | 1,036 (11.9%) | 38,343 (10.5%) | 4,251 (12.7%) | 61,994 (10.4%) | 6,319 (12.4%) | -0.06 |
| Use of anxiolytics/hypnotics; n (%) | 6,200 (5.4%) | 596 (6.7%) | 7,418 (6.5%) | 642 (7.3%) | 23,082 (6.3%) | 2,419 (7.2%) | 36,700 (6.2%) | 3,657 (7.2%) | -0.04 |
| Use of dementia meds; n (%) | 3,527 (3.1%) | 323 (3.6%) | 2,889 (2.5%) | 206 (2.4%) | 21,174 (5.8%) | 2,631 (7.9%) | 27,590 (4.6%) | 3,160 (6.2%) | -0.07 |
| Use of antiparkinsonian meds; n (%) | 2,831 (2.5%) | 261 (2.9%) | 2,799 (2.5%) | 207 (2.4%) | 13,280 (3.6%) | 1,369 (4.1%) | 18,910 (3.2%) | 1,837 (3.6%) | -0.02 |
| Any use of pramlintide; n (%) | 8 (0.0%) | 5 (0.1%) | 29 (0.0%) | 5 (0.1%) | ** | ** | ** | ** | #VALUE! |
| Any use of 1st generation sulfonylureas; n (%) | 34 (0.0%) | 1 (0.0%) | 92 (0.1%) | 1 (0.0%) | ** | ** | ** | ** | 0.00 |
| Entresto (sacubitril/valsartan); n (%) | 153 (0.1%) | 25 (0.3%) | 46 (0.0%) | 6 (0.1%) | 212 (0.1%) | 40 (0.1%) | 411 (0.1%) | 071 (0.1%) | 0.00 |
| Labs | | | | | | | 228,016 | 17,640 | |
| Lab values- HbA1c (%); n (%) | 38,300 (33.6%) | 3,628 (40.7%) | 7,256 (6.4%) | 411 (4.7%) | N/A | N/A | 45,556 (20.0%) | 4,039 (22.9%) | -0.07 |
| Lab values- HbA1c (%) (within 3 months); n (%) | 29,271 (25.7%) | 2,900 (32.6%) | 5,567 (4.9%) | 334 (3.8%) | N/A | N/A | 34,838 (15.3%) | 3,234 (18.3%) | -0.08 |
| Lab values- HbA1c (%) (within 6 months); n (%) | 38,300 (33.6%) | 3,628 (40.7%) | 7,256 (6.4%) | 411 (4.7%) | N/A | N/A | 45,556 (20.0%) | 4,039 (22.9%) | -0.07 |
| Lab values- BNP; n (%) | 940 (0.8%) | 116 (1.3%) | 159 (0.1%) | 11 (0.1%) | N/A | N/A | 1,099 (0.5%) | 127 (0.7%) | -0.03 |
| Lab values- BNP (within 3 months); n (%) | 586 (0.5%) | 66 (0.7%) | 96 (0.1%) | 8 (0.1%) | N/A | N/A | 682 (0.3%) | 074 (0.4%) | -0.02 |
| Lab values- BNP (within 6 months); n (%) | 940 (0.8%) | 116 (1.3%) | 159 (0.1%) | 11 (0.1%) | N/A | N/A | 1,099 (0.5%) | 127 (0.7%) | -0.03 |
| Lab values- BUN (mg/dl); n (%) | 39,671 (34.8%) | 3,848 (43.2%) | 5,599 (4.9%) | 460 (5.3%) | N/A | N/A | 45,270 (19.9%) | 4,308 (24.4%) | -0.11 |

| | | | | | | | | _ | |
|---|---|---|---|---|---|---|---|---|---|
| Lab values- BUN (mg/dl) (within 3 months); n (%) | 30,338 (26.6%) | 3,054 (34.3%) | 4,205 (3.7%) | 362 (4.1%) | N/A | N/A | 34,543 (15.1%) | 3,416 (19.4%) | -0.11 |
| Lab values- BUN (mg/dl) (within 6 months); n (%) | 39,671 (34.8%) | 3,848 (43.2%) | 5,599 (4.9%) | 460 (5.3%) | N/A | N/A | 45,270 (19.9%) | 4,308 (24.4%) | -0.11 |
| Lab values- Creatinine (mg/dl); n (%) | 40,504 (35.5%) | 3,967 (44.6%) | 5,824 (5.1%) | 501 (5.7%) | N/A | N/A | 46,328 (20.3%) | 4,468 (25.3%) | -0.12 |
| Lab vardes creatinine (mg/ar/), ir (70) | 40,504 (55.570) | 3,507 (44.070) | 3,624 (3.170) | 301 (3.770) | 19/5 | 19/6 | 40,320 (20.370) | 4,400 (23.370) | 0.12 |
| Lab values- Creatinine (mg/dl) (within 3 months); n (%) | 30,955 (27.2%) | 3,154 (35.4%) | 4,374 (3.8%) | 392 (4.5%) | N/A | N/A | 35,329 (15.5%) | 3,546 (20.1%) | -0.12 |
| Lab values- Creatinine (mg/dl) (within 6 months); n (%) | 40,504 (35.5%) | 3,967 (44.6%) | 5,824 (5.1%) | 501 (5.7%) | N/A | N/A | 46,328 (20.3%) | 4,468 (25.3%) | -0.12 |
| Lab values- HDL level (mg/dl); n (%) | 31,938 (28.0%) | 3,092 (34.7%) | 6,175 (5.4%) | 398 (4.6%) | N/A | N/A | 38,113 (16.7%) | 3,490 (19.8%) | -0.08 |
| tab values Tibe level (Ing. al.), II (70) | 32,330 (20.070) | 3,032 (3 70) | 0,173 (3.170) | 330 (1.0%) | .,,, | .,,,, | 50,115 (10.775) | 3,130 (23.070) | 0.00 |
| | // | | | | | | | | |
| Lab values- HDL level (mg/dl) (within 3 months); n (%) | 23,022 (20.2%) | 2,313 (26.0%) | 4,413 (3.9%) | 307 (3.5%) | N/A | N/A | 27,435 (12.0%) | 2,620 (14.9%) | -0.09 |
| Lab values- HDL level (mg/dl) (within 6 months); n (%) | 31,938 (28.0%) | 3,092 (34.7%) | 6,175 (5.4%) | 398 (4.6%) | N/A | N/A | 38,113 (16.7%) | 3,490 (19.8%) | -0.08 |
| Lab values- LDL level (mg/dl); n (%) | 32,964 (28.9%) | 3,182 (35.7%) | 6,625 (5.8%) | 403 (4.6%) | N/A | N/A | 39,589 (17.4%) | 3,585 (20.3%) | -0.07 |
| Lab values EBETever (IIIg/ai/, II (/v) | 32,304 (20.370) | 3,102 (33.770) | 0,023 (3.0%) | 403 (4.070) | 14/5 | 11/75 | 33,363 (17.476) | 3,303 (20.370) | 0.07 |
| | | | . === / / | | | | | | |
| Lab values- LDL level (mg/dl) (within 3 months); n (%) | 23,766 (20.8%) | 2,384 (26.8%) | 4,732 (4.1%) | 310 (3.5%) | N/A | N/A | 28,498 (12.5%) | 2,694 (15.3%) | -0.08 |
| Lab values- LDL level (mg/dl) (within 6 months); n (%) | 32,964 (28.9%) | 3,182 (35.7%) | 6,625 (5.8%) | 403 (4.6%) | N/A | N/A | 39,589 (17.4%) | 3,585 (20.3%) | -0.07 |
| Lab values- NT-proBNP; n (%) | 131 (0.1%) | 12 (0.1%) | 12 (0.0%) | 2 (0.0%) | N/A | N/A | 143 (0.1%) | 14 (0.1%) | 0.00 |
| Lab values- NT-proBNP (within 3 months); n (%) | 84 (0.1%) | 6 (0.1%) | 6 (0.0%) | 1 (0.0%) | N/A | N/A | 90 (0.0%) | 7 (0.0%) | 0.00 |
| | | | | | | | | | - |
| Lab values- NT-proBNP (within 6 months); n (%) | 131 (0.1%) | 12 (0.1%) | 12 (0.0%) | 2 (0.0%) | N/A | N/A | 143 (0.1%) | 14 (0.1%) | - |
| Lab values- Total cholesterol (mg/dl); n (%) | 32,336 (28.4%) | 3,154 (35.4%) | 6,131 (5.4%) | 405 (4.6%) | N/A | N/A | 38,467 (16.9%) | 3,559 (20.2%) | -0.08 |
| Lab values-Total cholesterol (mg/dl) (within 3 months); n | | | | | | | | | |
| (%) | 23,343 (20.5%) | 2,357 (26.5%) | 4,361 (3.8%) | 312 (3.6%) | N/A | N/A | 27,704 (12.2%) | 2,669 (15.1%) | -0.08 |
| • • | | 2,337 (20.3%) | 4,301 (3.8%) | 312 (3.0%) | N/A | 11// | 27,704 (12.276) | 2,009 (13.176) | -0.08 |
| Lab values-Total cholesterol (mg/dl) (within 6 months); n | | | | | | | | | |
| (%) | 32,336 (28.4%) | 3,154 (35.4%) | 6,131 (5.4%) | 405 (4.6%) | N/A | N/A | 38,467 (16.9%) | 3,559 (20.2%) | -0.08 |
| Lab values-Triglyceride level (mg/dl); n (%) | 32,012 (28.1%) | 3,140 (35.3%) | 6,014 (5.3%) | 400 (4.6%) | N/A | N/A | 38,026 (16.7%) | 3,540 (20.1%) | -0.09 |
| Lab values-Triglyceride level (mg/dl) (within 3 months); n | | | | | | | | | |
| (%) | 23,144 (20.3%) | 2,346 (26.3%) | 4,302 (3.8%) | 307 (3.5%) | N/A | N/A | 27,446 (12.0%) | 2,653 (15.0%) | -0.09 |
| | 23,144 (20.3%) | 2,346 (26.3%) | 4,302 (3.8%) | 307 (3.5%) | N/A | IN/A | 27,446 (12.0%) | 2,033 (13.0%) | -0.09 |
| Lab values-Triglyceride level (mg/dl) (within 6 months); n | | | | | | | | | |
| (%) | 32,012 (28.1%) | 3,140 (35.3%) | 6,014 (5.3%) | 400 (4.6%) | N/A | N/A | 38,026 (16.7%) | 3,540 (20.1%) | -0.09 |
| Lab result number- HbA1c (%) mean (only 2 to 20 | | | | | | | | | |
| included) | 38,074 | 3,615 | 5,890 | 390 | N/A | N/A | 43,964 | 4,005 | |
| | 7.99 (1.81) | 8.01 (1.81) | 8.11 (1.90) | 7.88 (1.83) | N/A | N/A | 8.01 (1.82) | 8.00 (1.81) | 0.01 |
| mean (sd) | | | | | | | | | |
| median [IQR] | 7.55 [6.80, 8.73] | 7.60 [6.70, 8.80] | 7.60 [6.80, 8.95] | 7.42 [6.60, 8.60] | N/A | N/A | 7.56 (1.82) | 7.58 (1.81) | -0.01 |
| Missing; n (%) | 75,917 (66.6%) | 5,289 (59.4%) | 108,135 (94.8%) | 8,346 (95.5%) | N/A | N/A | 184,052 (80.7%) | 13,635 (77.3%) | 0.08 |
| Lab result number- BNP mean | 940 | 116 | 159 | 11 | N/A | N/A | 1,099 | 127 | |
| mean (sd) | 227.35 (358.83) | 199.85 (371.31) | 2,946.36 (33,054.02) | 607.19 (1,393.52) | N/A | N/A | 620.73 (12554.50) | 235.13 (533.36) | 0.04 |
| | , , | | | | | | | , , | |
| median [IQR] | 97.30 [38.75, 251.23] | 82.60 [32.35, 208.35] | 109.00 [40.00, 327.00] | 49.00 [15.10, 188.00] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| | | | | | N/A | N/A | 226,917 (99.5%) | 17,513 (99.3%) | 0.03 |
| Missing; n (%) | 113,051 (99.2%) | 8,788 (98.7%) | 113,866 (99.9%) | 8,725 (99.9%) | ,,, | 11/7 | | | |
| - · · · · | | | | 8,725 (99.9%)<br>460 | | | | 4.308 | |
| Lab result number- BUN (mg/dl) mean | 39,671 | 3,848 | 5,599 | 460 | N/A | N/A | 45,270 | 4,308<br>52.40 (1978.94) | 0.02 |
| Lab result number- BUN (mg/dl) meanmean (sd) | 39,671<br>20.56 (9.20) | 3,848<br>22.06 (10.35) | 5,599<br>782.69 (11,615.02) | 460<br>306.16 (6,060.48) | N/A<br>N/A | N/A<br>N/A | 45,270<br>114.82 (4084.57) | 52.40 (1978.94) | 0.02 |
| Lab result number- BUN (mg/dl) mean<br>mean (sd)<br>median [IQR] | 39,671<br>20.56 (9.20)<br>18.50 [14.50, 24.00] | 3,848<br>22.06 (10.35)<br>19.67 [15.00, 27.00] | 5,599<br>782.69 (11,615.02)<br>17.00 [13.50, 22.00] | 460<br>306.16 (6,060.48)<br>18.25 [14.00, 25.88] | N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A | 45,270<br>114.82 (4084.57)<br>#VALUE! | 52.40 (1978.94)<br>#VALUE! | #VALUE! |
| Lab result number- BUN (mg/dl) meanmean (sd) | 39,671<br>20.56 (9.20) | 3,848<br>22.06 (10.35) | 5,599<br>782.69 (11,615.02) | 460<br>306.16 (6,060.48) | N/A<br>N/A | N/A<br>N/A | 45,270<br>114.82 (4084.57) | 52.40 (1978.94) | |
| Lab result number-BUN (mg/dl) mean<br>mean (sd)<br>median [IQR]<br>Missing; n (%) | 39,671<br>20.56 (9.20)<br>18.50 [14.50, 24.00] | 3,848<br>22.06 (10.35)<br>19.67 [15.00, 27.00] | 5,599<br>782.69 (11,615.02)<br>17.00 [13.50, 22.00] | 460<br>306.16 (6,060.48)<br>18.25 [14.00, 25.88] | N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A | 45,270<br>114.82 (4084.57)<br>#VALUE! | 52.40 (1978.94)<br>#VALUE! | #VALUE! |
| Lab result number-BUN (mg/dl) mean<br>mean (sd)<br>median [IQR]<br>Missing; n (%)<br>Lab result number-Creatinine (mg/dl) mean (only 0.1 to | 39,671<br>20.56 (9.20)<br>18.50 [14.50, 24.00]<br>74,320 (65.2%) | 3,848<br>22.06 (10.35)<br>19.67 [15.00, 27.00]<br>5,056 (56.8%) | 5,599<br>782.69 (11,615.02)<br>17.00 [13.50, 22.00]<br>108,426 (95.1%) | 460<br>306.16 (6,060.48)<br>18.25 [14.00, 25.88]<br>8,276 (94.7%) | N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A | 45,270<br>114.82 (4084.57)<br>#VALUE!<br>182,746 (80.1%) | 52.40 (1978.94)<br>#VALUE!<br>13,332 (75.6%) | #VALUE! |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included) | 39,671<br>20.56 (9.20)<br>18.50 [14.50, 24.00]<br>74,320 (65.2%)<br>40,229 | 3,848<br>22.06 (10.35)<br>19.67 [15.00, 27.00]<br>5,056 (56.8%) | 5,599<br>782.69 (11,615.02)<br>17.00 [13.50, 22.00]<br>108,426 (95.1%)<br>5,443 | 306.16 (6,060.48)<br>18.25 [14.00, 25.88]<br>8,276 (94.7%) | N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A | 45,270<br>114.82 (4084.57)<br>#VALUE!<br>182,746 (80.1%)<br>45,672 | 52.40 (1978.94)<br>#VALUE!<br>13,332 (75.6%) | #VALUE!<br>0.11 |
| Lab result number- BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number- Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd) | 39,671<br>20.56 (9.20)<br>18.50 [14.50, 24.00]<br>74,320 (65.2%)<br>40,229<br>1.14 (0.45) | 3,848<br>22.06 (10.35)<br>19.67 (15.00, 27.00)<br>5,056 (56.8%)<br>3,945<br>1.24 (0.52) | 5,599 782.69 (11,615.02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) | 460<br>306.16 (6,060.48)<br>18.25 [14.00, 25.88]<br>8,276 (94.7%)<br>469<br>1.18 (0.61) | N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A | 45,270<br>114.82 (4084.57)<br>#VALUE!<br>182,746 (80.1%)<br>45,672<br>1.13 (0.45) | 52.40 (1978.94)<br>#VALUE!<br>13,332 (75.6%)<br>4,414<br>1.23 (0.53) | #VALUE!<br>0.11 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included) | 39,671<br>20,56 (9,20)<br>18.50 [14.50, 24.00]<br>74,320 (65.2%)<br>40,229<br>1.14 (0.45)<br>1.04 [0.85, 1.32] | 3,848<br>22.06 (10.35)<br>19.67 [15.00, 27.00]<br>5,056 (56.8%)<br>3,945<br>1.24 (0.52)<br>1.14 [0.88, 1.48] | 5,599 782.69 (11,615.02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] | 460<br>306.16 (6,060.48)<br>18.25 [14.00, 25.88]<br>8,276 (94.7%)<br>469<br>1.18 (0.61)<br>1.02 [0.84, 1.35] | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | 45,270<br>114.82 (4084.57)<br>#VALUE!<br>182,746 (80.1%)<br>45,672<br>1.13 (0.45)<br>1.04 (0.45) | 52.40 (1978.94)<br>#VALUE!<br>13,332 (75.6%)<br>4,414<br>1.23 (0.53)<br>1.13 (0.53) | #VALUE!<br>0.11<br>-0.20<br>-0.18 |
| Lab result number- BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number- Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd) | 39,671<br>20.56 (9.20)<br>18.50 [14.50, 24.00]<br>74,320 (65.2%)<br>40,229<br>1.14 (0.45) | 3,848<br>22.06 (10.35)<br>19.67 (15.00, 27.00)<br>5,056 (56.8%)<br>3,945<br>1.24 (0.52) | 5,599 782.69 (11,615.02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) | 460<br>306.16 (6,060.48)<br>18.25 [14.00, 25.88]<br>8,276 (94.7%)<br>469<br>1.18 (0.61) | N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A | 45,270<br>114.82 (4084.57)<br>#VALUE!<br>182,746 (80.1%)<br>45,672<br>1.13 (0.45) | 52.40 (1978.94)<br>#VALUE!<br>13,332 (75.6%)<br>4,414<br>1.23 (0.53) | #VALUE!<br>0.11 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number- Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) | 39,671<br>20,56 (9,20)<br>18.50 [14.50, 24.00]<br>74,320 (65.2%)<br>40,229<br>1.14 (0.45)<br>1.04 [0.85, 1.32] | 3,848<br>22.06 (10.35)<br>19.67 [15.00, 27.00]<br>5,056 (56.8%)<br>3,945<br>1.24 (0.52)<br>1.14 [0.88, 1.48] | 5,599 782.69 (11,615.02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] | 460<br>306.16 (6,060.48)<br>18.25 [14.00, 25.88]<br>8,276 (94.7%)<br>469<br>1.18 (0.61)<br>1.02 [0.84, 1.35] | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | 45,270<br>114.82 (4084.57)<br>#VALUE!<br>182,746 (80.1%)<br>45,672<br>1.13 (0.45)<br>1.04 (0.45) | 52.40 (1978.94)<br>#VALUE!<br>13,332 (75.6%)<br>4,414<br>1.23 (0.53)<br>1.13 (0.53) | #VALUE!<br>0.11<br>-0.20<br>-0.18 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [lQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [lQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 | 39,671<br>20.56 (9.20)<br>18.50 [14.50, 24.00]<br>74,320 (65.2%)<br>40,229<br>1.14 (0.45)<br>1.04 [0.85, 1.32]<br>73,762 (64.7%) | 3,848 22.06 (10.35) 19.67 [15.00, 27.00] 5,056 (56.8%) 3,945 1.24 (0.52) 1.14 [0.88, 1.48] 4,959 (55.7%) | 5,599 782.69 (11,615.02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] 108,582 (95.2%) | 460<br>306.16 (6,060.48)<br>18.25 [14.00, 25.88]<br>8,276 (94.7%)<br>469<br>1.18 (0.61)<br>1.02 [0.84, 1.35]<br>8,267 (94.6%) | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | 45,270<br>114.82 (4084.57)<br>#VALUE!<br>182,746 (80.1%)<br>45,672<br>1.13 (0.45)<br>1.04 (0.45)<br>182,344 (80.0%) | 52.40 (1978.94)<br>#VALUEI<br>13,332 (75.6%)<br>4,414<br>1.23 (0.53)<br>1.13 (0.53)<br>13,226 (75.0%) | #VALUE!<br>0.11<br>-0.20<br>-0.18 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included) | 39,671<br>20.56 (9.20)<br>18.50 [14.50, 24.00]<br>74,320 (65.2%)<br>40,229<br>1.14 (0.45)<br>1.04 [0.85, 1.32]<br>73,762 (64.7%) | 3,848<br>22.06 (10.35)<br>19.67 [15.00, 27.00]<br>5,056 (56.8%)<br>3,945<br>1.24 (0.52)<br>1.14 [0.88, 1.48]<br>4,959 (55.7%) | 5,599 782.69 (11,615.02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] 108,582 (95.2%) | 460<br>306.16 (6,060.48)<br>18.25 [14.00, 25.88]<br>8,276 (94.7%)<br>469<br>1.18 (0.61)<br>1.02 [0.84, 1.35]<br>8,267 (94.6%) | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | 45,270<br>114.82 (4084.57)<br>#VALUEI<br>182,746 (80.1%)<br>45,672<br>1.13 (0.45)<br>1.04 (0.45)<br>182,344 (80.0%) | 52.40 (1978.94)<br>#VALUEI<br>13,332 (75.6%)<br>4,414<br>1.23 (0.53)<br>1.13 (0.53)<br>13,226 (75.0%) | #VALUE!<br>0.11<br>-0.20<br>-0.18<br>0.12 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)mean (sd) | 39,671<br>20.56 (9.20)<br>18.50 [14.50, 24.00]<br>74,320 (65.2%)<br>40,229<br>1.14 (0.45)<br>1.04 [0.85, 1.32]<br>73,762 (64.7%)<br>31,938<br>46.04 (13.96) | 3,848 22.06 (10.35) 19.67 [15.00, 27.00] 5,056 (56.8%) 3,945 1.24 (0.52) 1.14 [0.88, 1.48] 4,959 (55.7%) 3,092 46.52 (14.16) | 5,599 782.69 (11,615.02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] 108,582 (95.2%) 6,157 43.97 (14.10) | 460<br>306.16 (6,060.48)<br>18.25 [14.00, 25.88]<br>8,276 (94.7%)<br>469<br>1.18 (0.61)<br>1.02 [0.84, 1.35]<br>8,267 (94.6%)<br>397<br>51.75 (174.25) | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A | 45,270<br>114.82 (4084.57)<br>#VALUE!<br>182,746 (80.1%)<br>45,672<br>1.13 (0.45)<br>1.04 (0.45)<br>182,344 (80.0%)<br>38,095<br>45,71 (13.98) | 52.40 (1978.94) #WALUE! 13,332 (75.6%) 4,414 1.23 (0.53) 1.13 (0.53) 13,226 (75.0%) 3,489 47.12 (60.22) | #VALUE!<br>0.11<br>-0.20<br>-0.18<br>0.12 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included) | 39,671<br>20.56 (9.20)<br>18.50 [14.50, 24.00]<br>74,320 (65.2%)<br>40,229<br>1.14 (0.45)<br>1.04 [0.85, 1.32]<br>73,762 (64.7%) | 3,848<br>22.06 (10.35)<br>19.67 [15.00, 27.00]<br>5,056 (56.8%)<br>3,945<br>1.24 (0.52)<br>1.14 [0.88, 1.48]<br>4,959 (55.7%) | 5,599 782.69 (11,615.02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] 108,582 (95.2%) | 460<br>306.16 (6,060.48)<br>18.25 [14.00, 25.88]<br>8,276 (94.7%)<br>469<br>1.18 (0.61)<br>1.02 [0.84, 1.35]<br>8,267 (94.6%) | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | 45,270<br>114.82 (4084.57)<br>#VALUEI<br>182,746 (80.1%)<br>45,672<br>1.13 (0.45)<br>1.04 (0.45)<br>182,344 (80.0%) | 52.40 (1978.94)<br>#VALUEI<br>13,332 (75.6%)<br>4,414<br>1.23 (0.53)<br>1.13 (0.53)<br>13,226 (75.0%) | #VALUE!<br>0.11<br>-0.20<br>-0.18<br>0.12 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)mean (sd) | 39,671<br>20.56 (9.20)<br>18.50 [14.50, 24.00]<br>74,320 (65.2%)<br>40,229<br>1.14 (0.45)<br>1.04 [0.85, 1.32]<br>73,762 (64.7%)<br>31,938<br>46.04 [13.96)<br>44.00 [37.00, 53.00] | 3,848 22.06 (10.35) 19.67 [15.00, 27.00] 5,056 (56.8%) 3,945 1.24 (0.52) 1.14 [0.88, 1.48] 4,959 (55.7%) 3,092 46.52 [14.16) 44.50 [37.00, 54.00] | 5,599 782.69 (11,615.02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] 108,582 (95.2%) 6,157 43.97 (14.10) | 460<br>306.16 (6,060.48)<br>18.25 [14.00, 25.88]<br>8,276 (94.7%)<br>469<br>1.18 (0.61)<br>1.02 [0.84, 1.35]<br>8,267 (94.6%)<br>397<br>51.75 (174.25)<br>41.00 [34.00, 52.00] | N/A | N/A | 45,270<br>114.82 (4084.57)<br>#VALUE!<br>182,746 (80.1%)<br>45,672<br>1.13 (0.45)<br>1.04 (0.45)<br>182,344 (80.0%)<br>38,095<br>45,71 (13.98)<br>43.84 (13.98) | 52.40 (1978.94) #VALUEI 13,332 (75.6%) 4,414 1.23 (0.53) 1.13 (0.53) 13,226 (75.0%) 3,489 47.12 (60.22) 44.10 (60.22) | #VALUE!<br>0.11<br>-0.20<br>-0.18<br>0.12 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [lQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [lQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)mean (sd)mean (sd)mean (sd)mean (sd)mean (sd)median [lQR]Missing; n (%) | 39,671<br>20.56 (9.20)<br>18.50 [14.50, 24.00]<br>74,320 (65.2%)<br>40,229<br>1.14 (0.45)<br>1.04 [0.85, 1.32]<br>73,762 (64.7%)<br>31,938<br>46.04 (13.96) | 3,848 22.06 (10.35) 19.67 [15.00, 27.00] 5,056 (56.8%) 3,945 1.24 (0.52) 1.14 [0.88, 1.48] 4,959 (55.7%) 3,092 46.52 (14.16) | 5,599 782.69 (11,615.02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] 108,582 (95.2%) 6,157 43.97 (14.10) 43.00 [36.00, 51.00] | 460<br>306.16 (6,060.48)<br>18.25 [14.00, 25.88]<br>8,276 (94.7%)<br>469<br>1.18 (0.61)<br>1.02 [0.84, 1.35]<br>8,267 (94.6%)<br>397<br>51.75 (174.25) | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A | 45,270<br>114.82 (4084.57)<br>#VALUE!<br>182,746 (80.1%)<br>45,672<br>1.13 (0.45)<br>1.04 (0.45)<br>182,344 (80.0%)<br>38,095<br>45,71 (13.98) | 52.40 (1978.94) #WALUE! 13,332 (75.6%) 4,414 1.23 (0.53) 1.13 (0.53) 13,226 (75.0%) 3,489 47.12 (60.22) | #VALUEI 0.11 -0.20 -0.18 0.12 -0.03 -0.01 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included) | 39,671<br>20,56 (9,20)<br>18.50 [14.50, 24.00]<br>74,320 (65.2%)<br>40,229<br>1.14 (0.45)<br>1.04 [0.85, 1.32]<br>73,762 (64.7%)<br>31,938<br>46.04 (13.96)<br>44.00 [37.00, 53.00]<br>82,053 (72.0%) | 3,848 22.06 (10.35) 19.67 [15.00, 27.00] 5,056 (56.8%) 3,945 1.24 (0.52) 1.14 [0.88, 1.48] 4,959 (55.7%) 3,092 46.52 (14.16) 44.50 [37.00, 54.00] 5,812 (65.3%) | 5,599 782.69 (11,615.02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] 108,582 (95.2%) 6,157 43.97 (14.10) 43.00 [36.00, 51.00] 107,868 (94.6%) | 460 306.16 (6,060.48) 18.25 [14.00, 25.88] 8,276 (94.7%) 469 1.18 (0.61) 1.02 [0.84, 1.35] 8,267 (94.6%) 397 51.75 (174.25) 41.00 [34.00, 52.00] 8,339 (95.5%) | N/A | N/A | 45,270 114.82 (4084.57) #WALUEI 182,746 (80.1%) 45,672 1.13 (0.45) 1.04 (0.45) 182,344 (80.0%) 38,095 45.71 (13.98) 43.84 (13.98) 189,921 (83.3%) | 52.40 (1978.94) #VALUEI 13,332 (75.6%) 4,414 1.23 (0.53) 1.13 (0.53) 13,226 (75.0%) 3,489 47.12 (60.22) 44.10 (60.22) 14,151 (80.2%) | #VALUEI 0.11 -0.20 -0.18 0.12 -0.03 -0.01 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)median [iQR]median [iQR]median [iQR]median [iQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included) | 39,671<br>20.56 (9.20)<br>18.50 [14.50, 24.00]<br>74,320 (65.2%)<br>40,229<br>1.14 (0.45)<br>1.04 (0.85, 1.32]<br>73,762 (64.7%)<br>31,938<br>46.04 (13.96)<br>44.00 [37.00, 53.00]<br>82,053 (72.0%) | 3,848 22.06 (10.35) 19.67 [15.00, 27.00] 5,056 (56.8%) 3,945 1.24 (0.52) 1.14 [0.88, 1.48] 4,959 (55.7%) 3,092 46.52 [14.16) 44.50 [37.00, 54.00] 5,812 (65.3%) 3,111 | 5,599 782.69 (11,615.02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] 108,582 (95.2%) 6,157 43.97 (14.10) 43.00 [36.00, 51.00] 107,868 (94.6%) 5,964 | 460<br>306.16 (6,060.48)<br>18.25 [14.00, 25.88]<br>8,276 (94.7%)<br>469<br>1.18 (0.61)<br>1.02 [0.84, 1.35]<br>8,267 (94.6%)<br>397<br>51.75 (174.25)<br>41.00 [34.00, 52.00]<br>8,339 (95.5%) | N/A | N/A | 45,270 114.82 (4084.57) #VALUE! 182,746 (80.1%) 45,672 1.13 (0.45) 1.04 (0.45) 182,344 (80.0%) 38,095 45.71 (13.98) 43.84 (13.98) 189,921 (83.3%) | 52.40 (1978.94) #VALUEI 13,332 (75.6%) 4,414 1.23 (0.53) 1.13 (0.53) 13,226 (75.0%) 3,489 47.12 (60.22) 44.10 (60.22) 14,151 (80.2%) | #VALUEI 0.11 -0.20 -0.18 0.12 -0.03 -0.01 0.08 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number- Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number- HDL level (mg/dl) mean (only =<5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)mean (sd) | 39,671 20.56 (9.20) 18.50 [14.50, 24.00] 74,320 (65.2%) 40,229 1.14 (0.45) 1.04 [0.85, 1.32] 73,762 (64.7%) 31,938 46.04 (13.96) 44.00 [37.00, 53.00] 82,053 (72.0%) 32,245 85.89 (40.32) | 3,848 22.06 (10.35) 19.67 [15.00, 27.00] 5,056 (56.8%) 3,945 1.24 (0.52) 1.14 [0.88, 1.48] 4,959 (55.7%) 3,092 46.52 (14.16) 44.50 [37.00, 54.00] 5,812 (65.3%) 3,111 85.56 (40.40) | 5,599 782.69 (11,615.02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] 108,582 (95.2%) 6,157 43.97 (14.10) 43.00 [36.00, 51.00] 107,868 (94.6%) 5,964 87.23 (42.41) | 460<br>306.16 (6,060.48)<br>18.25 [14.00, 25.88]<br>8,276 (94.7%)<br>469<br>1.18 (0.61)<br>1.02 [0.84, 1.35]<br>8,267 (94.6%)<br>397<br>51.75 (174.25)<br>41.00 [34.00, 52.00]<br>8,339 (95.5%)<br>377<br>85.12 (45.45) | N/A | N/A | 45,270 114.82 (4084.57) #VALUE! 182,746 (80.1%) 45,672 1.13 (0.45) 1.04 (0.45) 182,344 (80.0%) 38,095 45.71 (13.98) 43.84 (13.98) 189,921 (83.3%) 38,209 86.10 (40.65) | 52.40 (1978.94) #VALUEI 13,332 (75.6%) 4,414 1.23 (0.53) 1.13 (0.53) 13,226 (75.0%) 3,489 47.12 (60.22) 14,151 (80.2%) 3,488 85.51 (40.98) | -0.20<br>-0.18<br>0.12<br>-0.03<br>-0.01<br>-0.08 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)median [iQR]median [iQR]median [iQR]median [iQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included) | 39,671<br>20,56 (9,20)<br>18.50 [14.50, 24.00]<br>74,320 (65.2%)<br>40,229<br>1.14 (0.45)<br>1.04 [0.85, 1.32]<br>73,762 (64.7%)<br>31,938<br>46.04 (13.96)<br>44.00 [37.00, 53.00]<br>82,053 (72.0%)<br>32,245<br>85.89 (40.32)<br>82.00 [61.00, 108.00] | 3,848 22.06 (10.35) 19.67 [15.00, 27.00] 5,056 (56.8%) 3,945 1.24 (0.52) 1.14 [0.88, 1.48] 4,959 (55.7%) 3,092 46.52 [14.16) 44.50 [37.00, 54.00] 5,812 (65.3%) 3,111 | 5,599 782.69 (11,615.02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] 108,582 (95.2%) 6,157 43.97 (14.10) 43.00 [36.00, 51.00] 107,868 (94.6%) 5,964 | 460<br>306.16 (6,060.48)<br>18.25 [14.00, 25.88]<br>8,276 (94.7%)<br>469<br>1.18 (0.61)<br>1.02 [0.84, 1.35]<br>8,267 (94.6%)<br>397<br>51.75 (174.25)<br>41.00 [34.00, 52.00]<br>8,339 (95.5%) | N/A | N/A | 45,270 114.82 (4084.57) #WALUEI 182,746 (80.1%) 45,672 1.13 (0.45) 1.04 (0.45) 182,344 (80.0%) 38,095 45.71 (13.98) 43.84 (13.98) 189,921 (83.3%) 38,209 86.10 (40.65) 82.39 (40.65) | 52.40 (1978.94) #VALUEI 13,332 (75.6%) 4,414 1.23 (0.53) 1.13 (0.53) 13,226 (75.0%) 3,489 47.12 (60.22) 44.10 (60.22) 14,151 (80.2%) 3,488 85.51 (40.98) 82.77 (40.98) | #VALUEI 0.11 -0.20 -0.18 0.12 -0.03 -0.01 0.08 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number- Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number- HDL level (mg/dl) mean (only =<5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)mean (sd) | 39,671 20.56 (9.20) 18.50 [14.50, 24.00] 74,320 (65.2%) 40,229 1.14 (0.45) 1.04 [0.85, 1.32] 73,762 (64.7%) 31,938 46.04 (13.96) 44.00 [37.00, 53.00] 82,053 (72.0%) 32,245 85.89 (40.32) | 3,848 22.06 (10.35) 19.67 [15.00, 27.00] 5,056 (56.8%) 3,945 1.24 (0.52) 1.14 [0.88, 1.48] 4,959 (55.7%) 3,092 46.52 (14.16) 44.50 [37.00, 54.00] 5,812 (65.3%) 3,111 85.56 (40.40) | 5,599 782.69 (11,615.02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] 108,582 (95.2%) 6,157 43.97 (14.10) 43.00 [36.00, 51.00] 107,868 (94.6%) 5,964 87.23 (42.41) | 460<br>306.16 (6,060.48)<br>18.25 [14.00, 25.88]<br>8,276 (94.7%)<br>469<br>1.18 (0.61)<br>1.02 [0.84, 1.35]<br>8,267 (94.6%)<br>397<br>51.75 (174.25)<br>41.00 [34.00, 52.00]<br>8,339 (95.5%)<br>377<br>85.12 (45.45) | N/A | N/A | 45,270 114.82 (4084.57) #VALUE! 182,746 (80.1%) 45,672 1.13 (0.45) 1.04 (0.45) 182,344 (80.0%) 38,095 45.71 (13.98) 43.84 (13.98) 189,921 (83.3%) 38,209 86.10 (40.65) | 52.40 (1978.94) #VALUEI 13,332 (75.6%) 4,414 1.23 (0.53) 1.13 (0.53) 13,226 (75.0%) 3,489 47.12 (60.22) 14,151 (80.2%) 3,488 85.51 (40.98) | -0.20<br>-0.18<br>0.12<br>-0.03<br>-0.01<br>-0.08 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)mean (sd)mean (sd)meaian [IQR] | 39,671<br>20,56 (9,20)<br>18.50 [14.50, 24.00]<br>74,320 (65.2%)<br>40,229<br>1.14 (0.45)<br>1.04 [0.85, 1.32]<br>73,762 (64.7%)<br>31,938<br>46.04 (13.96)<br>44.00 [37.00, 53.00]<br>82,053 (72.0%)<br>32,245<br>85.89 (40.32)<br>82.00 [61.00, 108.00] | 3,848 22.06 (10.35) 19.67 [15.00, 27.00] 5,056 (56.8%) 3,945 1.24 (0.52) 1.14 [0.88, 1.48] 4,959 (55.7%) 3,092 46.52 (14.16) 44.50 [37.00, 54.00] 5,812 (65.3%) 3,111 85.56 (40.40) 82.50 [61.00, 109.00] | 782.69 (11,615.02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] 108,582 (95.2%) 6,157 43.97 (14.10) 43.00 [36.00, 51.00] 107,868 (94.6%) 5,964 87.23 (42.41) 84,50 [63.00, 111.00] | 460 306.16 (6,060.48) 18.25 [14.00, 25.88] 8,276 (94.7%) 469 1.18 (0.61) 1.02 [0.84, 1.35] 8,267 (94.6%) 397 51.75 [174.25) 41.00 [34.00, 52.00] 8,339 (95.5%) 377 85.12 (45.45) 85.00 [59.00, 111.25] | N/A | N/A | 45,270 114.82 (4084.57) #WALUEI 182,746 (80.1%) 45,672 1.13 (0.45) 1.04 (0.45) 182,344 (80.0%) 38,095 45.71 (13.98) 43.84 (13.98) 189,921 (83.3%) 38,209 86.10 (40.65) 82.39 (40.65) | 52.40 (1978.94) #VALUEI 13,332 (75.6%) 4,414 1.23 (0.53) 1.13 (0.53) 13,226 (75.0%) 3,489 47.12 (60.22) 44.10 (60.22) 14,151 (80.2%) 3,488 85.51 (40.98) 82.77 (40.98) | #VALUEI 0.11 -0.20 -0.18 0.12 -0.03 -0.01 0.08 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only | 39,671 20.56 (9.20) 18.50 [14.50, 24.00] 74,320 (65.2%) 40,229 1.14 (0.45) 1.04 (0.85, 1.32] 73,762 (64.7%) 31,938 46.04 (13.96) 44.00 [37.00, 53.00] 82,053 (72.0%) 32,245 85.89 (40.32) 82.00 [61.00, 108.00] 81,746 (71.7%) | 3,848 22.06 (10.35) 19.67 [15.00, 27.00] 5,056 (56.8%) 3,945 1.24 (0.52) 1.14 [0.88, 1.48] 4,959 (55.7%) 3,092 46.52 [14.16) 44.50 [37.00, 54.00] 5,812 (65.3%) 3,111 85.56 (40.40) 82.50 [61.00, 109.00] 5,793 (65.1%) | 5,599 782.69 (11,615.02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] 108,582 (95.2%) 6,157 43.97 (14.10) 43.00 [36.00, 51.00] 107,868 (94.6%) 5,964 87.23 (42.41) 84.50 [63.00, 111.00] 108,061 (94.8%) | 460 306.16 (6,060.48) 18.25 [14.00, 25.88] 8,276 (94.7%) 469 1.18 (0.61) 1.02 [0.84, 1.35] 8,267 (94.6%) 397 51.75 (174.25) 41.00 [34.00, 52.00] 8,339 (95.5%) 377 85.12 (45.45) 85.00 [59.00, 111.25] 8,359 (95.7%) | N/A | N/A | 45,270 114.82 (4084.57) #VALUE! 182,746 (80.1%) 45,672 1.13 (0.45) 1.04 (0.45) 182,344 (80.0%) 38,095 45.71 (13.98) 43.84 (13.98) 189,921 (83.3%) 38,209 86.10 (40.65) 82.39 (40.65) 189,807 (83.2%) | 52.40 (1978.94) #VALUEI 13,332 (75.6%) 4,414 1.23 (0.53) 1.13 (0.53) 13,226 (75.0%) 3,489 47.12 (60.22) 44.10 (60.22) 14,151 (80.2%) 3,488 85.51 (40.98) 82.77 (40.98) 14,152 (80.2%) | #VALUEI 0.11 -0.20 -0.18 0.12 -0.03 -0.01 0.08 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only =<5000 included) | 39,671<br>20,56 (9,20)<br>18.50 [14.50, 24.00]<br>74,320 (65.2%)<br>40,229<br>1.14 (0.45)<br>1.04 [0.85, 1.32]<br>73,762 (64.7%)<br>31,938<br>46.04 (13.96)<br>44.00 [37.00, 53.00]<br>82,053 (72.0%)<br>32,245<br>85.89 (40.32)<br>82.00 [61.00, 108.00]<br>81,746 (71.7%) | 3,848 22.06 (10.35) 19.67 [15.00, 27.00] 5,056 (56.8%) 3,945 1.24 (0.52) 1.14 [0.88, 1.48] 4,959 (55.7%) 3,092 46.52 (14.16) 44.50 [37.00, 54.00] 5,812 (65.3%) 3,111 85.56 (40.40) 82.50 [61.00, 109.00] 5,793 (65.1%) | 78.269 (11,61,02) 782.69 (11,61,02) 17.00 [13.50,22.00) 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] 108,582 (95.2%) 6,157 43.97 (14.10) 43.00 [36.00, 51.00] 107,868 (94.6%) 5,964 87.23 (42.41) 84.50 [63.00, 111.00] 108,061 (94.8%) | 460 306.16 (6,060.48) 18.25 [14.00, 25.88] 8,276 [94.7%) 469 1.18 (0.61) 1.02 [0.84, 1.35] 8,267 (94.6%) 397 51.75 [174.25) 41.00 [34.00, 52.00] 8,339 (95.5%) 377 85.12 (45.45) 85.00 [59.00, 111.25] 8,359 (95.7%) | N/A | N/A | 45,270 114.82 (4084.57) #VALUEI 182,746 (80.1%) 45,672 1.13 (0.45) 1.04 (0.45) 182,344 (80.0%) 38,095 45.71 (13.98) 43.84 (13.98) 189,921 (83.3%) 38,209 86.10 (40.65) 82.39 (40.65) 189,807 (83.2%) | 52.40 (1978.94) #VALUEI 13,332 (75.6%) 4,414 1.23 (0.53) 1.13 (0.53) 13,226 (75.0%) 3,489 47.12 (60.22) 14,151 (80.2%) 3,488 85.51 (40.98) 82.77 (40.98) 14,152 (80.2%) | -0.20<br>-0.18<br>-0.12<br>-0.03<br>-0.01<br>-0.08<br>-0.01<br>-0.01<br>-0.01 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only | 39,671 20.56 (9.20) 18.50 [14.50, 24.00] 74,320 (65.2%) 40,229 1.14 (0.45) 1.04 (0.85, 1.32] 73,762 (64.7%) 31,938 46.04 (13.96) 44.00 [37.00, 53.00] 82,053 (72.0%) 32,245 85.89 (40.32) 82.00 [61.00, 108.00] 81,746 (71.7%) | 3,848 22.06 (10.35) 19.67 [15.00, 27.00] 5,056 (56.8%) 3,945 1.24 (0.52) 1.14 [0.88, 1.48] 4,959 (55.7%) 3,092 46.52 [14.16) 44.50 [37.00, 54.00] 5,812 (65.3%) 3,111 85.56 (40.40) 82.50 [61.00, 109.00] 5,793 (65.1%) | 5,599 782.69 (11,615.02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] 108,582 (95.2%) 6,157 43.97 (14.10) 43.00 [36.00, 51.00] 107,868 (94.6%) 5,964 87.23 (42.41) 84.50 [63.00, 111.00] 108,061 (94.8%) | 460 306.16 (6,060.48) 18.25 [14.00, 25.88] 8,276 (94.7%) 469 1.18 (0.61) 1.02 [0.84, 1.35] 8,267 (94.6%) 397 51.75 (174.25) 41.00 [34.00, 52.00] 8,339 (95.5%) 377 85.12 (45.45) 85.00 [59.00, 111.25] 8,359 (95.7%) | N/A | N/A | 45,270 114.82 (4084.57) #VALUE! 182,746 (80.1%) 45,672 1.13 (0.45) 1.04 (0.45) 182,344 (80.0%) 38,095 45.71 (13.98) 43.84 (13.98) 189,921 (83.3%) 38,209 86.10 (40.65) 82.39 (40.65) 189,807 (83.2%) | 52.40 (1978.94) #VALUEI 13,332 (75.6%) 4,414 1.23 (0.53) 1.13 (0.53) 13,226 (75.0%) 3,489 47.12 (60.22) 44.10 (60.22) 14,151 (80.2%) 3,488 85.51 (40.98) 82.77 (40.98) 14,152 (80.2%) | #VALUEI 0.11 -0.20 -0.18 0.12 -0.03 -0.01 0.08 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only =<5000 included) | 39,671<br>20,56 (9,20)<br>18.50 [14.50, 24.00]<br>74,320 (65.2%)<br>40,229<br>1.14 (0.45)<br>1.04 [0.85, 1.32]<br>73,762 (64.7%)<br>31,938<br>46.04 (13.96)<br>44.00 [37.00, 53.00]<br>82,053 (72.0%)<br>32,245<br>85.89 (40.32)<br>82.00 [61.00, 108.00]<br>81,746 (71.7%) | 3,848 22.06 (10.35) 19.67 [15.00, 27.00] 5,056 (56.8%) 3,945 1.24 (0.52) 1.14 [0.88, 1.48] 4,959 (55.7%) 3,092 46.52 (14.16) 44.50 [37.00, 54.00] 5,812 (65.3%) 3,111 85.56 (40.40) 82.50 [61.00, 109.00] 5,793 (65.1%) | 78.269 (11,61,02) 782.69 (11,61,02) 17.00 [13.50,22.00) 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] 108,582 (95.2%) 6,157 43.97 (14.10) 43.00 [36.00, 51.00] 107,868 (94.6%) 5,964 87.23 (42.41) 84.50 [63.00, 111.00] 108,061 (94.8%) | 460 306.16 (6,060.48) 18.25 [14.00, 25.88] 8,276 [94.7%) 469 1.18 (0.61) 1.02 [0.84, 1.35] 8,267 (94.6%) 397 51.75 [174.25) 41.00 [34.00, 52.00] 8,339 (95.5%) 377 85.12 (45.45) 85.00 [59.00, 111.25] 8,359 (95.7%) | N/A | N/A | 45,270 114.82 (4084.57) #VALUEI 182,746 (80.1%) 45,672 1.13 (0.45) 1.04 (0.45) 182,344 (80.0%) 38,095 45.71 (13.98) 43.84 (13.98) 189,921 (83.3%) 38,209 86.10 (40.65) 82.39 (40.65) 189,807 (83.2%) | 52.40 (1978.94) #VALUEI 13,332 (75.6%) 4,414 1.23 (0.53) 1.13 (0.53) 13,226 (75.0%) 3,489 47.12 (60.22) 14,151 (80.2%) 3,488 85.51 (40.98) 82.77 (40.98) 14,152 (80.2%) | -0.20<br>-0.18<br>-0.12<br>-0.03<br>-0.01<br>-0.08<br>-0.01<br>-0.01<br>-0.01 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only =<5000 included)mean (sd)mean (sd)mean (sd) | 39,671 20.56 (9.20) 18.50 [14.50, 24.00] 74,320 (65.2%) 40,229 1.14 (0.45) 1.04 [0.85, 1.32] 73,762 (64.7%) 31,938 46.04 (13.96) 44.00 [37.00, 53.00] 82,053 (72.0%) 32,245 85.89 (40.32) 82.00 [61.00, 108.00] 81,746 (71.7%) 32,317 172.24 (48.74) 165.50 [140.00, 197.00] | 3,848 22.06 (10.35) 19.67 [15.00, 27.00] 5,056 (56.8%) 3,945 1.24 (0.52) 1.14 [0.88, 1.48] 4,959 (55.7%) 46.52 (14.16) 44.50 [37.00, 54.00] 5,812 (65.3%) 3,111 85.56 (40.40) 82.50 [61.00, 109.00] 5,793 (65.1%) 3,153 173.80 (47.85) 166.00 [142.00, 197.50] | 782.69 (11.61.02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 (0.82, 1.21] 108,582 (95.2%) 6,157 43.97 (14.10) 43.00 [36.00, 51.00] 107,868 (94.6%) 5,964 87.23 (42.41) 84.50 [63.00, 111.00] 108,061 (94.8%) 6,112 173.02 (52.38) 168.00 [142.00, 200.00] | 460 306.16 (6,060.48) 18.25 [14.00, 25.88] 8,276 (94.7%) 469 1.18 (0.61) 1.02 [0.84, 1.35] 8,267 (94.6%) 397 51.75 (174.25) 41.00 [34.00, 52.00] 8,339 (95.5%) 377 85.12 (45.45) 85.00 [59.00, 111.25] 8,359 (95.7%) 403 174.06 (57.08) 170.00 [141.00, 205.00] | N/A | N/A | 45,270 114.82 (4084.57) #WALUE! 182,746 (80.1%) 45,672 1.13 (0.45) 1.04 (0.45) 182,344 (80.0%) 38,095 45.71 (13.98) 43.84 (13.98) 189,921 (83.3%) 38,209 86.10 (40.65) 82.39 (40.65) 189,807 (83.2%) 38,429 172.36 (49.34) 165.90 (49.34) | 52.40 (1978.94) #VALUEI 13,332 (75.6%) 4,414 1.23 (0.53) 1.13 (0.53) 13,226 (75.0%) 3,489 47.12 (60.22) 44.10 (60.22) 14,151 (80.2%) 3,488 85.51 (40.98) 82.77 (40.98) 14,152 (80.2%) 3,556 173.83 (48.99) 166.45 (48.99) | #VALUEI 0.11 -0.20 -0.18 0.12 -0.03 -0.01 0.08 0.01 -0.01 0.08 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) | 39,671 20.56 (9.20) 18.50 [14.50, 24.00] 74,320 (65.2%) 40,229 1.14 (0.45) 1.04 [0.85, 1.32] 73,762 (64.7%) 31,938 46.04 (13.96) 44.00 [37.00, 53.00] 82,053 (72.0%) 32,245 85.89 (40.32) 82.00 [61.00, 108.00] 81,746 (71.7%) 32,317 172.24 (48.74) | 3,848 22.06 (10.35) 19.67 [15.00, 27.00] 5,056 (56.8%) 3,945 1.24 (0.52) 1.14 [0.88, 1.48] 4,959 (55.7%) 3,092 46.52 (14.16) 44.50 [37.00, 54.00] 5,812 (65.3%) 3,111 85.56 (40.40) 82.50 [61.00, 109.00] 5,793 (65.1%) 3,153 173.80 (47.85) | 782.69 (11.61.02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] 108,582 (95.2%) 6,157 43.97 (14.10) 43.00 [36.00, 51.00] 107,868 (94.6%) 5,964 87.23 (42.41) 84.50 [63.00, 111.00] 108,061 (94.8%) 6,112 173.02 (52.38) | 460 306.16 (6,060.48) 18.25 [14.00, 25.88] 8,276 (94.7%) 469 1.18 (0.61) 1.02 [0.84, 1.35] 8,267 (94.6%) 397 51.75 (174.25) 41.00 [34.00, 52.00] 8,339 (95.5%) 377 85.12 (45.45) 85.00 [59.00, 111.25] 8,359 (95.7%) 403 174.06 (57.08) | N/A | N/A | 45,270 114.82 (4084.57) #WALUEI 182,746 (80.1%) 45,672 1.13 (0.45) 1.04 (0.45) 182,344 (80.0%) 38,095 45.71 (13.98) 43.84 (13.98) 189,921 (83.3%) 38,209 86.10 (40.65) 189,807 (83.2%) 38,429 172.36 (49.34) | 52.40 (1978.94) #VALUEI 13,332 (75.6%) 4,414 1.23 (0.53) 1.13 (0.53) 13,226 (75.0%) 3,489 47.12 (60.22) 44.10 (60.22) 14,151 (80.2%) 3,488 85.51 (40.98) 82.77 (40.98) 14,152 (80.2%) 3,556 173.83 (48.99) | #VALUEI 0.11 -0.20 -0.18 0.12 -0.03 -0.01 -0.01 -0.08 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-TDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]median [IQR]median [IQR]median [IQR]median [IQR] | 39,671 20,56 (9,20) 18.50 [14.50, 24.00] 74,320 (65.2%) 40,229 1.14 (0.45) 1.04 [0.85, 1.32] 73,762 (64.7%) 31,938 46.04 (13.96) 44.00 [37.00, 53.00] 82,053 (72.0%) 32,245 85.89 (40.32) 82.00 [61.00, 108.00] 81,746 (71.7%) 32,317 172.24 (48.74) 165.50 [140.00, 197.00] 81,674 (71.6%) | 3,848 22.06 (10.35) 19.67 [15.00, 27.00] 5,056 (56.8%) 3,945 1.24 (0.52) 1.14 [0.88, 1.48] 4,959 (55.7%) 3,092 46.52 [14.16) 44.50 [37.00, 54.00] 5,812 (65.3%) 3,111 85.56 (40.40) 82.50 [61.00, 109.00] 5,793 (65.1%) 3,153 173.80 (47.85) 166.00 [142.00, 197.50] 5,751 (64.6%) | 78.269 (11,615,02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] 108,582 (95.2%) 6,157 43.97 (14.10) 43.00 [36.00, 51.00] 107,868 (94.6%) 5,964 87.23 (42.41) 84.50 [63.00, 111.00] 108,061 (94.8%) 6,112 173.02 (52.38) 168.00 [142.00, 200.00] 107,913 (94.6%) | 460 306.16 (6,060.48) 18.25 [14.00, 25.88] 8,276 [94.7%) 469 1.18 (0.61) 1.02 [0.84, 1.35] 8,267 (94.6%) 397 51.75 [174.25) 41.00 [34.00, 52.00] 8,339 (95.5%) 377 85.12 (45.45) 85.00 [59.00, 111.25] 8,359 (95.7%) 403 174.06 (57.08) 170.00 [141.00, 205.00] 8,333 (95.4%) | N/A | N/A | 45,270 114.82 (4084.57) #WALUEI 182,746 (80.1%) 45,672 1.13 (0.45) 1.04 (0.45) 182,344 (80.0%) 38,095 45.71 (13.98) 43.84 (13.98) 189,921 (83.3%) 38,209 86.10 (40.65) 82.39 (40.65) 189,807 (83.2%) 38,429 172.36 (49.34) 165.90 (49.34) 189,587 (83.1%) | 52.40 (1978.94) #VALUEI 13,332 (75.6%) 4,414 1.23 (0.53) 1.13 (0.53) 13,226 (75.0%) 3,489 47.12 (60.22) 44.10 (60.22) 14,151 (80.2%) 3,488 85.51 (40.98) 82.77 (40.98) 14,152 (80.2%) 3,556 173.83 (48.99) 166.45 (48.99) 14,084 (79.8%) | #VALUEI 0.11 -0.20 -0.18 0.12 -0.03 -0.01 -0.01 -0.08 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Triglyceride level (mg/dl) mean (only =<5000 included) | 39,671 20.56 (9.20) 18.50 [14.50, 24.00] 74,320 (65.2%) 40,229 1.14 (0.45) 1.04 [0.85, 1.32] 73,762 (64.7%) 31,938 46.04 (13.96) 44.00 [37.00, 53.00] 82,053 (72.0%) 32,245 85.89 (40.32) 82.00 [61.00, 108.00] 81,746 (71.7%) 32,317 172.24 (48.74) 165.50 [140.00, 197.00] 81,674 (71.6%) 32,008 | 3,848 22.06 (10.35) 19.67 [15.00, 27.00] 5,056 (56.8%) 3,945 1.24 (0.52) 1.14 [0.88, 1.48] 4,959 (55.7%) 3,092 46.52 (14.16) 44.50 [37.00, 54.00] 5,812 (65.3%) 3,111 85.56 (40.40) 82.50 [61.00, 109.00] 5,793 (65.1%) 3,153 173.80 (47.85) 166.00 [142.00, 197.50] 5,751 (64.6%) | 782.69 (11.615.02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] 108,582 (95.2%) 6,157 43.97 (14.10) 43.00 [36.00, 51.00] 107,868 (94.6%) 5,964 87.23 (42.41) 84.50 [63.00, 111.00] 108,061 (94.8%) 6,112 173.02 (52.38) 168.00 [142.00, 200.00] 107,913 (94.6%) | 460 306.16 (6,060.48) 18.25 [14.00, 25.88] 8,276 [94.7%) 469 1.18 (0.61) 1.02 [0.84, 1.35] 8,267 (94.6%) 397 51.75 (174.25) 41.00 [34.00, 52.00] 8,339 (95.5%) 377 85.12 (45.45) 85.00 [59.00, 111.25] 8,359 (95.7%) 403 174.06 (57.08) 170.00 [141.00, 205.00] 8,333 (95.4%) 398 | N/A | N/A | 45,270 114.82 (4084.57) #WALUEI 182,746 (80.1%) 45,672 1.13 (0.45) 1.04 (0.45) 182,344 (80.0%) 38,095 45.71 (13.98) 43.84 (13.98) 189,921 (83.3%) 38,209 86.10 (40.65) 189,807 (83.2%) 38,429 172.36 (49.34) 165.90 (49.34) 189,587 (83.1%) | 52.40 (1978.94) #VALUEI 13,332 (75.6%) 4,414 1.23 (0.53) 1.13 (0.53) 1.13 (0.53) 13,226 (75.0%) 3,489 47.12 (60.22) 44.10 (60.22) 14,151 (80.2%) 3,488 85.51 (40.98) 82.77 (40.98) 14,152 (80.2%) 3,556 173.83 (48.99) 16.45 (48.99) 14,084 (79.8%) | #VALUEI 0.11 -0.20 -0.18 0.12 -0.03 -0.01 0.08 0.01 -0.01 0.08 -0.03 -0.01 0.08 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-TDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]median [IQR]median [IQR]median [IQR]median [IQR] | 39,671 20,56 (9,20) 18.50 [14.50, 24.00] 74,320 (65.2%) 40,229 1.14 (0.45) 1.04 [0.85, 1.32] 73,762 (64.7%) 31,938 46.04 (13.96) 44.00 [37.00, 53.00] 82,053 (72.0%) 32,245 85.89 (40.32) 82.00 [61.00, 108.00] 81,746 (71.7%) 32,317 172.24 (48.74) 165.50 [140.00, 197.00] 81,674 (71.6%) | 3,848 22.06 (10.35) 19.67 [15.00, 27.00] 5,056 (56.8%) 3,945 1.24 (0.52) 1.14 [0.88, 1.48] 4,959 (55.7%) 3,092 46.52 [14.16) 44.50 [37.00, 54.00] 5,812 (65.3%) 3,111 85.56 (40.40) 82.50 [61.00, 109.00] 5,793 (65.1%) 3,153 173.80 (47.85) 166.00 [142.00, 197.50] 5,751 (64.6%) | 78.269 (11,615,02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] 108,582 (95.2%) 6,157 43.97 (14.10) 43.00 [36.00, 51.00] 107,868 (94.6%) 5,964 87.23 (42.41) 84.50 [63.00, 111.00] 108,061 (94.8%) 6,112 173.02 (52.38) 168.00 [142.00, 200.00] 107,913 (94.6%) | 460 306.16 (6,060.48) 18.25 [14.00, 25.88] 8,276 [94.7%) 469 1.18 (0.61) 1.02 [0.84, 1.35] 8,267 (94.6%) 397 51.75 [174.25) 41.00 [34.00, 52.00] 8,339 (95.5%) 377 85.12 (45.45) 85.00 [59.00, 111.25] 8,359 (95.7%) 403 174.06 (57.08) 170.00 [141.00, 205.00] 8,333 (95.4%) | N/A | N/A | 45,270 114.82 (4084.57) #WALUEI 182,746 (80.1%) 45,672 1.13 (0.45) 1.04 (0.45) 182,344 (80.0%) 38,095 45.71 (13.98) 43.84 (13.98) 189,921 (83.3%) 38,209 86.10 (40.65) 82.39 (40.65) 189,807 (83.2%) 38,429 172.36 (49.34) 165.90 (49.34) 189,587 (83.1%) | 52.40 (1978.94) #VALUEI 13,332 (75.6%) 4,414 1.23 (0.53) 1.13 (0.53) 13,226 (75.0%) 3,489 47.12 (60.22) 44.10 (60.22) 14,151 (80.2%) 3,488 85.51 (40.98) 82.77 (40.98) 14,152 (80.2%) 3,556 173.83 (48.99) 166.45 (48.99) 14,084 (79.8%) | #VALUEI 0.11 -0.20 -0.18 0.12 -0.03 -0.01 -0.01 -0.08 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Triglyceride level (mg/dl) mean (only =<5000 included) | 39,671 20.56 (9.20) 18.50 [14.50, 24.00] 74,320 (65.2%) 40,229 1.14 (0.45) 1.04 [0.85, 1.32] 73,762 (64.7%) 31,938 46.04 (13.96) 44.00 [37.00, 53.00] 82,053 (72.0%) 32,245 85.89 (40.32) 82.00 [61.00, 108.00] 81,746 (71.7%) 32,317 172.24 (48.74) 165.50 [140.00, 197.00] 81,674 (71.6%) 32,008 | 3,848 22.06 (10.35) 19.67 [15.00, 27.00] 5,056 (56.8%) 3,945 1.24 (0.52) 1.14 [0.88, 1.48] 4,959 (55.7%) 3,092 46.52 (14.16) 44.50 [37.00, 54.00] 5,812 (65.3%) 3,111 85.56 (40.40) 82.50 [61.00, 109.00] 5,793 (65.1%) 3,153 173.80 (47.85) 166.00 [142.00, 197.50] 5,751 (64.6%) | 782.69 (11.615.02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] 108,582 (95.2%) 6,157 43.97 (14.10) 43.00 [36.00, 51.00] 107,868 (94.6%) 5,964 87.23 (42.41) 84.50 [63.00, 111.00] 108,061 (94.8%) 6,112 173.02 (52.38) 168.00 [142.00, 200.00] 107,913 (94.6%) | 460 306.16 (6,060.48) 18.25 [14.00, 25.88] 8,276 [94.7%) 469 1.18 (0.61) 1.02 [0.84, 1.35] 8,267 (94.6%) 397 51.75 (174.25) 41.00 [34.00, 52.00] 8,339 (95.5%) 377 85.12 (45.45) 85.00 [59.00, 111.25] 8,359 (95.7%) 403 174.06 (57.08) 170.00 [141.00, 205.00] 8,333 (95.4%) 398 | N/A | N/A | 45,270 114.82 (4084.57) #WALUEI 182,746 (80.1%) 45,672 1.13 (0.45) 1.04 (0.45) 182,344 (80.0%) 38,095 45.71 (13.98) 43.84 (13.98) 189,921 (83.3%) 38,209 86.10 (40.65) 189,807 (83.2%) 38,429 172.36 (49.34) 165.90 (49.34) 189,587 (83.1%) | 52.40 (1978.94) #VALUEI 13,332 (75.6%) 4,414 1.23 (0.53) 1.13 (0.53) 1.13 (0.53) 13,226 (75.0%) 3,489 47.12 (60.22) 44.10 (60.22) 14,151 (80.2%) 3,488 85.51 (40.98) 82.77 (40.98) 14,152 (80.2%) 3,556 173.83 (48.99) 16.45 (48.99) 14,084 (79.8%) | #VALUEI 0.11 -0.20 -0.18 0.12 -0.03 -0.01 0.08 0.01 -0.01 0.08 -0.03 -0.01 0.08 |
| Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only =<5000 included)mean (sd)mean (sd)mean (sd)mean (sd)mean (sd)mean (sd)mean (sd)median [IQR]Missing; n (%) Lab result number-Triglyceride level (mg/dl) mean (only =<5000 included)men (sd) | 39,671 20.56 (9.20) 18.50 [14.50, 24.00] 74,320 (65.2%) 40,229 1.14 (0.45) 1.04 [0.85, 1.32] 73,762 (64.7%) 31,938 46.04 (13.96) 44.00 [37.00, 53.00] 82,053 (72.0%) 32,245 85.89 (40.32) 82.00 [61.00, 108.00] 81,746 (71.7%) 32,317 172.24 (48.74) 165.50 [140.00, 197.00] 81,674 (71.6%) 32,008 185.40 (155.50) | 3,848 22.06 (10.35) 19.67 [15.00, 27.00] 5,056 (56.8%) 3,945 1.24 (0.52) 1.14 [0.88, 1.48] 4,959 (55.7%) 46.52 (14.16) 44.50 [37.00, 54.00] 5,812 (65.3%) 3,111 85.56 (40.40) 82.50 [61.00, 109.00] 5,793 (65.1%) 3,153 173.80 (47.85) 166.00 [142.00, 197.50] 5,751 (64.6%) 3,140 189.62 (172.91) | 78.269 (11,615,02) 17.00 [13.50, 22.00] 108,426 (95.1%) 5,443 1.09 (0.46) 1.00 [0.82, 1.21] 108,582 (95.2%) 6,157 43.97 (14.10) 43.00 [36.00, 51.00] 107,868 (94.6%) 5,964 87.23 (42.41) 84.50 [63.00, 111.00] 108,061 (94.8%) 6,112 173.02 (52.38) 168.00 [142.00, 200.00] 107,913 (94.6%) 5,996 193.09 (188.17) | 460 306.16 (6,060.48) 18.25 [14.00, 25.88] 8,276 (94.7%) 469 1.18 (0.61) 1.02 [0.84, 1.35] 8,267 (94.6%) 397 51.75 (174.25) 41.00 [34.00, 52.00] 8,339 (95.5%) 377 85.12 (45.45) 85.00 [59.00, 111.25] 8,359 (95.7%) 403 174.06 (57.08) 170.00 [141.00, 205.00] 8,333 (95.4%) 398 212.32 (232.65) | N/A | N/A | 45,270 114.82 (4084.57) #WALUE! 182,746 (80.1%) 45,672 1.13 (0.45) 1.04 (0.45) 182,344 (80.0%) 38,095 45.71 (13.98) 43.84 (13.98) 189,921 (83.3%) 38,209 86.10 (40.65) 82.39 (40.65) 82.39 (40.65) 189,807 (83.2%) 38,429 172.36 (49.34) 165.90 (49.34) 189,587 (83.1%) 38,004 186.61 (161.10) | 52.40 (1978.94) #VALUEI 13,332 (75.6%) 4,414 1.23 (0.53) 1.13 (0.53) 13,226 (75.0%) 3,489 47.12 (60.22) 44.10 (60.22) 14,151 (80.2%) 3,488 85.51 (40.98) 82.77 (40.98) 14,152 (80.2%) 3,556 173.83 (48.99) 14,084 (79.8%) 3,538 192.17 (180.63) | **VALUEI 0.11 -0.20 -0.18 0.12 -0.03 -0.01 -0.08 -0.03 -0.01 -0.08 -0.03 -0.01 -0.08 |

| Lab annula arraban Harrandahia anna (antro Oinglordad) | 28,631 | 2.000 | 2.766 | 252 | N1/A | N1/A | 32,397 | 2.262 | |
|---|---|---|---|---|---|---|---|---|---|
| Lab result number- Hemoglobin mean (only >0 included)mean (sd) | 13.29 (1.75) | 2,909<br>13.17 (1.73) | 3,766<br>6,103.13 (230,642.43) | 353<br>443.69 (8,089.45) | N/A<br>N/A | N/A<br>N/A | 721.21 (78630.20) | 3,262<br>59.76 (2658.57) | 0.01 |
| median [IQR] | 13.30 [12.10, 14.50] | 13.20 [11.95, 14.40] | 13.60 [12.30, 14.75] | 13.30 [12.00, 14.53] | N/A<br>N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Missing; n (%) | 85,360 (74.9%) | 5,995 (67.3%) | 110,259 (96.7%) | 8,383 (96.0%) | N/A<br>N/A | N/A | 195,619 (85.8%) | 14,378 (81.5%) | 0.12 |
| | 65,560 (74.9%) | 3,993 (07.3%) | 110,239 (90.7%) | 0,303 (90.0%) | N/A | IN/A | 193,019 (03.0%) | 14,576 (61.5%) | 0.12 |
| Lab result number- Serum sodium mean (only > 90 and < 190 included) | 39,251 | 3,841 | 5,097 | 458 | N/A | N/A | 44,348 | 4,299 | |
| mean (sd) | 139.42 (2.88) | 139.59 (2.83) | 138.84 (2.83) | 139.10 (2.65) | N/A | N/A | 139.35 (2.87) | 139.54 (2.81) | -0.07 |
| median [IQR] | 139.75 [138.00, 141.00] | 140.00 [138.00, 141.50] | 139.00 [137.00, 141.00] | 139.37 [137.00, 141.00] | N/A | N/A | 139.66 (2.87) | 139.93 (2.81) | -0.10 |
| Missing; n (%) | 74,740 (65.6%) | 5,063 (56.9%) | 108,928 (95.5%) | 8,278 (94.8%) | N/A | N/A | 183,668 (80.6%) | 13,341 (75.6%) | 0.12 |
| Lab result number- Albumin mean (only >0 and <=10 | 74,740 (03.070) | 3,003 (30.3%) | 108,328 (33.376) | 8,278 (34.878) | N/A | IN/A | 183,008 (80.0%) | 13,341 (73.070) | 0.12 |
| included) | 36.154 | 3,614 | 4.374 | 398 | N/A | N/A | 40,528 | 4,012 | |
| mean (sd) | 4.21 (0.33) | 4.21 (0.36) | 4.12 (0.64) | 4.09 (0.71) | N/A | N/A | 4.20 (0.38) | 4.20 (0.41) | 0.00 |
| median [IQR] | 4.20 [4.00, 4.40] | 4.20 [4.00, 4.45] | 4.20 [4.00, 4.40] | 4.20 [4.00, 4.40] | N/A | N/A | 4.20 (0.38) | 4.20 (0.41) | 0.00 |
| Missing; n (%) | 77,837 (68.3%) | 5,290 (59.4%) | 109,651 (96.2%) | 8,338 (95.4%) | N/A | N/A | 187,488 (82.2%) | 13,628 (77.3%) | 0.12 |
| Lab result number- Glucose (fasting or random) mean | 77,037 (00.370) | 3,230 (33.170) | 103,031 (30.270) | 0,550 (55.170) | .,,,, | .,,,, | 107,100 (02.270) | 13,020 (77.370) | 0.12 |
| (only 10-1000 included) | 39.051 | 3.838 | 4.988 | 457 | N/A | N/A | 44.039 | 4,295 | |
| mean (sd) | 168.55 (73.40) | 164.67 (71.92) | 177.16 (79.94) | 166.24 (76.35) | N/A | N/A | 169.53 (74.17) | 164.84 (72.41) | 0.06 |
| median [IQR] | 150.00 [121.00, 195.00] | 146.00 [118.50, 187.00] | 156.00 [124.00, 208.00] | 145.00 [120.92, 188.00] | N/A | N/A | 150.68 (74.17) | 145.89 (72.41) | 0.07 |
| Missing; n (%) | 74,940 (65.7%) | 5,066 (56.9%) | 109,037 (95.6%) | 8,279 (94.8%) | N/A | N/A | 183,977 (80.7%) | 13,345 (75.7%) | 0.12 |
| | , (,-, | 2,222 (22.27.2) | | -,= () | | | | | |
| Lab result number- Potassium mean (only 1-7 included) | 40,186 | 3,936 | 5,475 | 450 | N/A | N/A | 45,661 | 4,386 | |
| mean (sd) | 4.47 (0.45) | 4.49 (0.46) | 4.35 (0.46) | 4.36 (0.50) | N/A | N/A | 4.46 (0.45) | 4.48 (0.46) | -0.04 |
| median [IQR] | 4.45 [4.20, 4.75] | 4.50 [4.20, 4.80] | 4.32 [4.00, 4.60] | 4.38 [4.07, 4.70] | N/A | N/A | 4.43 (0.45) | 4.49 (0.46) | -0.13 |
| Missing; n (%) | 73,805 (64.7%) | 4,968 (55.8%) | 108,550 (95.2%) | 8,286 (94.8%) | N/A | N/A | 182,355 (80.0%) | 13,254 (75.1%) | 0.12 |
| Comorbidity Scores | | | | | | | | | |
| CCI (180 days)- ICD9 and ICD10 | | | | | | | | | |
| mean (sd) | 2.99 (2.02) | 3.36 (2.10) | 2.08 (1.78) | 2.46 (1.86) | 3.19 (2.08) | 3.77 (2.11) | 2.94 (2.01) | 3.47 (2.07) | -0.26 |
| median [IQR] | 3.00 [1.00, 4.00] | 3.00 [2.00, 5.00] | 2.00 [1.00, 3.00] | 2.00 [1.00, 4.00] | 3.00 [2.00, 4.00] | 4.00 [2.00, 5.00] | 2.81 (2.01) | 3.48 (2.07) | -0.33 |
| Frailty Score: Qualitative Version 365 days as Categories, | | | | | | | | | |
| v1 | | | | | | | | | |
| 0; n (%) | 44,743 (39.3%) | 4,273 (48.0%) | 28,949 (25.4%) | 2,610 (29.9%) | 87,576 (23.9%) | 9,710 (29.1%) | 161,268 (27.1%) | 16,593 (32.5%) | -0.12 |
| 1 to 2; n (%) | 39,522 (34.7%) | 2,883 (32.4%) | 50,470 (44.3%) | 3,722 (42.6%) | 119,132 (32.5%) | 10,236 (30.6%) | 209,124 (35.2%) | 16,841 (33.0%) | 0.05 |
| 3 or more; n (%) | 29,726 (26.1%) | 1,748 (19.6%) | 34,606 (30.3%) | 2,404 (27.5%) | 159,428 (43.5%) | 13,455 (40.3%) | 223,760 (37.7%) | 17,607 (34.5%) | 0.07 |
| Facility Course Francision Marriag 200 days as Catanagian | | | | | | | | | |
| Frailty Score: Empirical Version 365 days as Categories,<0.12908; n (%) | 14,662 (12.9%) | 1,228 (13.8%) | 16,898 (14.8%) | 1,340 (15.3%) | 20,704 (5.7%) | 1,564 (4.7%) | 52,264 (8.8%) | 4,132 (8.1%) | 0.03 |
| <0.12908; n (%)<br>0.12908 - 0.1631167; n (%) | 33,703 (29.6%) | 2,522 (28.3%) | 33,908 (29.7%) | 2,586 (29.6%) | 67,558 (18.5%) | 5,402 (16.2%) | 135,169 (22.7%) | 10,510 (20.6%) | 0.03 |
| | | 5,154 (57.9%) | | | 277,874 (75.9%) | 26,435 (79.1%) | 406,719 (68.5%) | 36,399 (71.3%) | -0.06 |
| >= 0.1631167; n (%) | 65,626 (57.6%) | | 63,219 (55.4%) | 4,810 (55.1%) | | | | | 0.01 |
| Non-Frailty; n (%) | 63,097 (55.4%) | 5,173 (58.1%) | 55,924 (49.0%) | 4,718 (54.0%) | 15,747 (4.3%) | 1,403 (4.2%) | 134,768 (22.7%) | 11,294 (22.1%) | 0.01 |
| Frailty Score (mean): Qualitative Version 365 days, v1 | | | | | | | | | |
| mean (sd) | 1.68 (2.08) | 1.33 (1.90) | 1.97 (1.98) | 1.79 (1.89) | 2.57 (2.41) | 2.36 (2.39) | 2.28 (2.27) | 2.08 (2.23) | 0.09 |
| median [IQR] | 1.00 [0.00, 3.00] | 1.00 [0.00, 2.00] | 2.00 [0.00, 3.00] | 1.00 [0.00, 3.00] | | 2.00 [0.00, 4.00] | 1.81 (2.27) | 1.65 (2.23) | 0.07 |
| Frailty Score (mean): Empirical Version 365 days, | | | | | | | , , | ` ' | |
| mean (sd) | 0.18 (0.06) | 0.18 (0.06) | 0.17 (0.05) | 0.17 (0.05) | 0.21 (0.07) | 0.21 (0.07) | 0.20 (0.06) | 0.20 (0.07) | 0.00 |
| median [IQR] | 0.17 [0.14, 0.21] | 0.17 [0.14, 0.21] | 0.16 [0.14, 0.20] | 0.16 [0.14, 0.19] | 0.20 [0.16, 0.24] | 0.20 [0.17, 0.25] | 0.19 (0.06) | 0.19 (0.07) | 0.00 |
| Healthcare Utilization | | | | | | | | | |
| Any hospitalization; n (%) | 11,956 (10.5%) | 920 (10.3%) | 13,485 (11.8%) | 899 (10.3%) | 50,583 (13.8%) | 4,291 (12.8%) | 76,024 (12.8%) | 6,110 (12.0%) | 0.02 |
| Any hospitalization within prior 30 days; n (%) | 4,508 (4.0%) | 319 (3.6%) | 4,953 (4.3%) | 263 (3.0%) | 18,266 (5.0%) | 1,389 (4.2%) | 27,727 (4.7%) | 1,971 (3.9%) | 0.04 |
| Any hospitalization during prior 31-180 days; n (%) | 8,158 (7.2%) | 653 (7.3%) | 9,220 (8.1%) | 679 (7.8%) | 35,844 (9.8%) | 3,185 (9.5%) | 53,222 (9.0%) | 4,517 (8.8%) | 0.01 |
| Endocrinologist Visit; n (%) | 6,826 (6.0%) | 1,500 (16.8%) | 7,000 (6.1%) | 1,485 (17.0%) | 27,770 (7.6%) | 5,512 (16.5%) | 41,596 (7.0%) | 8,497 (16.6%) | -0.30 |
| Endocrinologist Visit (30 days prior); n (%) | 3,954 (3.5%) | 1,079 (12.1%) | 4,239 (3.7%) | 1,088 (12.5%) | 15,203 (4.2%) | 3,902 (11.7%) | 23,396 (3.9%) | 6,069 (11.9%) | -0.30 |
| Endocrinologist Visit (31 to 180 days prior); n (%) | 4,733 (4.2%) | 966 (10.8%) | 4,701 (4.1%) | 963 (11.0%) | 20,849 (5.7%) | 3,759 (11.3%) | 30,283 (5.1%) | 5,688 (11.1%) | -0.22 |
| Internal medicine/family medicine visits; n (%) | 98,689 (86.6%) | 7,064 (79.3%) | 94,269 (82.7%) | 7,569 (86.6%) | 306,858 (83.8%) | 27,861 (83.4%) | 499,816 (84.1%) | 42,494 (83.3%) | 0.02 |
| Internal medicine/family medicine visits (30 days prior); | | | | | | | | | |
| n (%) | 72,530 (63.6%) | 5,239 (58.8%) | 68,880 (60.4%) | 5,670 (64.9%) | 214,056 (58.5%) | 20,278 (60.7%) | 355,466 (59.8%) | 31,187 (61.1%) | -0.03 |
| Internal medicine/family medicine visits (31 to 180 days | | | | | | | | | |
| prior); n (%) | 85,493 (75.0%) | 6,235 (70.0%) | 79,062 (69.3%) | 6,601 (75.6%) | 268,278 (73.3%) | 25,080 (75.1%) | 432,833 (72.8%) | 37,916 (74.3%) | -0.03 |
| Cardiologist visit; n (%) | 40,644 (35.7%) | 3,396 (38.1%) | 33,564 (29.4%) | 2,878 (32.9%) | 153,453 (41.9%) | 14,288 (42.8%) | 227,661 (38.3%) | 20,562 (40.3%) | -0.04 |
| Number of Cardiologist visits (30 days prior); n (%) | 14,207 (12.5%) | 1,245 (14.0%) | 11,295 (9.9%) | 980 (11.2%) | 52,867 (14.4%) | 4,868 (14.6%) | 78,369 (13.2%) | 7,093 (13.9%) | -0.02 |
| Number of Conditional Assistant (24 to 100 do 100 d | 24 450 (20 20) | 2 800 /22 52/1 | 20.626/25.40/ | 2 400 (20 50() | 122 570 /26 22/ | 42 504 (27 70) | 105 662 (22 694) | 17.000 (25.20) | 0.65 |
| Number of Cardiologist visits (31 to 180 days prior); n (%) | 34,459 (30.2%) | 2,890 (32.5%) | 28,626 (25.1%) | 2,486 (28.5%) | 132,578 (36.2%) | 12,584 (37.7%) | 195,663 (32.9%) | 17,960 (35.2%) | -0.05 |
| Electrocardiogram ; n (%) | 39,835 (34.9%) | 3,371 (37.9%) | 39,798 (34.9%) | 3,239 (37.1%) | 142,743 (39.0%) | 13,763 (41.2%) | 222,376 (37.4%) | 20,373 (39.9%) | -0.05 |
| Use of glucose test strips; n (%) | 3,782 (3.3%) | 428 (4.8%) | 3,883 (3.4%) | 401 (4.6%) | 12,324 (3.4%) | 1,343 (4.0%) | 19,989 (3.4%) | 2,172 (4.3%) | -0.05 |
| Dialysis; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| Naive new user ; n (%) | 34,575 (30.3%) | 2,522 (28.3%) | 35,230 (30.9%) | 2,410 (27.6%) | 97,997 (26.8%) | 8,357 (25.0%) | 167,802 (28.2%) | 13,289 (26.0%) | 0.05 |

| N antidiabetic drugs at index date | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| mean (sd) | 1.67 (0.64) | 1.75 (0.68) | 1.70 (0.65) | 1.77 (0.71) | 1.66 (0.63) 1.73 (0.6 | 1.67 (0.64) | 1.74 (0.68) | -0.11 |
| median [IQR] | 2.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 2.00 [1.00, 2.00] 2.00 [1.00, 2.00 | | 2.00 (0.68) | 0.00 |
| | (,, | ,, | ,, | ,, | | | () | |
| number of different/distinct medication prescriptions | | | | | | | | |
| mean (sd) | 9.76 (4.67) | 11.09 (5.37) | 9.57 (4.62) | 10.67 (5.07) | 10.00 (4.50) 11.47 (5.0) | 9.87 (4.56) | 11.27 (5.10) | -0.29 |
| median [IQR] | 9.00 [6.00, 12.00] | 10.00 [7.00, 14.00] | 9.00 [6.00, 12.00] | 10.00 [7.00, 14.00] | 9.00 [7.00, 12.00] 11.00 [8.00, 14.00 | | 10.65 (5.10) | -0.34 |
| Number of Hospitalizations | (,, | | (,, | | (, ==, == (, = | , | | 0.0 |
| mean (sd) | 0.13 (0.41) | 0.13 (0.41) | 0.14 (0.41) | 0.12 (0.39) | 0.18 (0.50) 0.16 (0.4) | 0.16 (0.47) | 0.15 (0.45) | 0.02 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] 0.00 [0.00, 0.00 | | 0.00 (0.45) | 0.00 |
| Number of hospital days | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] 0.00 [0.00, 0.00 | 0.00 (0.47) | 0.00 (0.43) | 0.00 |
| | 0.69 (3.15) | 0.67 (2.66) | 0.77 (3.34) | 0.66 (2.86) | 1.09 (4.32) 1.02 (3.9 | 0.95 (3.94) | 0.90 (3.60) | 0.01 |
| mean (sd)<br>median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] 0.00 [0.00, 0.00 | | 0.00 (3.60) | 0.01 |
| Number of Emergency Department (ED) visits | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] 0.00 [0.00, 0.00 | 0.00 (3.34) | 0.00 (3.00) | 0.00 |
| | 0.47 (1.25) | 0.40 (1.40) | 0.22 (1.51) | 0.10/1.26\ | 0.64 (1.48) 0.63 (1.44 | 0.53 (1.44) | 0.53 (1.40) | 0.00 |
| mean (sd) | | 0.49 (1.40) | 0.22 (1.51) | 0.19 (1.26) | | | | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] 0.00 [0.00, 0.00 | 0.00 (1.44) | 0.00 (1.40) | 0.00 |
| Number of Office visits | 4.04 (2.04) | 5.54(4.27) | 4.00 (4.40) | 5.07 (4.22) | 5 40 (4 27) | 5 24 (4 24) | C 45 (4 C2) | 0.20 |
| mean (sd) | 4.81 (3.84) | 5.54 (4.37) | 4.90 (4.19) | 5.87 (4.32) | 5.48 (4.37) 6.38 (4.7) | | 6.15 (4.63) | -0.20 |
| median [IQR] | 4.00 [2.00, 6.00] | 5.00 [3.00, 7.00] | 4.00 [2.00, 6.00] | 5.00 [3.00, 8.00] | 4.00 [2.00, 7.00] 5.00 [3.00, 9.00 | 9] 4.00 (4.24) | 5.00 (4.63) | -0.23 |
| Number of Endocrinologist visits | | | | | | | | |
| mean (sd) | 0.26 (1.68) | 0.81 (2.91) | 0.26 (1.60) | 0.84 (3.11) | 0.41 (2.46) 0.95 (3.73 | | 0.91 (3.49) | -0.19 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] 0.00 [0.00, 0.00 | 0.00 (2.18) | 0.00 (3.49) | 0.00 |
| Number of internal medicine/family medicine visits | | | | | | | | |
| mean (sd) | 10.22 (13.48) | 9.35 (14.19) | 6.96 (10.00) | 7.84 (9.99) | 8.22 (10.66) 8.99 (11.6) | | 8.86 (11.85) | -0.04 |
| median [IQR] | 6.00 [2.00, 13.00] | 5.00 [1.00, 12.00] | 4.00 [1.00, 9.00] | 5.00 [2.00, 10.00] | 5.00 [2.00, 11.00] 6.00 [2.00, 12.00 | 5.00 (11.14) | 5.65 (11.85) | -0.06 |
| Number of Cardiologist visits | | | | | | | | |
| mean (sd) | 1.70 (3.99) | 1.95 (4.52) | 1.27 (3.33) | 1.48 (3.46) | 2.19 (4.88) 2.34 (5.13 | 1.92 (4.46) | 2.12 (4.81) | -0.04 |
| median [IQR] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 2.00] 0.00 [0.00, 2.00 | 0.00 (4.46) | 0.00 (4.81) | 0.00 |
| Number electrocardiograms received | | | | | | | | |
| mean (sd) | 0.71 (1.48) | 0.76 (1.50) | 0.66 (1.30) | 0.67 (1.23) | 0.82 (1.50) 0.86 (1.50 | 0.77 (1.46) | 0.81 (1.46) | -0.03 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] 0.00 [0.00, 1.00 | 0.00 (1.46) | 0.00 (1.46) | 0.00 |
| Number of HbA1c tests ordered | | | | | | | | |
| mean (sd) | 1.14 (0.90) | 1.30 (0.95) | 0.81 (0.87) | 0.98 (0.94) | 1.26 (0.88) 1.47 (0.9) | 1.15 (0.88) | 1.36 (0.92) | -0.23 |
| median [IQR] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | 1.00 [1.00, 2.00] 1.00 [1.00, 2.00 | 1.00 (0.88) | 1.00 (0.92) | 0.00 |
| Number of glucose tests ordered | | | | | | | | |
| mean (sd) | 0.47 (2.91) | 1.00 (8.11) | 0.38 (1.34) | 0.49 (1.26) | 0.39 (1.05) 0.58 (1.33 | 9) 0.40 (1.63) | 0.64 (3.59) | -0.09 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] 0.00 [0.00, 1.00 | 0.00 (1.63) | 0.00 (3.59) | 0.00 |
| Number of lipid tests ordered | | | | | | | | |
| mean (sd) | 0.91 (0.94) | 1.03 (1.00) | 0.69 (1.15) | 0.86 (1.33) | 0.92 (0.83) 1.08 (0.90 | 0.87 (0.92) | 1.03 (1.00) | -0.17 |
| median [IQR] | 1.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] 1.00 [0.00, 2.00 | 0.81 (0.92) | 1.00 (1.00) | -0.20 |
| Number of creatinine tests ordered | | | | | | | | |
| mean (sd) | 0.06 (0.35) | 0.07 (0.47) | 0.10 (0.49) | 0.07 (0.58) | 0.10 (0.43) 0.09 (0.44 | 0.09 (0.43) | 0.08 (0.45) | 0.02 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] 0.00 [0.00, 0.00 | | 0.00 (0.45) | 0.00 |
| Number of BUN tests ordered | | | | | | | | |
| mean (sd) | 0.04 (0.29) | 0.04 (0.38) | 0.06 (0.40) | 0.05 (0.58) | 0.06 (0.34) 0.06 (0.33 | 2) 0.06 (0.34) | 0.05 (0.39) | 0.03 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] 0.00 [0.00, 0.00 | | 0.00 (0.39) | 0.00 |
| Number of tests for microalbuminuria | | | | | | | ( , | |
| mean (sd) | 0.73 (1.16) | 0.87 (1.32) | 0.44 (0.92) | 0.58 (1.05) | 0.42 (0.70) 0.57 (0.84 | 0.48 (0.85) | 0.62 (0.98) | -0.15 |
| median [IQR] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] 0.00 [0.00, 1.00 | | 0.00 (0.98) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd digit | ()) | ( | ( | ( | | | () | |
| level | | | | | | | | |
| mean (sd) | 5.56 (7.61) | 7.38 (8.79) | 2.27 (5.00) | 2.87 (5.40) | 6.02 (8.58) 7.70 (9.44 | 5.21 (7.83) | 6.82 (8.76) | -0.19 |
| median [IQR] | 3.00 [0.00, 9.00] | 5.00 [0.00, 11.00] | 0.00 [0.00, 3.00] | 0.00 [0.00, 4.00] | 3.00 [0.00, 9.00] 5.00 [0.00, 12.00 | | 4.14 (8.76) | -0.21 |
| | | | | | | . () | (3.1. 4) | |
| Use of thiazide; n (%) | 14,325 (12.6%) | 1,077 (12.1%) | 13,611 (11.9%) | 1,008 (11.5%) | 50,169 (13.7%) 4,605 (13.8% | 78,105 (13.1%) | 6,690 (13.1%) | 0.00 |
| Use of beta blockers; n (%) | 57,310 (50.3%) | 4,545 (51.0%) | 57,096 (50.1%) | 4,427 (50.7%) | 202,981 (55.4%) 19,093 (57.2% | | 28,065 (55.0%) | -0.03 |
| Use of calcium channel blockers; n (%) | 35,824 (31.4%) | 3,051 (34.3%) | 33,870 (29.7%) | 2,789 (31.9%) | 128,069 (35.0%) 13,043 (39.0% | | 18,883 (37.0%) | -0.08 |
| | | -, (,) | | , (- 2/-) | , | , | -,, | |

| | Optur | n I | MarketS | Scan I | Medica | are | | POOLED | |
|---|---|---|---|---|---|---|---|---|---|
| | Reference-2nd | • | Reference-2nd | - | Reference-2nd | • | Reference-2nd | | |
| Variable | Generation SUs | Exposure-Linagliptin | Generation SUs | Exposure-Linagliptin | Generation SUs | Exposure-Linagliptin | Generation SUs | Exposure-Linagliptin | St. Diff |
| Number of patients | 8880 | 8880 | 8716 | 8716 | 33319 | 33319 | 50,915 | 50,915 | |
| Age | CC 0C (10 0.1) | CC OC (11 C3) | C2 05 (14 54) | 62.76 (44.52) | 75 02 /7 22 | 75.07.(7.44) | 72 20 (0 00) | 72 24 (0.00) | 2.22 |
| mean (sd) | 66.96 (10.94) | 66.96 (11.63) | 63.85 (11.51) | 63.76 (11.53) | 75.92 (7.38) | 75.97 (7.44) | 72.29 (8.90) | 72.31 (9.09) | 0.00 |
| median [IQR] | 68.00 [60.00, 75.00] | 67.00 [59.00, 76.00] | 63.00 [56.00, 72.00] | 62.00 [56.00, 71.00] | 75.00 [70.00, 81.00] | 75.00 [70.00, 81.00] | 71.72 (8.90) | 71.38 (9.09) | 0.04 |
| Age categories | 1 227 (12 00/) | 1 242 (44 000) | 1 736 (40 000) | 1 745 /40 70/ | 0.00.000 | 0 (0 00/) | 2.052 (5.00() | 2 020 /5 00/\ | 0.00 |
| 18 - 54; n (%)<br>55 - 64; n (%) | 1,227 (13.8%)<br>1,986 (22.4%) | 1,313 (14.8%)<br>2,434 (27.4%) | 1,726 (19.8%)<br>3,404 (39.1%) | 1,715 (19.7%)<br>3,524 (40.4%) | 0 (0.0%)<br>307 (0.9%) | 0 (0.0%)<br>339 (1.0%) | 2,953 (5.8%)<br>5,697 (11.2%) | 3,028 (5.9%)<br>6,297 (12.4%) | 0.00<br>-0.04 |
| 65 - 74; n (%) | 3,436 (38.7%) | 2,634 (29.7%) | 1,870 (21.5%) | 1,781 (20.4%) | 15,789 (47.4%) | 15,632 (46.9%) | 21,095 (41.4%) | 20,047 (39.4%) | 0.04 |
| >= 75; n (%) | 2,231 (25.1%) | 2,499 (28.1%) | 1,716 (19.7%) | 1,696 (19.5%) | 17,223 (51.7%) | 17,348 (52.1%) | 21,170 (41.6%) | 21,543 (42.3%) | -0.01 |
| Gender | _,_51 (25.170) | _, .55 (25.270) | _,. 10 (15 70) | _,( | ,_25 (52., 70) | ,0(52.12,0) | , 0 (.1.0,0) | ,3 (12.374) | 3.01 |
| Males; n (%) | 4,699 (52.9%) | 4,669 (52.6%) | 4,973 (57.1%) | 5,039 (57.8%) | 14,083 (42.3%) | 14,131 (42.4%) | 23,755 (46.7%) | 23,839 (46.8%) | 0.00 |
| Females; n (%) | 4,181 (47.1%) | 4,211 (47.4%) | 3,743 (42.9%) | 3,677 (42.2%) | 19,236 (57.7%) | 19,188 (57.6%) | 27,160 (53.3%) | 27,076 (53.2%) | 0.00 |
| Race | | | | | | | | | |
| White; n (%) | N/A | N/A | N/A | N/A | 23,508 (70.6%) | 23,421 (70.3%) | 23,508 (70.6%) | 23,421 (70.3%) | 0.01 |
| Black; n (%) | N/A | N/A | N/A | N/A | 4,254 (12.8%) | 4,256 (12.8%) | 4,254 (12.8%) | 4,256 (12.8%) | 0.00 |
| Asian; n (%) | N/A | N/A | N/A | N/A | 2,120 (6.4%) | 2,151 (6.5%) | 2,120 (6.4%) | 2,151 (6.5%) | 0.00 |
| Hispanic; n (%) | N/A | N/A | N/A | N/A | 1,819 (5.5%) | 1,861 (5.6%) | 1,819 (5.5%) | 1,861 (5.6%) | 0.00 |
| North American Native; n (%) | N/A | N/A | N/A | N/A | 273 (0.8%) | 270 (0.8%) | 273 (0.8%) | 270 (0.8%) | 0.00 |
| Other/Unknown; n (%) Region (lumping missing&other category with | N/A | N/A | N/A | N/A | 1,345 (4.0%) | 1,360 (4.1%) | 1,345 (4.0%) | 1,360 (4.1%) | -0.01 |
| West) | | | | | | | | | |
| Northeast; n (%) | 1,134 (12.8%) | 1,141 (12.8%) | 1,872 (21.5%) | 1,936 (22.2%) | 6,759 (20.3%) | 6,789 (20.4%) | 9,765 (19.2%) | 9,866 (19.4%) | -0.01 |
| South; n (%) | 4,622 (52.0%) | 4,611 (51.9%) | 1,654 (19.0%) | 1,644 (18.9%) | 14,504 (43.5%) | 14,319 (43.0%) | 20,780 (40.8%) | 20,574 (40.4%) | 0.01 |
| Midwest; n (%) | 1,575 (17.7%) | 1,590 (17.9%) | 4,154 (47.7%) | 4,147 (47.6%) | 5,737 (17.2%) | 5,801 (17.4%) | 11,466 (22.5%) | 11,538 (22.7%) | 0.00 |
| West; n (%) | 1,549 (17.4%) | 1,538 (17.3%) | 934 (10.7%) | 895 (10.3%) | 6,319 (19.0%) | 6,410 (19.2%) | 8,802 (17.3%) | 8,843 (17.4%) | 0.00 |
| Unknown+missing; n (%) | N/A | N/A | 102 (1.2%) | 94 (1.1%) | N/A | N/A | 102 (1.2%) | 94 (1.1%) | 0.01 |
| CV Covariates | 2 400 (20 27) | 2.450/20.550 | 2 200 (25) | 2 020 (24 ==*) | 40.740./44.000 | 42.754 (44.260) | 20 220 (20 27) | 20 240 (20 00) | |
| Ischemic heart disease; n (%) | 3,488 (39.3%)<br>203 (2.3%) | 3,469 (39.1%)<br>211 (2.4%) | 3,098 (35.5%)<br>156 (1.8%) | 3,028 (34.7%)<br>164 (1.9%) | 13,743 (41.2%)<br>583 (1.7%) | 13,751 (41.3%)<br>570 (1.7%) | 20,329 (39.9%)<br>942 (1.9%) | 20,248 (39.8%)<br>945 (1.9%) | 0.00 |
| Acute MI; n (%) ACS/unstable angina; n (%) | 203 (2.3%)<br>133 (1.5%) | 211 (2.4%)<br>117 (1.3%) | 156 (1.8%) | 164 (1.9%)<br>125 (1.4%) | 459 (1.4%) | 570 (1.7%)<br>440 (1.3%) | 942 (1.9%)<br>712 (1.4%) | 945 (1.9%)<br>682 (1.3%) | 0.00 |
| Old MI; n (%) | 416 (4.7%) | 428 (4.8%) | 242 (2.8%) | 241 (2.8%) | 1,583 (4.8%) | 1,570 (4.7%) | 2,241 (4.4%) | 2,239 (4.4%) | 0.00 |
| Stable angina; n (%) | 547 (6.2%) | 539 (6.1%) | 387 (4.4%) | 381 (4.4%) | 1,727 (5.2%) | 1,702 (5.1%) | 2,661 (5.2%) | 2,622 (5.1%) | 0.00 |
| Coronary atherosclerosis and other forms of chronic | () | (/0) | (/9) | () | , (xy) | , == (=:=:-, | , ( ) | , (, | 3.00 |
| ischemic heart disease; n (%) | 3,205 (36.1%) | 3,212 (36.2%) | 2,873 (33.0%) | 2,834 (32.5%) | 13,040 (39.1%) | 13,022 (39.1%) | 19,118 (37.5%) | 19,068 (37.5%) | 0.00 |
| Other atherosclerosis with ICD10; n (%) | 94 (1.1%) | 114 (1.3%) | 92 (1.1%) | 107 (1.2%) | 657 (2.0%) | 680 (2.0%) | 843 (1.7%) | 901 (1.8%) | -0.01 |
| Previous cardiac procedure (CABG or PTCA or Stent); | | | | | | | | | |
| n (%) | 55 (0.6%) | 56 (0.6%) | 66 (0.8%) | 80 (0.9%) | 168 (0.5%) | 170 (0.5%) | 289 (0.6%) | 306 (0.6%) | 0.00 |
| History of CABG or PTCA; n (%) | 755 (8.5%) | 776 (8.7%) | 363 (4.2%) | 380 (4.4%) | 3,490 (10.5%) | 3,405 (10.2%) | 4,608 (9.1%) | 4,561 (9.0%) | 0.00 |
| Any stroke; n (%) | 337 (3.8%) | 343 (3.9%) | 345 (4.0%) | 353 (4.1%) | 1,782 (5.3%) | 1,830 (5.5%) | 2,464 (4.8%) | 2,526 (5.0%) | -0.01 |
| Ischemic stroke (w and w/o mention of cerebral infarction); n (%) | 333 (3.8%) | 335 (3.8%) | 341 (3.9%) | 347 (4.0%) | 1,754 (5.3%) | 1,810 (5.4%) | 2,428 (4.8%) | 2,492 (4.9%) | 0.00 |
| Hemorrhagic stroke; n (%) | 6 (0.1%) | 13 (0.1%) | 7 (0.1%) | 10 (0.1%) | 33 (0.1%) | 32 (0.1%) | 2,428 (4.8%) | 2,492 (4.9%)<br>055 (0.1%) | 0.00 |
| TIA; n (%) | 57 (0.6%) | 56 (0.6%) | 52 (0.6%) | 62 (0.7%) | 329 (1.0%) | 336 (1.0%) | 438 (0.9%) | 454 (0.9%) | 0.00 |
| Other cerebrovascular disease; n (%) | 198 (2.2%) | 177 (2.0%) | 98 (1.1%) | 111 (1.3%) | 957 (2.9%) | 948 (2.8%) | 1,253 (2.5%) | 1,236 (2.4%) | 0.01 |
| Late effects of cerebrovascular disease; n (%) | 172 (1.9%) | 170 (1.9%) | 73 (0.8%) | 70 (0.8%) | 822 (2.5%) | 842 (2.5%) | 1,067 (2.1%) | 1,082 (2.1%) | 0.00 |
| Cerebrovascular procedure; n (%) | 4 (0.0%) | 3 (0.0%) | 4 (0.0%) | 3 (0.0%) | 13 (0.0%) | 11 (0.0%) | 021 (0.0%) | 017 (0.0%) | #DIV/0! |
| Heart failure (CHF); n (%) | 1,118 (12.6%) | 1,140 (12.8%) | 839 (9.6%) | 820 (9.4%) | 5,351 (16.1%) | 5,337 (16.0%) | 7,308 (14.4%) | 7,297 (14.3%) | 0.00 |
| Peripheral Vascular Disease (PVD) or PVD Surgery ; n | | | | | | | | | |
| (%) | 878 (9.9%) | 872 (9.8%) | 593 (6.8%) | 558 (6.4%) | 4,957 (14.9%) | 4,955 (14.9%) | 6,428 (12.6%) | 6,385 (12.5%) | 0.00 |
| Atrial fibrillation; n (%) | 835 (9.4%) | 845 (9.5%) | 738 (8.5%) | 733 (8.4%) | 4,861 (14.6%) | 4,884 (14.7%) | 6,434 (12.6%) | 6,462 (12.7%) | 0.00 |
| Other cardiac dysrhythmia; n (%) | 1,125 (12.7%) | 1,103 (12.4%) | 799 (9.2%) | 800 (9.2%) | 5,521 (16.6%) | 5,531 (16.6%) | 7,445 (14.6%) | 7,434 (14.6%) | 0.00 |
| Cardiac conduction disorders; n (%) | 336 (3.8%) | 329 (3.7%) | 248 (2.8%) | 238 (2.7%) | 1,680 (5.0%) | 1,576 (4.7%) | 2,264 (4.4%) | 2,143 (4.2%) | 0.01 |
| Other CVD; n (%) | 1,272 (14.3%) | 1,278 (14.4%) | 1,147 (13.2%) | 1,134 (13.0%) | 6,324 (19.0%) | 6,350 (19.1%) | 8,743 (17.2%) | 8,762 (17.2%) | 0.00 |
| Diabetes-related complications Diabetic retinopathy; n (%) | 630 (7.1%) | 670 (7.5%) | 375 (4.3%) | 397 (4.6%) | 2,635 (7.9%) | 2,651 (8.0%) | 3,640 (7.1%) | 3,718 (7.3%) | -0.01 |
| Diabetes with other ophthalmic manifestations; n | 030 (7.1%) | 070 (7.5%) | 3/3(4.3%) | 337 (4.0%) | 2,033 (1.9%) | 2,031 (0.0%) | 3,040 (7.170) | 3,710(7.370) | -0.01 |
| (%) | 74 (0.8%) | 58 (0.7%) | 258 (3.0%) | 254 (2.9%) | 953 (2.9%) | 937 (2.8%) | 1,285 (2.5%) | 1,249 (2.5%) | 0.00 |
| Retinal detachment, vitreous hemorrhage, | ,/ | (- /-/ | () | - (/ | , | - , , | (/ | | |
| vitrectomy; n (%) | 44 (0.5%) | 61 (0.7%) | 36 (0.4%) | 52 (0.6%) | 137 (0.4%) | 163 (0.5%) | 217 (0.4%) | 276 (0.5%) | -0.01 |
| Retinal laser coagulation therapy; n (%) | 41 (0.5%) | 70 (0.8%) | 51 (0.6%) | 67 (0.8%) | 205 (0.6%) | 253 (0.8%) | 297 (0.6%) | 390 (0.8%) | -0.02 |
| Occurrence of Diabetic Neuropathy ; n (%) | 1,816 (20.5%) | 1,833 (20.6%) | 1,090 (12.5%) | 1,109 (12.7%) | 7,317 (22.0%) | 7,280 (21.8%) | 10,223 (20.1%) | 10,222 (20.1%) | 0.00 |

| Occurrence of diabetic nephropathy with ICD10; n | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| (%) | 2,215 (24.9%) | 2,268 (25.5%) | 1,124 (12.9%) | 1,114 (12.8%) | 6,355 (19.1%) | 6,416 (19.3%) | 9,694 (19.0%) | 9,798 (19.2%) | -0.01 |
| Hypoglycemia; n (%) | 216 (2.4%) | 226 (2.5%) | 195 (2.2%) | 207 (2.4%) | 1,053 (3.2%) | 1,079 (3.2%) | 1,464 (2.9%) | 1,512 (3.0%) | -0.01 |
| Hyperglycemia; n (%) | 568 (6.4%) | 544 (6.1%) | 348 (4.0%) | 342 (3.9%) | 2,120 (6.4%) | 2,159 (6.5%) | 3,036 (6.0%) | 3,045 (6.0%) | 0.00 |
| Disorders of fluid electrolyte and acid-base balance; n | | | | | | | | | |
| (%) | 1,091 (12.3%) | 1,051 (11.8%) | 568 (6.5%) | 617 (7.1%) | 4,041 (12.1%) | 4,017 (12.1%) | 5,700 (11.2%) | 5,685 (11.2%) | 0.00 |
| Diabetic ketoacidosis; n (%) | 37 (0.4%) | 35 (0.4%) | 41 (0.5%) | 24 (0.3%) | 171 (0.5%) | 126 (0.4%) | 249 (0.5%) | 185 (0.4%) | 0.01 |
| Hyperosmolar hyperglycemic nonketotic syndrome (HONK); n (%) | 49 (0.6%) | 55 (0.6%) | 37 (0.4%) | 41 (0.5%) | 205 (0.6%) | 216 (0.6%) | 291 (0.6%) | 312 (0.6%) | 0.00 |
| Diabetes with peripheral circulatory disorders with | 45 (0.0%) | 33 (0.0%) | 37 (0.470) | 41 (0.3%) | 203 (0.0%) | 210 (0.076) | 231 (0.0%) | 312 (0.0%) | 0.00 |
| ICD-10 ; n (%) | 808 (9.1%) | 808 (9.1%) | 373 (4.3%) | 400 (4.6%) | 3,068 (9.2%) | 3,123 (9.4%) | 4,249 (8.3%) | 4,331 (8.5%) | -0.01 |
| Diabetic Foot; n (%) | 268 (3.0%) | 269 (3.0%) | 184 (2.1%) | 199 (2.3%) | 1,098 (3.3%) | 1,078 (3.2%) | 1,550 (3.0%) | 1,546 (3.0%) | 0.00 |
| Gangrene; n (%) | 31 (0.3%) | 31 (0.3%) | 14 (0.2%) | 16 (0.2%) | 107 (0.3%) | 101 (0.3%) | 152 (0.3%) | 148 (0.3%) | 0.00 |
| Lower extremity amputation; n (%) | 80 (0.9%) | 96 (1.1%) | 31 (0.4%) | 38 (0.4%) | 277 (0.8%) | 276 (0.8%) | 388 (0.8%) | 410 (0.8%) | 0.00 |
| Osteomyelitis; n (%) | 66 (0.7%) | 78 (0.9%) | 54 (0.6%) | 46 (0.5%) | 240 (0.7%) | 210 (0.6%) | 360 (0.7%) | 334 (0.7%) | 0.00 |
| Skin infections ; n (%) | 569 (6.4%) | 539 (6.1%) | 501 (5.7%) | 522 (6.0%) | 2,480 (7.4%) | 2,528 (7.6%) | 3,550 (7.0%) | 3,589 (7.0%) | 0.00 |
| Erectile dysfunction; n (%) | 246 (2.8%) | 241 (2.7%) | 220 (2.5%) | 216 (2.5%) | 644 (1.9%) | 644 (1.9%) | 1,110 (2.2%) | 1,101 (2.2%) | 0.00 |
| Diabetes with unspecified complication; n (%) | 627 (7.1%) | 606 (6.8%) | 370 (4.2%) | 388 (4.5%) | 2,097 (6.3%) | 2,070 (6.2%) | 3,094 (6.1%) | 3,064 (6.0%) | 0.00 |
| Diabetes mellitus without mention of complications; | | // | | | | | | | |
| n (%) | 7,608 (85.7%) | 7,607 (85.7%) | 7,937 (91.1%) | 7,943 (91.1%) | 30,740 (92.3%) | 30,751 (92.3%) | 46,285 (90.9%) | 46,301 (90.9%) | 0.00 |
| Hypertension: 1 inpatient or 2 outpatient claims | 7.873 (88.7%) | 7,855 (88.5%) | 6.785 (77.8%) | 6,815 (78.2%) | 31,536 (94.6%) | 31,451 (94.4%) | 46.194 (90.7%) | 46,121 (90.6%) | 0.00 |
| within 365 days; n (%)<br>Hyperlipidemia ; n (%) | 6,695 (75.4%) | 6,689 (75.3%) | 5,614 (64.4%) | 5,628 (64.6%) | 26,315 (79.0%) | 26,388 (79.2%) | 38,624 (75.9%) | 38,705 (76.0%) | 0.00 |
| Edema; n (%) | 818 (9.2%) | 809 (9.1%) | 556 (6.4%) | 553 (6.3%) | 4,504 (13.5%) | 4,434 (13.3%) | 5,878 (11.5%) | 5,796 (11.4%) | 0.00 |
| Renal Dysfunction (non-diabetic) ; n (%) | 3,697 (41.6%) | 3,732 (42.0%) | 2,456 (28.2%) | 2,511 (28.8%) | 13,956 (41.9%) | 14,275 (42.8%) | 20,109 (39.5%) | 20,518 (40.3%) | -0.02 |
| Occurrence of acute renal disease ; n (%) | 643 (7.2%) | 603 (6.8%) | 422 (4.8%) | 419 (4.8%) | 2,452 (7.4%) | 2,378 (7.1%) | 3,517 (6.9%) | 3,400 (6.7%) | 0.01 |
| Occurrence of chronic renal insufficiency; n (%) | 3,381 (38.1%) | 3,371 (38.0%) | 2,101 (24.1%) | 2,150 (24.7%) | 12,524 (37.6%) | 12,774 (38.3%) | 18,006 (35.4%) | 18,295 (35.9%) | -0.01 |
| Chronic kidney disease ; n (%) | 3,319 (37.4%) | 3,314 (37.3%) | 2,065 (23.7%) | 2,102 (24.1%) | 12,176 (36.5%) | 12,358 (37.1%) | 17,560 (34.5%) | 17,774 (34.9%) | -0.01 |
| CKD Stage 3-4; n (%) | 2,764 (31.1%) | 2,781 (31.3%) | 1,669 (19.1%) | 1,702 (19.5%) | 9,803 (29.4%) | 9,776 (29.3%) | 14,236 (28.0%) | 14,259 (28.0%) | 0.00 |
| Occurrence of hypertensive nephropathy; n (%) | 1,472 (16.6%) | 1,471 (16.6%) | 723 (8.3%) | 751 (8.6%) | 5,364 (16.1%) | 5,361 (16.1%) | 7,559 (14.8%) | 7,583 (14.9%) | 0.00 |
| Occurrence of miscellaneous renal insufficiency; n | | | | | | | | | |
| (%) | 800 (9.0%) | 790 (8.9%) | 601 (6.9%) | 586 (6.7%) | 3,837 (11.5%) | 3,718 (11.2%) | 5,238 (10.3%) | 5,094 (10.0%) | 0.01 |
| Glaucoma or cataracts ; n (%) | 1,689 (19.0%) | 1,764 (19.9%) | 1,481 (17.0%) | 1,507 (17.3%) | 9,097 (27.3%) | 9,110 (27.3%) | 12,267 (24.1%) | 12,381 (24.3%) | 0.00 |
| Cellulitis or abscess of toe; n (%) | 166 (1.9%) | 138 (1.6%) | 82 (0.9%) | 101 (1.2%) | 570 (1.7%) | 591 (1.8%) | 818 (1.6%) | 830 (1.6%) | 0.00 |
| Foot ulcer; n (%) | 250 (2.8%) | 257 (2.9%) | 185 (2.1%) | 194 (2.2%) | 1,091 (3.3%) | 1,069 (3.2%) | 1,526 (3.0%) | 1,520 (3.0%) | 0.00 |
| Bladder stones; n (%) | 17 (0.2%) | 16 (0.2%) | 17 (0.2%) | 17 (0.2%) | 70 (0.2%) | 66 (0.2%) | 104 (0.2%) | 099 (0.2%) | 0.00 |
| Kidney stones; n (%) | 290 (3.3%) | 272 (3.1%) | 270 (3.1%) | 260 (3.0%) | 1,031 (3.1%) | 1,010 (3.0%) | 1,591 (3.1%) | 1,542 (3.0%) | 0.01 |
| Urinary tract infections (UTIs); n (%) | 1,036 (11.7%)<br>3,574 (40.2%) | 1,013 (11.4%) | 622 (7.1%)<br>2,997 (34.4%) | 641 (7.4%)<br>3,094 (35.5%) | 6,198 (18.6%) | 6,107 (18.3%) | 7,856 (15.4%)<br>22,097 (43.4%) | 7,761 (15.2%) | 0.01<br>-0.03 |
| Dipstick urinalysis; n (%) Non-dipstick urinalysis; n (%) | 4,002 (45.1%) | 3,671 (41.3%)<br>3,900 (43.9%) | 2,841 (32.6%) | 2,809 (32.2%) | 15,526 (46.6%)<br>14,418 (43.3%) | 16,153 (48.5%)<br>14,601 (43.8%) | 21,261 (41.8%) | 22,918 (45.0%)<br>21,310 (41.9%) | 0.00 |
| Urine function test; n (%) | 264 (3.0%) | 209 (2.4%) | 267 (3.1%) | 280 (3.2%) | 1,361 (4.1%) | 1,370 (4.1%) | 1,892 (3.7%) | 1,859 (3.7%) | 0.00 |
| Cytology; n (%) | 81 (0.9%) | 88 (1.0%) | 105 (1.2%) | 120 (1.4%) | 438 (1.3%) | 437 (1.3%) | 624 (1.2%) | 645 (1.3%) | -0.01 |
| Cystos; n (%) | 114 (1.3%) | 111 (1.2%) | 154 (1.8%) | 150 (1.7%) | 666 (2.0%) | 561 (1.7%) | 934 (1.8%) | 822 (1.6%) | 0.02 |
| Other Covariates | , , | , , | , | , | , , | , | , , , | ,, | |
| Liver disease; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| Osteoarthritis; n (%) | 1,546 (17.4%) | 1,513 (17.0%) | 1,091 (12.5%) | 1,080 (12.4%) | 8,803 (26.4%) | 8,745 (26.2%) | 11,440 (22.5%) | 11,338 (22.3%) | 0.00 |
| Other arthritis, arthropathies and musculoskeletal | | | | | | | | | |
| pain; n (%) | 3,601 (40.6%) | 3,513 (39.6%) | 2,985 (34.2%) | 2,986 (34.3%) | 16,525 (49.6%) | 16,480 (49.5%) | 23,111 (45.4%) | 22,979 (45.1%) | 0.01 |
| Dorsopathies; n (%) | 2,069 (23.3%) | 2,033 (22.9%) | 1,824 (20.9%) | 1,828 (21.0%) | 9,548 (28.7%) | 9,466 (28.4%) | 13,441 (26.4%) | 13,327 (26.2%) | 0.00 |
| Fractures; n (%) | 297 (3.3%) | 304 (3.4%) | 232 (2.7%) | 222 (2.5%) | 1,576 (4.7%) | 1,511 (4.5%) | 2,105 (4.1%) | 2,037 (4.0%) | 0.01 |
| Falls; n (%) | 385 (4.3%) | 392 (4.4%) | 97 (1.1%) | 107 (1.2%) | 1,769 (5.3%) | 1,804 (5.4%) | 2,251 (4.4%) | 2,303 (4.5%) | 0.00 |
| Osteoporosis; n (%) | 547 (6.2%) | 538 (6.1%) | 266 (3.1%) | 262 (3.0%) | 3,873 (11.6%) | 3,962 (11.9%) | 4,686 (9.2%) | 4,762 (9.4%) | -0.01 |
| Hyperthyroidism; n (%) | 76 (0.9%) | 97 (1.1%) | 52 (0.6%) | 55 (0.6%) | 415 (1.2%) | 425 (1.3%) | 543 (1.1%) | 577 (1.1%) | 0.00<br>0.01 |
| Hypothyroidism; n (%) Other disorders of thyroid gland; n (%) | 1,610 (18.1%)<br>377 (4.2%) | 1,667 (18.8%)<br>415 (4.7%) | 1,178 (13.5%)<br>349 (4.0%) | 1,119 (12.8%)<br>382 (4.4%) | 5,372 (16.1%)<br>1,687 (5.1%) | 5,234 (15.7%)<br>1,772 (5.3%) | 8,160 (16.0%)<br>2,413 (4.7%) | 8,020 (15.8%)<br>2,569 (5.0%) | -0.01 |
| Depression; n (%) | 817 (9.2%) | 801 (9.0%) | 567 (6.5%) | 557 (6.4%) | 3,892 (11.7%) | 3,839 (11.5%) | 5,276 (10.4%) | 5,197 (10.2%) | 0.01 |
| Anxiety; n (%) | 788 (8.9%) | 781 (8.8%) | 438 (5.0%) | 448 (5.1%) | 3,208 (9.6%) | 3,189 (9.6%) | 4,434 (8.7%) | 4,418 (8.7%) | 0.00 |
| Sleep_Disorder; n (%) | 602 (6.8%) | 590 (6.6%) | 882 (10.1%) | 870 (10.0%) | 2,750 (8.3%) | 2,717 (8.2%) | 4,234 (8.3%) | 4,177 (8.2%) | 0.00 |
| Dementia; n (%) | 534 (6.0%) | 533 (6.0%) | 247 (2.8%) | 223 (2.6%) | 3,583 (10.8%) | 3,529 (10.6%) | 4,364 (8.6%) | 4,285 (8.4%) | 0.01 |
| Delirium; n (%) | 143 (1.6%) | 147 (1.7%) | 72 (0.8%) | 72 (0.8%) | 837 (2.5%) | 848 (2.5%) | 1,052 (2.1%) | 1,067 (2.1%) | 0.00 |
| Psychosis; n (%) | 112 (1.3%) | 129 (1.5%) | 57 (0.7%) | 55 (0.6%) | 795 (2.4%) | 792 (2.4%) | 964 (1.9%) | 976 (1.9%) | 0.00 |
| Obesity; n (%) | 1,752 (19.7%) | 1,655 (18.6%) | 1,002 (11.5%) | 983 (11.3%) | 3,985 (12.0%) | 3,909 (11.7%) | 6,739 (13.2%) | 6,547 (12.9%) | 0.01 |
| Overweight; n (%) | 576 (6.5%) | 587 (6.6%) | 146 (1.7%) | 164 (1.9%) | 1,351 (4.1%) | 1,340 (4.0%) | 2,073 (4.1%) | 2,091 (4.1%) | 0.00 |
| Smoking; n (%) | 1,147 (12.9%) | 1,120 (12.6%) | 445 (5.1%) | 472 (5.4%) | 4,307 (12.9%) | 4,230 (12.7%) | 5,899 (11.6%) | 5,822 (11.4%) | 0.01 |
| Alcohol abuse or dependence; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| Drug abuse or dependence; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| COPD; n (%) | 947 (10.7%) | 878 (9.9%) | 636 (7.3%) | 617 (7.1%) | 4,686 (14.1%) | 4,669 (14.0%) | 6,269 (12.3%) | 6,164 (12.1%) | 0.01 |

| Asthma; n (%) | 572 (6.4%) | 566 (6.4%) | 453 (5.2%) | 423 (4.9%) | 2,227 (6.7%) | 2,213 (6.6%) | 3,252 (6.4%) | 3,202 (6.3%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Obstructive sleep apnea; n (%) | 916 (10.3%) | 873 (9.8%) | 947 (10.9%) | 934 (10.7%) | 2,238 (6.7%) | 2,212 (6.6%) | 4,101 (8.1%) | 4,019 (7.9%) | 0.01 |
| Pneumonia; n (%) | 325 (3.7%) | 313 (3.5%) | 229 (2.6%) | 240 (2.8%) | 1,503 (4.5%) | 1,501 (4.5%) | 2,057 (4.0%) | 2,054 (4.0%) | 0.00 |
| Imaging; n (%) | 9 (0.1%) | 17 (0.2%) | 11 (0.1%) | 7 (0.1%) | 74 (0.2%) | 54 (0.2%) | 94 (0.2%) | 78 (0.2%) | 0.00 |
| Diabetes Medications DM Medications - AGIs; n (%) | 40 (0.5%) | 32 (0.4%) | 33 (0.4%) | 32 (0.4%) | 210 (0.6%) | 194 (0.6%) | 283 (0.6%) | 258 (0.5%) | 0.01 |
| DM Medications - Adis, it (%) DM Medications - Glitazones; n (%) | 625 (7.0%) | 616 (6.9%) | 856 (9.8%) | 836 (9.6%) | 2,492 (7.5%) | 2,468 (7.4%) | 3,973 (7.8%) | 3,920 (7.7%) | 0.00 |
| DM Medications - Insulin; n (%) | 2,377 (26.8%) | 2,402 (27.0%) | 1,870 (21.5%) | 1,896 (21.8%) | 9,270 (27.8%) | 9,320 (28.0%) | 13,517 (26.5%) | 13,618 (26.7%) | 0.00 |
| DM Medications - Meglitinides; n (%) | 171 (1.9%) | 179 (2.0%) | 249 (2.9%) | 240 (2.8%) | 1,105 (3.3%) | 1,154 (3.5%) | 1,525 (3.0%) | 1,573 (3.1%) | -0.01 |
| DM Medications - Metformin; n (%) | 5,016 (56.5%) | 4,907 (55.3%) | 5,021 (57.6%) | 4,978 (57.1%) | 17,725 (53.2%) | 17,642 (52.9%) | 27,762 (54.5%) | 27,527 (54.1%) | 0.01 |
| Concomitant initiation or current use of SGLT2i; n | 3,010 (30.376) | 4,507 (33.376) | 3,021 (37.0%) | 4,578 (57.178) | 17,723 (33.270) | 17,042 (32.376) | 27,702 (34.370) | 27,327 (34.170) | 0.01 |
| (%) | 51 (0.6%) | 267 (3.0%) | 62 (0.7%) | 559 (6.4%) | 22 (0.1%) | 412 (1.2%) | #VALUE! | 1,238 (2.4%) | #VALUE! |
| Concomitant initiation or current use of AGIs; n (%) | 31 (0.3%) | 26 (0.3%) | 26 (0.3%) | 23 (0.3%) | 138 (0.4%) | 128 (0.4%) | 195 (0.4%) | 177 (0.3%) | 0.02 |
| Concomitant initiation or current use of Glitazones; | () | == (=:=,-, | == (=:=:-) | (0.07.7) | | === (=:, | () | | ***- |
| n (%) | 427 (4.8%) | 423 (4.8%) | 539 (6.2%) | 525 (6.0%) | 1,750 (5.3%) | 1,734 (5.2%) | 2,716 (5.3%) | 2,682 (5.3%) | 0.00 |
| Concomitant initiation or current use of Insulin; n | | | | | | | | | |
| (%) | 1,806 (20.3%) | 1,841 (20.7%) | 1,393 (16.0%) | 1,435 (16.5%) | 7,081 (21.3%) | 7,195 (21.6%) | 10,280 (20.2%) | 10,471 (20.6%) | -0.01 |
| Concomitant initiation or current use of | | | | | | | | | |
| Meglitinides; n (%) | 118 (1.3%) | 129 (1.5%) | 191 (2.2%) | 187 (2.1%) | 821 (2.5%) | 860 (2.6%) | 1,130 (2.2%) | 1,176 (2.3%) | -0.01 |
| Concomitant initiation or current use of Metformin; | | | | | | | | | |
| n (%) | 4,016 (45.2%) | 3,909 (44.0%) | 4,013 (46.0%) | 3,970 (45.5%) | 13,978 (42.0%) | 13,920 (41.8%) | 22,007 (43.2%) | 21,799 (42.8%) | 0.01 |
| Past use of SGLT2i; n (%) | 0 (0.0%) | 0 (0.0%) | 1 (0.0%) | 1 (0.0%) | 0 (0.0%) | 0 (0.0%) | 001 (0.0%) | 001 (0.0%) | #DIV/0! |
| Past use of AGIs ; n (%) | 9 (0.1%) | 6 (0.1%) | 7 (0.1%) | 9 (0.1%) | 72 (0.2%) | 66 (0.2%) | 088 (0.2%) | 081 (0.2%) | 0.00 |
| Past use of Glitazones ; n (%) | 198 (2.2%) | 193 (2.2%) | 317 (3.6%) | 311 (3.6%) | 742 (2.2%) | 734 (2.2%) | 1,257 (2.5%) | 1,238 (2.4%) | 0.01 |
| Past use of Insulin ; n (%) | 571 (6.4%) | 561 (6.3%) | 477 (5.5%) | 461 (5.3%) | 2,189 (6.6%) | 2,125 (6.4%) | 3,237 (6.4%) | 3,147 (6.2%) | 0.01 |
| Past use of Meglitinides ; n (%) | 53 (0.6%) | 50 (0.6%) | 58 (0.7%) | 53 (0.6%) | 284 (0.9%) | 294 (0.9%) | 395 (0.8%) | 397 (0.8%) | 0.00 |
| Past use of metformin ; n (%) | 1,000 (11.3%) | 998 (11.2%) | 1,008 (11.6%) | 1,008 (11.6%) | 3,747 (11.2%) | 3,722 (11.2%) | 5,755 (11.3%) | 5,728 (11.3%) | 0.00 |
| Other Medications | | | | | | | | | |
| Use of ACE inhibitors; n (%) | 3,677 (41.4%) | 3,668 (41.3%) | 3,499 (40.1%) | 3,486 (40.0%) | 12,931 (38.8%) | 12,775 (38.3%) | 20,107 (39.5%) | 19,929 (39.1%) | 0.01 |
| Use of ARBs; n (%) | 2,818 (31.7%) | 2,768 (31.2%) | 2,906 (33.3%) | 2,848 (32.7%) | 11,910 (35.7%) | 11,911 (35.7%) | 17,634 (34.6%) | 17,527 (34.4%) | 0.00 |
| Use of Loop Diuretics ; n (%) | 1,851 (20.8%) | 1,824 (20.5%) | 1,700 (19.5%) | 1,683 (19.3%) | 8,927 (26.8%) | 8,978 (26.9%) | 12,478 (24.5%) | 12,485 (24.5%) | 0.00 |
| Use of other diuretics; n (%) | 441 (5.0%) | 433 (4.9%) | 413 (4.7%) | 439 (5.0%) | 1,637 (4.9%) | 1,626 (4.9%) | 2,491 (4.9%) | 2,498 (4.9%) | 0.00 |
| Use of nitrates-United; n (%) | 753 (8.5%) | 769 (8.7%) | 730 (8.4%) | 744 (8.5%) | 3,871 (11.6%) | 3,853 (11.6%) | 5,354 (10.5%) | 5,366 (10.5%) | 0.00 |
| Use of other hypertension drugs; n (%) | 886 (10.0%) | 915 (10.3%) | 768 (8.8%) | 793 (9.1%) | 3,857 (11.6%) | 3,850 (11.6%) | 5,511 (10.8%) | 5,558 (10.9%) | 0.00 |
| Use of digoxin; n (%) | 202 (2.3%) | 219 (2.5%) | 280 (3.2%) | 272 (3.1%) | 1,335 (4.0%) | 1,344 (4.0%) | 1,817 (3.6%) | 1,835 (3.6%) | 0.00 |
| Use of Anti-arrhythmics; n (%) | 160 (1.8%) | 176 (2.0%) | 211 (2.4%) | 216 (2.5%) | 1,078 (3.2%) | 1,054 (3.2%) | 1,449 (2.8%) | 1,446 (2.8%) | 0.00<br>0.00 |
| Use of COPD/asthma meds; n (%) | 1,624 (18.3%) | 1,602 (18.0%) | 1,488 (17.1%) | 1,459 (16.7%) | 6,907 (20.7%) | 6,986 (21.0%) | 10,019 (19.7%) | 10,047 (19.7%) | 0.00 |
| Use of statins; n (%) | 6,456 (72.7%) | 6,428 (72.4%) | 6,090 (69.9%) | 6,081 (69.8%) | 24,525 (73.6%) | 24,594 (73.8%) | 37,071 (72.8%) | 37,103 (72.9%) | 0.00 |
| Use of other lipid-lowering drugs; n (%) Use of antiplatelet agents; n (%) | 1,261 (14.2%)<br>1,797 (20.2%) | 1,221 (13.8%) | 1,542 (17.7%) | 1,522 (17.5%) | 4,758 (14.3%) | 4,860 (14.6%) | 7,561 (14.9%)<br>10,873 (21.4%) | 7,603 (14.9%) | 0.00 |
| Use of oral anticoagulants (Dabigatran, Rivaroxaban, | 1,797 (20.2%) | 1,745 (19.7%) | 1,849 (21.2%) | 1,859 (21.3%) | 7,227 (21.7%) | 7,176 (21.5%) | 10,673 (21.4%) | 10,780 (21.2%) | 0.00 |
| Apixaban, Warfarin); n (%) | 738 (8.3%) | 745 (8.4%) | 777 (8.9%) | 791 (9.1%) | 3,971 (11.9%) | 4,016 (12.1%) | 5,486 (10.8%) | 5,552 (10.9%) | 0.00 |
| Use of heparin and other low-molecular weight | 750 (0.570) | 743 (0.470) | 777 (0.570) | 731 (3.170) | 3,371 (11.370) | 4,010 (12.170) | 3,400 (10.070) | 3,332 (10.370) | 0.00 |
| heparins; n (%) | 48 (0.5%) | 50 (0.6%) | 0 (0.0%) | 1 (0.0%) | 153 (0.5%) | 157 (0.5%) | 201 (0.4%) | 208 (0.4%) | 0.00 |
| Use of NSAIDs; n (%) | 1,244 (14.0%) | 1,269 (14.3%) | 1,257 (14.4%) | 1,290 (14.8%) | 5,605 (16.8%) | 5,590 (16.8%) | 8,106 (15.9%) | 8,149 (16.0%) | 0.00 |
| Use of oral corticosteroids; n (%) | 1,594 (18.0%) | 1,591 (17.9%) | 1,506 (17.3%) | 1,498 (17.2%) | 6,811 (20.4%) | 6,858 (20.6%) | 9,911 (19.5%) | 9,947 (19.5%) | 0.00 |
| Use of bisphosphonate (United); n (%) | 251 (2.8%) | 227 (2.6%) | 145 (1.7%) | 137 (1.6%) | 1,662 (5.0%) | 1,654 (5.0%) | 2,058 (4.0%) | 2,018 (4.0%) | 0.00 |
| Use of opioids; n (%) | 2,261 (25.5%) | 2,252 (25.4%) | 2,322 (26.6%) | 2,292 (26.3%) | 9,179 (27.5%) | 9,004 (27.0%) | 13,762 (27.0%) | 13,548 (26.6%) | 0.01 |
| Use of antidepressants; n (%) | 2,221 (25.0%) | 2,233 (25.1%) | 2,105 (24.2%) | 2,136 (24.5%) | 9,564 (28.7%) | 9,481 (28.5%) | 13,890 (27.3%) | 13,850 (27.2%) | 0.00 |
| Use of antipsychotics; n (%) | 299 (3.4%) | 303 (3.4%) | 225 (2.6%) | 213 (2.4%) | 1,538 (4.6%) | 1,500 (4.5%) | 2,062 (4.0%) | 2,016 (4.0%) | 0.00 |
| Use of anticonvulsants; n (%) | 1,634 (18.4%) | 1,672 (18.8%) | 1,336 (15.3%) | 1,314 (15.1%) | 6,898 (20.7%) | 7,000 (21.0%) | 9,868 (19.4%) | 9,986 (19.6%) | -0.01 |
| Use of lithium; n (%) | 16 (0.2%) | 9 (0.1%) | 20 (0.2%) | 15 (0.2%) | 55 (0.2%) | 40 (0.1%) | 091 (0.2%) | 064 (0.1%) | 0.03 |
| Use of Benzos; n (%) | 1,041 (11.7%) | 1,028 (11.6%) | 1,030 (11.8%) | 1,033 (11.9%) | 4,194 (12.6%) | 4,237 (12.7%) | 6,265 (12.3%) | 6,298 (12.4%) | 0.00 |
| Use of anxiolytics/hypnotics; n (%) | 592 (6.7%) | 594 (6.7%) | 633 (7.3%) | 641 (7.4%) | 2,449 (7.4%) | 2,406 (7.2%) | 3,674 (7.2%) | 3,641 (7.2%) | 0.00 |
| Use of dementia meds; n (%) | 333 (3.8%) | 319 (3.6%) | 234 (2.7%) | 206 (2.4%) | 2,601 (7.8%) | 2,618 (7.9%) | 3,168 (6.2%) | 3,143 (6.2%) | 0.00 |
| Use of antiparkinsonian meds; n (%) | 283 (3.2%) | 259 (2.9%) | 222 (2.5%) | 207 (2.4%) | 1,350 (4.1%) | 1,365 (4.1%) | 1,855 (3.6%) | 1,831 (3.6%) | 0.00 |
| Any use of pramlintide; n (%) | 0 (0.0%) | 5 (0.1%) | 10 (0.1%) | 5 (0.1%) | ** | ** | ** | ** | ** |
| Any use of 1st generation sulfonylureas; n (%) | 4 (0.0%) | 1 (0.0%) | 2 (0.0%) | 1 (0.0%) | ** | ** | ** | ** | ** |
| Entresto (sacubitril/valsartan); n (%) | 12 (0.1%) | 25 (0.3%) | 8 (0.1%) | 6 (0.1%) | 29 (0.1%) | 40 (0.1%) | 049 (0.1%) | 071 (0.1%) | 0.00 |
| Labs | | | | | | | 17,596 | 17,596 | |
| Lab values- HbA1c (%); n (%) | 3,567 (40.2%) | 3,619 (40.8%) | 591 (6.8%) | 410 (4.7%) | N/A | N/A | 4,158 (23.6%) | 4,029 (22.9%) | 0.02 |
| Lab values- HbA1c (%) (within 3 months); n (%) | 2,757 (31.0%) | 2,895 (32.6%) | 460 (5.3%) | 333 (3.8%) | N/A | N/A | 3,217 (18.3%) | 3,228 (18.3%) | 0.00 |
| Lab values- HbA1c (%) (within 6 months); n (%) | 3,567 (40.2%) | 3,619 (40.8%) | 591 (6.8%) | 410 (4.7%) | N/A | N/A | 4,158 (23.6%) | 4,029 (22.9%) | 0.02 |
| Lab values- BNP; n (%) | 75 (0.8%) | 116 (1.3%) | 9 (0.1%) | 11 (0.1%) | N/A | N/A | 084 (0.5%) | 127 (0.7%) | -0.03 |
| Lab values- BNP (within 3 months); n (%) | 54 (0.6%) | 66 (0.7%) | 5 (0.1%) | 8 (0.1%) | N/A | N/A | 059 (0.3%) | 074 (0.4%) | -0.02 |
| Lab values- BNP (within 6 months); n (%) | 75 (0.8%) | 116 (1.3%) | 9 (0.1%) | 11 (0.1%) | N/A | N/A | 084 (0.5%) | 127 (0.7%) | -0.03 |
| Lab values- BUN (mg/dl); n (%) | 3,723 (41.9%) | 3,839 (43.2%) | 534 (6.1%) | 459 (5.3%) | N/A | N/A | 4,257 (24.2%) | 4,298 (24.4%) | 0.00 |

| Lab values- BUN (mg/dl) (within 3 months); n (%) | 2,904 (32.7%) | 3,046 (34.3%) | 411 (4.7%) | 361 (4.1%) | N/A | N/A | 3,315 (18.8%) | 3,407 (19.4%) | -0.02 |
|---|---|---|---|---|---|---|---|---|---|
| Lab values- BUN (mg/dl) (within 6 months); n (%) | 3,723 (41.9%) | 3,839 (43.2%) | 534 (6.1%) | 459 (5.3%) | N/A | N/A | 4,257 (24.2%) | 4,298 (24.4%) | 0.00 |
| Lab values- Creatinine (mg/dl); n (%) | 3,814 (43.0%) | 3,958 (44.6%) | 567 (6.5%) | 500 (5.7%) | N/A | N/A | 4,381 (24.9%) | 4,458 (25.3%) | -0.01 |
| | 3,014 (43.070) | 3,556 (44.070) | 307 (0.370) | 300 (3.770) | 14/5 | 14/15 | 4,501 (24.570) | 4,430 (23.370) | 0.01 |
| Lab values- Creatinine (mg/dl) (within 3 months); n | | | | | | | | | |
| (%) | 2,972 (33.5%) | 3,146 (35.4%) | 436 (5.0%) | 391 (4.5%) | N/A | N/A | 3,408 (19.4%) | 3,537 (20.1%) | -0.02 |
| Lab values- Creatinine (mg/dl) (within 6 months); n | | | | | | | | | |
| (%) | 3,814 (43.0%) | 3,958 (44.6%) | 567 (6.5%) | 500 (5.7%) | N/A | N/A | 4,381 (24.9%) | 4,458 (25.3%) | -0.01 |
| Lab values- HDL level (mg/dl); n (%) | 2,999 (33.8%) | 3,087 (34.8%) | 502 (5.8%) | 397 (4.6%) | N/A | N/A | 3,501 (19.9%) | 3,484 (19.8%) | 0.00 |
| Lab values-TIDE level (Hig/GI), II (70) | 2,333 (33.8%) | 3,087 (34.8%) | 302 (3.8%) | 397 (4.0%) | IN/A | IN/A | 3,301 (19.9%) | 3,484 (13.876) | 0.00 |
| Lab values- HDL level (mg/dl) (within 3 months); n (%) | 2,179 (24.5%) | 2,308 (26.0%) | 362 (4.2%) | 306 (3.5%) | N/A | N/A | 2,541 (14.4%) | 2,614 (14.9%) | -0.01 |
| Lab values- HDL level (mg/dl) (within 6 months); n (%) | 2,999 (33.8%) | 3,087 (34.8%) | 502 (5.8%) | 397 (4.6%) | N/A | N/A | 3,501 (19.9%) | 3,484 (19.8%) | 0.00 |
| Lab values-LDL level (mg/dl); n (%) | 3,088 (34.8%) | 3,177 (35.8%) | 528 (6.1%) | 402 (4.6%) | N/A | N/A | 3,616 (20.6%) | 3,579 (20.3%) | 0.01 |
| Edb values EDE level (IIIg/al/, II (70) | 3,000 (34.0%) | 3,177 (33.670) | 320 (0.170) | 402 (4.0%) | 14/5 | 14/15 | 3,010 (20.070) | 3,373 (20.370) | 0.01 |
| | | | | /// | | | | | |
| Lab values- LDL level (mg/dl) (within 3 months); n (%) | 2,230 (25.1%) | 2,379 (26.8%) | 374 (4.3%) | 309 (3.5%) | N/A | N/A | 2,604 (14.8%) | 2,688 (15.3%) | -0.01 |
| Lab values- LDL level (mg/dl) (within 6 months); n (%) | 3,088 (34.8%) | 3,177 (35.8%) | 528 (6.1%) | 402 (4.6%) | N/A | N/A | 3,616 (20.6%) | 3,579 (20.3%) | 0.01 |
| Lab values- NT-proBNP; n (%) | 15 (0.2%) | 12 (0.1%) | 0 (0.0%) | 2 (0.0%) | N/A | N/A | 15 (0.1%) | 0 (0.1%) | _ |
| Lab values- NT-proBNP (within 3 months); n (%) | 10 (0.1%) | | 0 (0.0%) | 1 (0.0%) | N/A | N/A | 10 (0.1%) | 0 (0.0%) | |
| | | 6 (0.1%) | | | | | | | |
| Lab values- NT-proBNP (within 6 months); n (%) | 15 (0.2%) | 12 (0.1%) | 0 (0.0%) | 2 (0.0%) | N/A | N/A | 15 (0.1%) | 14 (0.1%) | - |
| Lab values-Total cholesterol (mg/dl); n (%) | 3,051 (34.4%) | 3,149 (35.5%) | 505 (5.8%) | 404 (4.6%) | N/A | N/A | 3,556 (20.2%) | 3,553 (20.2%) | 0.00 |
| Lab values-Total cholesterol (mg/dl) (within 3 | | | | | | | | | |
| months); n (%) | 2,212 (24.9%) | 2,352 (26.5%) | 361 (4.1%) | 311 (3.6%) | N/A | N/A | 2,573 (14.6%) | 2,663 (15.1%) | -0.01 |
| ** * * | 2,212 (24.576) | 2,332 (20.376) | 301 (4.176) | 311 (3.0%) | IN/A | IN/A | 2,373 (14.0%) | 2,003 (13.176) | -0.01 |
| Lab values-Total cholesterol (mg/dl) (within 6 | | | | | | | | | |
| months); n (%) | 3,051 (34.4%) | 3,149 (35.5%) | 505 (5.8%) | 404 (4.6%) | N/A | N/A | 3,556 (20.2%) | 3,553 (20.2%) | 0.00 |
| Lab values-Triglyceride level (mg/dl); n (%) | 3,015 (34.0%) | 3,135 (35.3%) | 500 (5.7%) | 399 (4.6%) | N/A | N/A | 3,515 (20.0%) | 3,534 (20.1%) | 0.00 |
| Lab values- Triglyceride level (mg/dl) (within 3 | | | | | | | | | |
| months); n (%) | 2,190 (24.7%) | 2,341 (26.4%) | 355 (4.1%) | 306 (3.5%) | N/A | N/A | 2,545 (14.5%) | 2,647 (15.0%) | -0.01 |
| | 2,190 (24.7%) | 2,341 (20.4%) | 333 (4.1%) | 300 (3.3%) | N/A | IN/A | 2,343 (14.3%) | 2,647 (13.0%) | -0.01 |
| Lab values- Triglyceride level (mg/dl) (within 6 | | | | | | | | | |
| months); n (%) | 3,015 (34.0%) | 3,135 (35.3%) | 500 (5.7%) | 399 (4.6%) | N/A | N/A | 3,515 (20.0%) | 3,534 (20.1%) | 0.00 |
| Lab result number- HbA1c (%) mean (only 2 to 20 | | | | | | | | | |
| included) | 3,541 | 3,606 | 529 | 389 | N/A | N/A | 4,070 | 3,995 | |
| | 8.14 (1.86) | 8.00 (1.81) | 8.11 (1.85) | 7.88 (1.83) | N/A | N/A | 8.14 (1.86) | 7.99 (1.81) | 0.08 |
| mean (sd) | | | | | | | | | |
| median [IQR] | 7.70 [6.85, 9.04] | 7.60 [6.70, 8.80] | 7.60 [6.80, 9.00] | 7.45 [6.60, 8.60] | N/A | N/A | 7.69 (1.86) | 7.59 (1.81) | 0.05 |
| Missing; n (%) | 5,339 (60.1%) | 5,274 (59.4%) | 8,187 (93.9%) | 8,327 (95.5%) | N/A | N/A | 13,526 (76.9%) | 13,601 (77.3%) | -0.01 |
| Lab result number- BNP mean | 75 | 116 | 9 | 11 | N/A | N/A | 84 | 127 | |
| mean (sd) | 182.81 (288.14) | 199.85 (371.31) | 209.22 (333.71) | 607.19 (1,393.52) | N/A | N/A | 185.64 (294.70) | 235.13 (533.36) | -0.11 |
| | 102.01 (200.14) | | | | | | | | |
| | | | | | | | ` | | |
| median [IQR] | 65.50 [32.60, 167.50] | 82.60 [32.35, 208.35] | 80.00 [47.00, 204.50] | 49.00 [15.10, 188.00] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| median [IQR]<br>Missing; n (%) | | 82.60 [32.35, 208.35]<br>8,764 (98.7%) | | | | | #VALUE!<br>17,512 (99.5%) | | |
| Missing; n (%) | 65.50 [32.60, 167.50] | | 80.00 [47.00, 204.50] | 49.00 [15.10, 188.00] | N/A | N/A | | #VALUE! | #VALUE! |
| Missing; n (%)<br>Lab result number-BUN (mg/dl) mean | 65.50 [32.60, 167.50]<br>8,805 (99.2%)<br>3,723 | 8,764 (98.7%)<br>3,839 | 80.00 [47.00, 204.50]<br>8,707 (99.9%)<br>534 | 49.00 [15.10, 188.00]<br>8,705 (99.9%)<br>459 | N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A | 17,512 (99.5%)<br><mark>4,257</mark> | #VALUE!<br>17,469 (99.3%)<br>4,298 | #VALUE!<br>0.03 |
| Missing; n (%)<br>Lab result number-BUN (mg/dl) mean<br>mean (sd) | 65.50 [32.60, 167.50]<br>8,805 (99.2%)<br>3,723<br>21.39 (9.92) | 8,764 (98.7%)<br>3,839<br>22.02 (10.30) | 80.00 [47.00, 204.50]<br>8,707 (99.9%)<br>534<br>550.42 (9,028.78) | 49.00 [15.10, 188.00]<br>8,705 (99.9%)<br>459<br>306.80 (6,067.08) | N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A | 17,512 (99.5%)<br><mark>4,257</mark><br>87.75 (3195.92) | #VALUE!<br>17,469 (99.3%)<br>4,298<br>52.43 (1981.24) | #VALUE!<br>0.03<br>0.01 |
| Missing; n (%)<br>Lab result number- BUN (mg/dl) mean<br>mean (sd)<br>median [IQR] | 65.50 [32.60, 167.50]<br>8,805 (99.2%)<br>3,723<br>21.39 (9.92)<br>19.00 [15.00, 25.50] | 8,764 (98.7%) 3,839 22.02 (10.30) 19.50 [15.00, 27.00] | 80.00 [47.00, 204.50]<br>8,707 (99.9%)<br>534<br>550.42 (9,028.78)<br>18.00 [13.50, 24.00] | 49.00 [15.10, 188.00]<br>8,705 (99.9%)<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00] | N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A | 17,512 (99.5%)<br>4,257<br>87.75 (3195.92)<br>#VALUE! | #VALUE!<br>17,469 (99.3%)<br>4,298<br>52.43 (1981.24)<br>#VALUE! | #VALUE!<br>0.03<br>0.01<br>#VALUE! |
| Missing; n (%)<br>Lab result number-BUN (mg/dl) mean<br>mean (sd) | 65.50 [32.60, 167.50]<br>8,805 (99.2%)<br>3,723<br>21.39 (9.92) | 8,764 (98.7%)<br>3,839<br>22.02 (10.30) | 80.00 [47.00, 204.50]<br>8,707 (99.9%)<br>534<br>550.42 (9,028.78) | 49.00 [15.10, 188.00]<br>8,705 (99.9%)<br>459<br>306.80 (6,067.08) | N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A | 17,512 (99.5%)<br><mark>4,257</mark><br>87.75 (3195.92) | #VALUE!<br>17,469 (99.3%)<br>4,298<br>52.43 (1981.24) | #VALUE!<br>0.03<br>0.01 |
| Missing; n (%)<br>Lab result number- BUN (mg/dl) mean<br>mean (sd)<br>median [IQR] | 65.50 [32.60, 167.50]<br>8,805 (99.2%)<br>3,723<br>21.39 (9.92)<br>19.00 [15.00, 25.50] | 8,764 (98.7%) 3,839 22.02 (10.30) 19.50 [15.00, 27.00] | 80.00 [47.00, 204.50]<br>8,707 (99.9%)<br>534<br>550.42 (9,028.78)<br>18.00 [13.50, 24.00] | 49.00 [15.10, 188.00]<br>8,705 (99.9%)<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00] | N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A | 17,512 (99.5%)<br>4,257<br>87.75 (3195.92)<br>#VALUE! | #VALUE!<br>17,469 (99.3%)<br>4,298<br>52.43 (1981.24)<br>#VALUE! | #VALUE!<br>0.03<br>0.01<br>#VALUE! |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 | 65.50 [32.60, 167.50]<br>8,805 (99.2%)<br>3,723<br>21.39 (9.92)<br>19.00 [15.00, 25.50]<br>5,157 (58.1%) | 8,764 (98.7%)<br>3,839<br>22.02 (10.30)<br>19.50 [15.00, 27.00]<br>5,041 (56.8%) | 80.00 [47.00, 204.50]<br>8,707 (99.9%)<br>534<br>550.42 (9,028.78)<br>18.00 [13.50, 24.00]<br>8,182 (93.9%) | 49.00 [15.10, 188.00]<br>8,705 (99.9%)<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 (94.7%) | N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A | 17,512 (99.5%)<br>4,257<br>87.75 (3195.92)<br>#VALUE!<br>13,339 (75.8%) | #VALUE!<br>17,469 (99.3%)<br>4,298<br>52.43 (1981.24)<br>#VALUE!<br>13,298 (75.6%) | #VALUE!<br>0.03<br>0.01<br>#VALUE! |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included) | 65.50 [32.60, 167.50]<br>8,805 [99.2%)<br>3,723<br>21.39 [9.92)<br>19.00 [15.00, 25.50]<br>5,157 (58.1%)<br>3,791 | 8,764 (98.7%)<br>3,839<br>22.02 (10.30)<br>19.50 [15.00, 27.00]<br>5,041 (56.8%) | 80.00 [47.00, 204.50]<br>8,707 (99.9%)<br>534<br>550.42 (9,028.78)<br>18.00 [13.50, 24.00]<br>8,182 (93.9%) | 49.00 [15.10, 188.00]<br>8,705 [99.9%]<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 [94.7%] | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) #VALUE! 13,339 (75.8%) 4,311 | #VALUE!<br>17,469 (99.3%)<br>4,298<br>52.43 (1981.24)<br>#VALUE!<br>13,298 (75.6%)<br>4,404 | #VALUE!<br>0.03<br>0.01<br>#VALUE!<br>0.00 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd) | 65.50 [32.60, 167.50]<br>8,805 [99.2%]<br>3,723<br>21.39 [9.92)<br>19.00 [15.00, 25.50]<br>5,157 (58.1%)<br>3,791<br>1.20 (0.50) | 8,764 (98.7%)<br>3,839<br>22.02 (10.30)<br>19.50 (15.00, 27.00)<br>5,041 (56.8%)<br>3,936<br>1.24 (0.51) | 80.00 [47.00, 204.50]<br>8,707 [99.9%]<br>534<br>550.42 [9,028.78]<br>18.00 [13.50, 24.00]<br>8,182 [93.9%]<br>520<br>1.15 [0.52] | 49.00 [15.10, 188.00]<br>8,705 (99.9%)<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 (94.7%)<br>468<br>1.18 (0.61) | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) #VALUEI 13,339 (75.8%) 4,311 1.19 (0.50) | #VALUEI<br>17,469 (99.3%)<br>4,298<br>52.43 (1981.24)<br>#VALUEI<br>13,298 (75.6%)<br>4,404<br>1.23 (0.52) | #VALUE!<br>0.03<br>0.01<br>#VALUE!<br>0.00 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR] | 65.50 [32.60, 167.50]<br>8,805 [99.2%]<br>3,723<br>21.39 [9.92)<br>19.00 [15.00, 25.50]<br>5,157 (58.1%)<br>3,791<br>1.20 [0.50]<br>1.08 [0.87, 1.41] | 8,764 (98.7%)<br>3,839<br>22.02 (10.30)<br>19.50 (15.00, 27.00)<br>5,041 (56.8%)<br>3,936<br>1.24 (0.51)<br>1.14 [0.88, 1.48] | 80.00 [47.00, 204.50]<br>8,707 [99.9%]<br>534<br>550.42 (9,028.78)<br>18.00 [13.50, 24.00]<br>8,182 (93.9%)<br>520<br>1.15 (0.52)<br>1.00 [0.84, 1.36] | 49.00 [15.10, 188.00]<br>8,705 (99.9%)<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 (94.7%)<br>468<br>1.18 (0.61)<br>1.01 [0.84, 1.35] | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) 74,410E 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) | #VALUEI<br>17,469 (99.3%)<br>4,298<br>52.43 (1981.24)<br>#VALUEI<br>13,298 (75.6%)<br>4,404<br>1.23 (0.52)<br>1.13 (0.52) | #VALUE!<br>0.03<br>0.01<br>#VALUE!<br>0.00<br>-0.08<br>-0.12 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd) | 65.50 [32.60, 167.50]<br>8,805 [99.2%]<br>3,723<br>21.39 [9.92)<br>19.00 [15.00, 25.50]<br>5,157 (58.1%)<br>3,791<br>1.20 (0.50) | 8,764 (98.7%)<br>3,839<br>22.02 (10.30)<br>19.50 (15.00, 27.00)<br>5,041 (56.8%)<br>3,936<br>1.24 (0.51) | 80.00 [47.00, 204.50]<br>8,707 [99.9%]<br>534<br>550.42 [9,028.78]<br>18.00 [13.50, 24.00]<br>8,182 [93.9%]<br>520<br>1.15 [0.52] | 49.00 [15.10, 188.00]<br>8,705 (99.9%)<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 (94.7%)<br>468<br>1.18 (0.61) | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) #VALUEI 13,339 (75.8%) 4,311 1.19 (0.50) | #VALUEI<br>17,469 (99.3%)<br>4,298<br>52.43 (1981.24)<br>#VALUEI<br>13,298 (75.6%)<br>4,404<br>1.23 (0.52) | #VALUE!<br>0.03<br>0.01<br>#VALUE!<br>0.00 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) | 65.50 [32.60, 167.50]<br>8,805 [99.2%]<br>3,723<br>21.39 [9.92)<br>19.00 [15.00, 25.50]<br>5,157 (58.1%)<br>3,791<br>1.20 [0.50]<br>1.08 [0.87, 1.41] | 8,764 (98.7%)<br>3,839<br>22.02 (10.30)<br>19.50 (15.00, 27.00)<br>5,041 (56.8%)<br>3,936<br>1.24 (0.51)<br>1.14 [0.88, 1.48] | 80.00 [47.00, 204.50]<br>8,707 [99.9%]<br>534<br>550.42 (9,028.78)<br>18.00 [13.50, 24.00]<br>8,182 (93.9%)<br>520<br>1.15 (0.52)<br>1.00 [0.84, 1.36] | 49.00 [15.10, 188.00]<br>8,705 (99.9%)<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 (94.7%)<br>468<br>1.18 (0.61)<br>1.01 [0.84, 1.35] | N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) 74,410E 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) | #VALUEI<br>17,469 (99.3%)<br>4,298<br>52.43 (1981.24)<br>#VALUEI<br>13,298 (75.6%)<br>4,404<br>1.23 (0.52)<br>1.13 (0.52) | #VALUE!<br>0.03<br>0.01<br>#VALUE!<br>0.00<br>-0.08<br>-0.12 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only | 65.50 [32.60, 167.50]<br>8,805 [99.2%]<br>3,723<br>21.39 [9.92)<br>19.00 [15.00, 25.50]<br>5,157 [58.1%]<br>3,791<br>1.20 [0.50)<br>1.08 [0.87, 1.41]<br>5,089 [57.3%] | 8,764 (98.7%)<br>3,839<br>22.02 (10.30)<br>19.50 (15.00, 27.00)<br>5,041 (56.8%)<br>3,936<br>1.24 (0.51)<br>1.14 [0.88, 1.48]<br>4,944 (55.7%) | 80.00 [47.00, 204.50]<br>8,707 [99.9%)<br>534<br>550.42 (9,028.78)<br>18.00 [13.50, 24.00]<br>8,182 (93.9%)<br>520<br>1.15 (0.52)<br>1.00 [0.84, 1.36]<br>8,196 (94.0%) | 49.00 [15.10, 188.00]<br>8,705 [99.9%]<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 [94.7%]<br>468<br>1.18 (0.61)<br>1.01 [0.84, 1.35]<br>8,248 (94.6%) | N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) #VALUEI 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) 13,285 (75.5%) | #VALUEI 17,469 (99.3%) 4,298 52.43 (1981.24) #VALUEI 13,298 (75.6%) 4,404 1.23 (0.52) 1.13 (0.52) 13,192 (75.0%) | #VALUE!<br>0.03<br>0.01<br>#VALUE!<br>0.00<br>-0.08<br>-0.12 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only e | 65.50 [32.60, 167.50]<br>8,805 [99.2%]<br>3,723<br>21.39 [9.92)<br>19.00 [15.00, 25.50]<br>5,157 (58.1%)<br>3,791<br>1.20 (0.50)<br>1.08 [0.87, 1.41]<br>5,089 (57.3%) | 8,764 (98.7%)<br>3,839<br>22.02 (10.30)<br>19.50 (15.00, 27.00)<br>5,041 (56.8%)<br>3,936<br>1.24 (0.51)<br>1.14 [0.88, 1.48]<br>4,944 (55.7%) | 80.00 [47.00, 204.50]<br>8,707 [99.9%)<br>534<br>550.42 [9,028.78]<br>18.00 [13.50, 24.00]<br>8,182 [93.9%)<br>520<br>1.15 [0.52)<br>1.00 [0.84, 1.36]<br>8,196 [94.0%) | 49.00 [15.10, 188.00]<br>8,705 (99.9%)<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 (94.7%)<br>468<br>1.18 (0.61)<br>1.01 [0.84, 1.35]<br>8,248 (94.6%) | N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) #VALUEI 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) 13,285 (75.5%) | #VALUEI 17,469 (99.3%) 4,298 52.43 (1981.24) #VALUEI 13,298 (75.6%) 4,404 1.23 (0.52) 1.13 (0.52) 13,192 (75.0%) 3,483 | #VALUE! 0.03 0.01 #VALUE! 0.00 -0.08 -0.12 0.01 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only 9.1 to 15 included)mean (sd) | 65.50 [32.60, 167.50]<br>8,805 [99.2%]<br>3,723<br>21.39 [9.92)<br>19.00 [15.00, 25.50]<br>5,157 (58.1%)<br>3,791<br>1.20 (0.50)<br>1.08 [0.87, 1.41]<br>5,089 (57.3%)<br>2,999<br>45.64 (13.89) | 8,764 (98.7%)<br>3,839<br>22.02 (10.30)<br>19.50 (15.00, 27.00)<br>5,041 (56.8%)<br>3,936<br>1.24 (0.51)<br>1.14 [0.88, 1.48]<br>4,944 (55.7%)<br>3,087<br>46.51 (14.12) | 80.00 [47.00, 204.50]<br>8,707 [99.9%)<br>534<br>550.42 (9,028.78)<br>18.00 [13.50, 24.00]<br>8,182 (93.9%)<br>520<br>1.15 (0.52)<br>1.00 [0.84, 1.36]<br>8,196 (94.0%)<br>501<br>43.93 (15.31) | 49.00 [15.10, 188.00]<br>8,705 (99.9%)<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 (94.7%)<br>468<br>1.18 (0.61)<br>1.01 [0.84, 1.35]<br>8,248 (94.6%)<br>396<br>51.64 (174.45) | N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) #VALUEI 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) 13,285 (75.5%) 3,500 45.40 (14.10) | #VALUEI 17,469 (99.3%) 4,298 52.43 (1981.24) #VALUEI 13,298 (75.6%) 4,404 1.23 (0.52) 1.13 (0.52) 13,192 (75.0%) 3,483 47.09 (60.26) | #VALUE! 0.03 0.01 #VALUE! 0.00 -0.08 -0.12 0.01 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only e | 65.50 [32.60, 167.50]<br>8,805 [99.2%]<br>3,723<br>21.39 [9.92)<br>19.00 [15.00, 25.50]<br>5,157 (58.1%)<br>3,791<br>1.20 (0.50)<br>1.08 [0.87, 1.41]<br>5,089 (57.3%) | 8,764 (98.7%)<br>3,839<br>22.02 (10.30)<br>19.50 (15.00, 27.00)<br>5,041 (56.8%)<br>3,936<br>1.24 (0.51)<br>1.14 [0.88, 1.48]<br>4,944 (55.7%) | 80.00 [47.00, 204.50]<br>8,707 [99.9%)<br>534<br>550.42 [9,028.78]<br>18.00 [13.50, 24.00]<br>8,182 [93.9%)<br>520<br>1.15 [0.52)<br>1.00 [0.84, 1.36]<br>8,196 [94.0%) | 49.00 [15.10, 188.00]<br>8,705 (99.9%)<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 (94.7%)<br>468<br>1.18 (0.61)<br>1.01 [0.84, 1.35]<br>8,248 (94.6%) | N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) #VALUEI 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) 13,285 (75.5%) | #VALUEI 17,469 (99.3%) 4,298 52.43 (1981.24) #VALUEI 13,298 (75.6%) 4,404 1.23 (0.52) 1.13 (0.52) 13,192 (75.0%) 3,483 | #VALUE! 0.03 0.01 #VALUE! 0.00 -0.08 -0.12 0.01 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only 9.1 to 15 included)median [IQR]Missing; n (%) | 65.50 [32.60, 167.50]<br>8,805 [99.2%]<br>3,723<br>21.39 [9.92]<br>19.00 [15.00, 25.50]<br>5,157 (58.1%)<br>3,791<br>1.20 (0.50)<br>1.08 [0.87, 1.41]<br>5,089 (57.3%)<br>2,999<br>45.64 (13.89)<br>44.00 [36.00, 53.00] | 8,764 (98.7%) 3,839 22.02 (10.30) 19.50 (15.00, 27.00) 5,041 (56.8%) 3,936 1.24 (0.51) 1.14 [0.88, 1.48] 4,944 (55.7%) 3,087 46.51 (14.12) 44.50 [37.00, 54.00] | 80.00 [47.00, 204.50]<br>8,707 [99.9%)<br>534<br>550.42 [9.028.78]<br>18.00 [13.50, 24.00]<br>8,182 [93.9%)<br>520<br>1.15 [0.52)<br>1.00 [0.84, 1.36]<br>8,196 [94.0%)<br>501<br>43.93 [15.31]<br>42.50 [35.00, 52.00] | 49.00 [15.10, 188.00]<br>8,705 [99.9%]<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 [94.7%]<br>468<br>1.18 (0.61)<br>1.01 [0.84, 1.35]<br>8,248 [94.6%]<br>396<br>51.64 (174.45)<br>41.00 [34.00, 52.00] | N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) #WALUEI 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) 13,285 (75.5%) 3,500 45.40 (14.10) 43.79 (14.10) | #VALUEI 17,469 (99.3%) 4,298 52.43 (1981.24) #VALUEI 13,298 (75.6%) 4,404 1.23 (0.52) 1.13 (0.52) 13,192 (75.0%) 3,483 47.09 (60.26) 44.10 (60.26) | #VALUE! 0.03 0.01 #VALUE! 0.00 -0.08 -0.12 0.01 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only e<5000 included)mean (sd)mean (sd)mean (sd)mean [IQR] | 65.50 [32.60, 167.50]<br>8,805 [99.2%]<br>3,723<br>21.39 [9.92)<br>19.00 [15.00, 25.50]<br>5,157 (58.1%)<br>3,791<br>1.20 (0.50)<br>1.08 [0.87, 1.41]<br>5,089 (57.3%)<br>2,999<br>45.64 (13.89) | 8,764 (98.7%)<br>3,839<br>22.02 (10.30)<br>19.50 (15.00, 27.00)<br>5,041 (56.8%)<br>3,936<br>1.24 (0.51)<br>1.14 [0.88, 1.48]<br>4,944 (55.7%)<br>3,087<br>46.51 (14.12) | 80.00 [47.00, 204.50]<br>8,707 [99.9%)<br>534<br>550.42 (9,028.78)<br>18.00 [13.50, 24.00]<br>8,182 (93.9%)<br>520<br>1.15 (0.52)<br>1.00 [0.84, 1.36]<br>8,196 (94.0%)<br>501<br>43.93 (15.31) | 49.00 [15.10, 188.00]<br>8,705 (99.9%)<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 (94.7%)<br>468<br>1.18 (0.61)<br>1.01 [0.84, 1.35]<br>8,248 (94.6%)<br>396<br>51.64 (174.45) | N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) #VALUEI 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) 13,285 (75.5%) 3,500 45.40 (14.10) | #VALUEI 17,469 (99.3%) 4,298 52.43 (1981.24) #VALUEI 13,298 (75.6%) 4,404 1.23 (0.52) 1.13 (0.52) 13,192 (75.0%) 3,483 47.09 (60.26) | #VALUE! 0.03 0.01 #VALUE! 0.00 -0.08 -0.12 0.01 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only e<5000 included)mean (sd)median [IQR]median [IQR]median [IQR]median [IQR] | 65.50 [32.60, 167.50]<br>8,805 [99.2%]<br>3,723<br>21.39 [9.92)<br>19.00 [15.00, 25.50]<br>5,157 [58.1%]<br>3,791<br>1.20 (0.50)<br>1.08 [0.87, 1.41]<br>5,089 [57.3%)<br>2,999<br>45.64 [13.89]<br>44.00 [36.00, 53.00]<br>5,881 [66.2%] | 8,764 (98.7%) 3,839 22.02 (10.30) 19.50 (15.00, 27.00) 5,041 (56.8%) 3,936 1.24 (0.51) 1.14 [0.88, 1.48] 4,944 (55.7%) 3,087 46.51 (14.12) 44.50 [37.00, 54.00] 5,793 (65.2%) | 80.00 [47.00, 204.50]<br>8,707 [99.9%)<br>534<br>550.42 [9,028.78]<br>18.00 [13.50, 24.00]<br>8,182 [93.9%)<br>520<br>1.15 [0.52)<br>1.00 [0.84, 1.36]<br>8,196 [94.0%)<br>501<br>43.93 [15.31)<br>42.50 [35.00, 52.00]<br>8,215 [94.3%) | 49.00 [15.10, 188.00]<br>8,705 [99.9%]<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 (94.7%)<br>468<br>1.18 (0.61)<br>1.01 [0.84, 1.35]<br>8,248 (94.6%)<br>396<br>51.64 (174.45)<br>41.00 [34.00, 52.00]<br>8,320 (95.5%) | N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) #VALUEI 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) 13,285 (75.5%) 3,500 45.40 (14.10) 43.79 (14.10) 14,096 (80.1%) | #VALUEI 17,469 (99.3%) 4,298 52.43 (1981.24) #VALUEI 13,298 (75.6%) 4,404 1.23 (0.52) 1.13 (0.52) 1.3,192 (75.0%) 3,483 47.09 (60.26) 44.10 (60.26) 14,113 (80.2%) | #VALUE! 0.03 0.01 #VALUE! 0.00 -0.08 -0.12 0.01 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [lQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [lQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only <>5000 included)mean (sd)median [lQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only <>5000 included) | 65.50 (32.60, 167.50)<br>8,805 (99.2%)<br>3,723<br>21.39 (9.92)<br>19.00 [15.00, 25.50]<br>5,157 (58.1%)<br>3,791<br>1.20 (0.50)<br>1.08 [0.87, 1.41]<br>5,089 (57.3%)<br>2,999<br>45.64 (13.89)<br>44.00 [36.00, 53.00]<br>5,881 (66.2%) | 8,764 (98.7%) 3,839 22.02 (10.30) 19.50 (15.00, 27.00) 5,041 (56.8%) 3,936 1.24 (0.51) 1.14 [0.88, 1.48] 4,944 (55.7%) 3,087 46.51 (14.12) 44.50 [37.00, 54.00] 5,793 (65.2%) 3,106 | 80.00 [47.00, 204.50]<br>8,707 [99.9%)<br>534<br>550.42 (9.028.78)<br>18.00 [13.50, 24.00]<br>8,182 [93.9%)<br>520<br>1.15 (0.52)<br>1.00 [0.84, 1.36]<br>8,196 [94.0%)<br>501<br>43.93 (15.31)<br>42.50 [35.00, 52.00]<br>8,215 [94.3%) | 49.00 [15.10, 188.00]<br>8,705 [99.9%]<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 [94.7%]<br>468<br>1.18 (0.61)<br>1.01 [0.84, 1.35]<br>8,248 [94.6%]<br>396<br>51.64 (174.45)<br>41.00 [34.00,52.00]<br>8,320 [95.5%] | N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) 47ALUEI 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) 13,285 (75.5%) 3,500 45.40 (14.10) 43.79 (14.10) 14,096 (80.1%) | #VALUEI 17,469 (99.3%) 4,298 52.43 (1981.24) #VALUEI 13,298 (75.6%) 4,404 1.23 (0.52) 1.13 (0.52) 1.3192 (75.0%) 3,483 47.09 (60.26) 44.10 (60.26) 14,113 (80.2%) 3,482 | #VALUE! 0.03 0.01 #VALUE! 0.00 -0.08 -0.12 0.01 -0.04 -0.04 -0.01 0.00 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number- Creatinine (mg/dl) mean (only 0.1 to 15 included)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)mean (sd)mean (sd)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)median [IQR] | 65.50 [32.60, 167.50]<br>8,805 [99.2%]<br>3,723<br>21.39 [9.92]<br>19.00 [15.00, 25.50]<br>5,157 [58.1%]<br>3,791<br>1.20 [0.50]<br>1.08 [0.87, 1.41]<br>5,089 [57.3%]<br>2,999<br>45.64 (13.89)<br>44.00 [36.00, 53.00]<br>5,881 (66.2%)<br>3,014<br>85.21 (41.48) | 8,764 (98.7%) 3,839 22.02 (10.30) 19.50 (15.00, 27.00) 5,041 (56.8%) 3,936 1.24 (0.51) 1.14 [0.88, 1.48] 4,944 (55.7%) 3,087 46.51 (14.12) 44.50 (37.00, 54.00) 5,793 (65.2%) 3,106 85.59 (40.41) | 80.00 [47.00, 204.50]<br>8,707 [99.9%)<br>534<br>550.42 (9.028.78)<br>18.00 [13.50, 24.00]<br>8,182 [93.9%)<br>520<br>1.15 [0.52)<br>1.00 [0.84, 1.36]<br>8,196 [94.0%)<br>501<br>43.93 [15.31)<br>42.50 [35.00, 52.00]<br>8,215 [94.3%)<br>481<br>86.93 (43.78) | 49.00 [15.10, 188.00]<br>8,705 [99.9%]<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 [94.7%]<br>468<br>1.18 [0.61]<br>1.01 [0.84, 1.35]<br>8,248 [94.6%]<br>396<br>51.64 (174.45)<br>41.00 [34.00, 52.00]<br>8,320 [95.5%]<br>376<br>85.05 (45.50) | N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) #VALUEI 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) 13,285 (75.5%) 3,500 45.40 (14.10) 43.79 (14.10) 14,096 (80.1%) 3,495 85.45 (41.81) | #VALUEI 17,469 (99.3%) 4,298 52.43 (1981.24) #VALUEI 13,298 (75.6%) 4,404 1.23 (0.52) 1.13 (0.52) 13,192 (75.0%) 3,483 47.09 (60.26) 44.10 (60.26) 14,113 (80.2%) 3,482 85.53 (40.99) | #VALUE! 0.03 0.01 #VALUE! 0.00 -0.08 -0.12 0.01 -0.04 -0.01 0.00 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [lQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [lQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only <>5000 included)mean (sd)median [lQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only <>5000 included) | 65.50 (32.60, 167.50)<br>8,805 (99.2%)<br>3,723<br>21.39 (9.92)<br>19.00 [15.00, 25.50]<br>5,157 (58.1%)<br>3,791<br>1.20 (0.50)<br>1.08 [0.87, 1.41]<br>5,089 (57.3%)<br>2,999<br>45.64 (13.89)<br>44.00 [36.00, 53.00]<br>5,881 (66.2%) | 8,764 (98.7%) 3,839 22.02 (10.30) 19.50 (15.00, 27.00) 5,041 (56.8%) 3,936 1.24 (0.51) 1.14 [0.88, 1.48] 4,944 (55.7%) 3,087 46.51 (14.12) 44.50 [37.00, 54.00] 5,793 (65.2%) 3,106 | 80.00 [47.00, 204.50]<br>8,707 [99.9%)<br>534<br>550.42 (9.028.78)<br>18.00 [13.50, 24.00]<br>8,182 [93.9%)<br>520<br>1.15 (0.52)<br>1.00 [0.84, 1.36]<br>8,196 [94.0%)<br>501<br>43.93 (15.31)<br>42.50 [35.00, 52.00]<br>8,215 [94.3%) | 49.00 [15.10, 188.00]<br>8,705 [99.9%]<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 [94.7%]<br>468<br>1.18 (0.61)<br>1.01 [0.84, 1.35]<br>8,248 [94.6%]<br>396<br>51.64 (174.45)<br>41.00 [34.00,52.00]<br>8,320 [95.5%] | N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) #VALUEI 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) 13,285 (75.5%) 3,500 45.40 (14.10) 43.79 (14.10) 14,096 (80.1%) 3,495 85.45 (41.81) 82.20 (41.81) | #VALUEI 17,469 (99.3%) 4,298 52.43 (1981.24) #VALUEI 13,298 (75.6%) 4,404 1.23 (0.52) 1.13 (0.52) 13,192 (75.0%) 3,483 47.09 (60.26) 44.10 (60.26) 14,113 (80.2%) 3,482 85.53 (40.99) 82.94 (40.99) | #VALUE! 0.03 0.01 #VALUE! 0.00 -0.08 -0.12 -0.01 -0.04 -0.01 -0.00 -0.00 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number- Creatinine (mg/dl) mean (only 0.1 to 15 included)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)mean (sd)mean (sd)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)median [IQR] | 65.50 [32.60, 167.50]<br>8,805 [99.2%]<br>3,723<br>21.39 [9.92]<br>19.00 [15.00, 25.50]<br>5,157 [58.1%]<br>3,791<br>1.20 [0.50]<br>1.08 [0.87, 1.41]<br>5,089 [57.3%]<br>2,999<br>45.64 (13.89)<br>44.00 [36.00, 53.00]<br>5,881 (66.2%)<br>3,014<br>85.21 (41.48) | 8,764 (98.7%) 3,839 22.02 (10.30) 19.50 (15.00, 27.00) 5,041 (56.8%) 3,936 1.24 (0.51) 1.14 [0.88, 1.48] 4,944 (55.7%) 3,087 46.51 (14.12) 44.50 (37.00, 54.00) 5,793 (65.2%) 3,106 85.59 (40.41) | 80.00 [47.00, 204.50]<br>8,707 [99.9%)<br>554<br>550.42 (9.028.78)<br>18.00 [13.50, 24.00]<br>8,182 [93.9%)<br>520<br>1.15 (0.52)<br>1.00 [0.84, 1.36]<br>8,196 (94.0%)<br>501<br>43.93 [15.31)<br>42.50 [35.00, 52.00]<br>8,215 [94.3%)<br>481<br>86.93 (43.78)<br>85.00 [62.00, 109.58] | 49.00 [15.10, 188.00]<br>8,705 [99.9%]<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 [94.7%]<br>468<br>1.18 [0.61]<br>1.01 [0.84, 1.35]<br>8,248 [94.6%]<br>396<br>51.64 (174.45)<br>41.00 [34.00, 52.00]<br>8,320 [95.5%]<br>376<br>85.05 (45.50) | N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) #VALUEI 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) 13,285 (75.5%) 3,500 45.40 (14.10) 43.79 (14.10) 14,096 (80.1%) 3,495 85.45 (41.81) | #VALUEI 17,469 (99.3%) 4,298 52.43 (1981.24) #VALUEI 13,298 (75.6%) 4,404 1.23 (0.52) 1.13 (0.52) 13,192 (75.0%) 3,483 47.09 (60.26) 44.10 (60.26) 14,113 (80.2%) 3,482 85.53 (40.99) | #VALUE! 0.03 0.01 #VALUE! 0.00 -0.08 -0.12 0.01 -0.04 -0.01 0.00 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only <>5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only <>5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only <>5000 included)mean (sd)mean (sd)median [IQR]Missing; n (%) | 65.50 [32.60, 167.50]<br>8,805 [99.2%]<br>3,723<br>21.39 [9.92)<br>19.00 [15.00, 25.50]<br>5,157 [58.1%]<br>3,791<br>1.20 [0.50)<br>1.08 [0.87, 1.41]<br>5,089 [57.3%)<br>2,999<br>45.64 [13.89]<br>44.00 [36.00, 53.00]<br>5,881 [66.2%]<br>3,014<br>85.21 [41.48]<br>81.75 [60.00, 108.00] | 8,764 (98.7%) 3,839 22.02 (10.30) 19.50 (15.00, 27.00) 5,041 (56.8%) 3,936 1.24 (0.51) 1.14 [0.88, 1.48] 4,944 (55.7%) 3,087 46.51 (14.12) 44.50 [37.00, 54.00] 5,793 (65.2%) 3,106 85.59 (40.41) 82.75 [61.00, 109.00] | 80.00 [47.00, 204.50]<br>8,707 [99.9%)<br>534<br>550.42 (9.028.78)<br>18.00 [13.50, 24.00]<br>8,182 [93.9%)<br>520<br>1.15 [0.52)<br>1.00 [0.84, 1.36]<br>8,196 [94.0%)<br>501<br>43.93 [15.31)<br>42.50 [35.00, 52.00]<br>8,215 [94.3%)<br>481<br>86.93 (43.78) | 49.00 [15.10, 188.00]<br>8,705 [99.9%]<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 [94.7%]<br>468<br>1.18 (0.61)<br>1.01 [0.84, 1.35]<br>8,248 [94.6%]<br>396<br>51.64 (174.45)<br>41.00 [34.00, 52.00]<br>8,320 [95.5%]<br>376<br>85.05 [45.50]<br>84.50 [59.00, 111.38] | N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) #VALUEI 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) 13,285 (75.5%) 3,500 45.40 (14.10) 43.79 (14.10) 14,096 (80.1%) 3,495 85.45 (41.81) 82.20 (41.81) | #VALUEI 17,469 (99.3%) 4,298 52.43 (1981.24) #VALUEI 13,298 (75.6%) 4,404 1.23 (0.52) 1.13 (0.52) 13,192 (75.0%) 3,483 47.09 (60.26) 44.10 (60.26) 14,113 (80.2%) 3,482 85.53 (40.99) 82.94 (40.99) | #VALUE! 0.03 0.01 #VALUE! 0.00 -0.08 -0.12 -0.01 -0.04 -0.01 -0.00 -0.00 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only <5000 included)mean (sd)mean (sd)mean (sd)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only <5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only <5000 included)median [IQR]median [IQR]median [IQR] | 65.50 [32.60, 167.50] 8,805 [99.2%) 3,723 21.39 [9.92) 19.00 [15.00, 25.50] 5,157 [58.1%) 3,791 1.20 [0.50) 1.08 [0.87, 1.41] 5,089 [57.3%) 2,999 45.64 [13.89) 44.00 [36.00, 53.00] 5,881 [66.2%) 3,014 85.21 [41.48) 81.75 [60.00, 108.00] 5,866 (66.1%) | 8,764 (98.7%) 3,839 22.02 (10.30) 19.50 (15.00, 27.00) 5,041 (56.8%) 3,936 1.24 (0.51) 1.14 [0.88, 1.48] 4,944 (55.7%) 3,087 46.51 (14.12) 44.50 [37.00, 54.00] 5,793 (65.2%) 3,106 85.59 (40.41) 82.75 [61.00, 109.00] 5,774 (65.0%) | 80.00 [47.00, 204.50]<br>8,707 [99.9%)<br>534<br>550.42 [9.028.78]<br>18.00 [13.50, 24.00]<br>8,182 [93.9%)<br>520<br>1.15 [0.52)<br>1.00 [0.84, 1.36]<br>8,196 [94.0%)<br>501<br>43.93 [15.31]<br>42.50 [35.00, 52.00]<br>8,215 [94.3%)<br>481<br>86.93 (43.78)<br>85.00 [62.00, 109.58]<br>8,235 [94.5%) | 49.00 [15.10, 188.00]<br>8,705 [99.9%]<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 [94.7%]<br>468<br>1.18 [0.61]<br>1.01 [0.84, 1.35]<br>8,248 [94.6%]<br>396<br>51.64 (174.45)<br>41.00 [34.00, 52.00]<br>8,320 [95.5%]<br>376<br>85.05 (45.50)<br>84.50 [59.00, 111.38]<br>8,340 (95.7%) | N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) 47ALUEI 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) 13,285 (75.5%) 3,500 45.40 (14.10) 43.79 (14.10) 14,096 (80.1%) 3,495 85.45 (41.81) 82.20 (41.81) 14,101 (80.1%) | #VALUEI 17,469 (99.3%) 4,298 52.43 (1981.24) #VALUEI 13,298 (75.6%) 4,404 1.23 (0.52) 1.13 (0.52) 13,192 (75.0%) 3,483 47.09 (60.26) 44.10 (60.26) 14,113 (80.2%) 3,482 85.53 (40.99) 82.94 (40.99) 14,114 (80.2%) | #VALUE! 0.03 0.01 #VALUE! 0.00 -0.08 -0.12 -0.01 -0.04 -0.01 -0.00 -0.00 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only =<5000 included) | 65.50 [32.60, 167.50] 8,805 [99.2%] 3,723 21.39 [9.92) 19.00 [15.00, 25.50] 5,157 [58.1%] 3,791 1.20 [0.50] 1.08 [0.87, 1.41] 5,089 [57.3%] 2,999 45.64 [13.89] 44.00 [36.00, 53.00] 5,881 (66.2%) 3,014 85.21 (41.48) 81.75 [60.00, 108.00] 5,866 (66.1%) | 8,764 (98.7%) 3,839 22.02 (10.30) 19.50 (15.00, 27.00) 5,041 (56.8%) 3,936 1.24 (0.51) 1.14 [0.88, 1.48] 4,944 (55.7%) 3,087 46.51 (14.12) 44.50 (37.00, 54.00) 5,793 (65.2%) 3,106 85.59 (40.41) 82.75 [61.00, 109.00] 5,774 (65.0%) 3,148 | 80.00 [47.00, 204.50]<br>8,707 [99.9%)<br>534<br>550.42 (9,028.78)<br>18.00 [13.50, 24.00]<br>8,182 (93.9%)<br>520<br>1.15 (0.52)<br>1.00 [0.84, 1.36]<br>8,196 (94.0%)<br>501<br>43.93 (15.31)<br>42.50 [35.00, 52.00]<br>8,215 (94.3%)<br>481<br>86.93 (43.78)<br>85.00 [62.00, 109.58]<br>8,235 (94.5%) | 49.00 [15.10, 188.00]<br>8,705 [99.9%]<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 [94.7%]<br>468<br>1.18 (0.61)<br>1.01 [0.84, 1.35]<br>8,248 (94.6%)<br>396<br>51.64 (174.45)<br>41.00 [34.00, 52.00]<br>8,320 (95.5%)<br>376<br>85.05 (45.50)<br>84.50 [59.00, 111.38]<br>8,340 (95.7%) | N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) #VALUEI 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) 13,285 (75.5%) 3,500 45.40 (14.10) 43.79 (14.10) 14,096 (80.1%) 3,495 85.45 (41.81) 82.20 (41.81) 14,101 (80.1%) | #VALUEI 17,469 (99.3%) 4,298 52.43 (1981.24) #VALUEI 13,298 (75.6%) 4,404 1.23 (0.52) 1.13 (0.52) 1.3,192 (75.0%) 3,483 47.09 (60.26) 44.10 (60.26) 14,113 (80.2%) 3,482 85.53 (40.99) 82.94 (40.99) 14,114 (80.2%) 3,550 | #VALUE! 0.03 0.01 #VALUE! 0.00 -0.08 -0.12 0.01 -0.04 -0.01 0.00 0.00 -0.02 0.00 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only <5000 included)mean (sd)mean (sd)mean (sd)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only <5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only <5000 included)median [IQR]median [IQR]median [IQR] | 65.50 [32.60, 167.50] 8,805 [99.2%) 3,723 21.39 [9.92) 19.00 [15.00, 25.50] 5,157 [58.1%) 3,791 1.20 [0.50) 1.08 [0.87, 1.41] 5,089 [57.3%) 2,999 45.64 [13.89) 44.00 [36.00, 53.00] 5,881 [66.2%) 3,014 85.21 [41.48) 81.75 [60.00, 108.00] 5,866 (66.1%) | 8,764 (98.7%) 3,839 22.02 (10.30) 19.50 (15.00, 27.00) 5,041 (56.8%) 3,936 1.24 (0.51) 1.14 [0.88, 1.48] 4,944 (55.7%) 3,087 46.51 (14.12) 44.50 [37.00, 54.00] 5,793 (65.2%) 3,106 85.59 (40.41) 82.75 [61.00, 109.00] 5,774 (65.0%) | 80.00 [47.00, 204.50]<br>8,707 [99.9%)<br>534<br>550.42 [9.028.78]<br>18.00 [13.50, 24.00]<br>8,182 [93.9%)<br>520<br>1.15 [0.52)<br>1.00 [0.84, 1.36]<br>8,196 [94.0%)<br>501<br>43.93 [15.31]<br>42.50 [35.00, 52.00]<br>8,215 [94.3%)<br>481<br>86.93 (43.78)<br>85.00 [62.00, 109.58]<br>8,235 [94.5%) | 49.00 [15.10, 188.00]<br>8,705 [99.9%]<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 [94.7%]<br>468<br>1.18 [0.61]<br>1.01 [0.84, 1.35]<br>8,248 [94.6%]<br>396<br>51.64 (174.45)<br>41.00 [34.00, 52.00]<br>8,320 [95.5%]<br>376<br>85.05 (45.50)<br>84.50 [59.00, 111.38]<br>8,340 (95.7%) | N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) 47ALUEI 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) 13,285 (75.5%) 3,500 45.40 (14.10) 43.79 (14.10) 14,096 (80.1%) 3,495 85.45 (41.81) 82.20 (41.81) 14,101 (80.1%) | #VALUEI 17,469 (99.3%) 4,298 52.43 (1981.24) #VALUEI 13,298 (75.6%) 4,404 1.23 (0.52) 1.13 (0.52) 13,192 (75.0%) 3,483 47.09 (60.26) 44.10 (60.26) 14,113 (80.2%) 3,482 85.53 (40.99) 82.94 (40.99) 14,114 (80.2%) | #VALUE! 0.03 0.01 #VALUE! 0.00 -0.08 -0.12 -0.01 -0.04 -0.01 -0.00 -0.00 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only =<5000 included) | 65.50 [32.60, 167.50] 8,805 [99.2%] 3,723 21.39 [9.92) 19.00 [15.00, 25.50] 5,157 [58.1%] 3,791 1.20 [0.50] 1.08 [0.87, 1.41] 5,089 [57.3%] 2,999 45.64 [13.89] 44.00 [36.00, 53.00] 5,881 (66.2%) 3,014 85.21 (41.48) 81.75 [60.00, 108.00] 5,866 (66.1%) | 8,764 (98.7%) 3,839 22.02 (10.30) 19.50 (15.00, 27.00) 5,041 (56.8%) 3,936 1.24 (0.51) 1.14 [0.88, 1.48] 4,944 (55.7%) 3,087 46.51 (14.12) 44.50 [37.00, 54.00] 5,793 (65.2%) 3,106 85.59 (40.41) 82.75 [61.00, 109.00] 5,774 (65.0%) 3,148 173.80 (47.86) | 80.00 [47.00, 204.50]<br>8,707 [99.9%)<br>534<br>550.42 (9,028.78)<br>18.00 [13.50, 24.00]<br>8,182 (93.9%)<br>520<br>1.15 (0.52)<br>1.00 [0.84, 1.36]<br>8,196 (94.0%)<br>501<br>43.93 (15.31)<br>42.50 [35.00, 52.00]<br>8,215 (94.3%)<br>481<br>86.93 (43.78)<br>85.00 [62.00, 109.58]<br>8,235 (94.5%) | 49.00 [15.10, 188.00]<br>8,705 [99.9%]<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 [94.7%]<br>468<br>1.18 (0.61)<br>1.01 [0.84, 1.35]<br>8,248 (94.6%)<br>396<br>51.64 (174.45)<br>41.00 [34.00, 52.00]<br>8,320 (95.5%)<br>376<br>85.05 (45.50)<br>84.50 [59.00, 111.38]<br>8,340 (95.7%) | N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) #VALUEI 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) 13,285 (75.5%) 3,500 45.40 (14.10) 43.79 (14.10) 14,096 (80.1%) 3,495 85.45 (41.81) 82.20 (41.81) 14,101 (80.1%) | #VALUEI 17,469 (99.3%) 4,298 52.43 (1981.24) #VALUEI 13,298 (75.6%) 4,404 1.23 (0.52) 1.13 (0.52) 1.3,192 (75.0%) 3,483 47.09 (60.26) 44.10 (60.26) 14,113 (80.2%) 3,482 85.53 (40.99) 82.94 (40.99) 14,114 (80.2%) 3,550 | #VALUE! 0.03 0.01 #VALUE! 0.00 -0.08 -0.12 0.01 -0.04 -0.01 0.00 0.00 -0.02 0.00 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only =<5000 included)mean (sd)median [IQR] | 65.50 [32.60, 167.50] 8,805 [99.2%) 3,723 21.39 [9.92) 19.00 [15.00, 25.50] 5,157 (58.1%) 3,791 1.20 (0.50) 1.08 [0.87, 1.41] 5,089 (57.3%) 2,999 45.64 (13.89) 44.00 [36.00, 53.00] 5,881 (66.2%) 3,014 85.21 (41.48) 81.75 [60.00, 108.00] 5,866 (66.1%) 3,048 172.69 (47.81) 166.00 [141.00, 199.00] | 8,764 (98.7%) 3,839 22.02 (10.30) 19.50 (15.00, 27.00) 5,041 (56.8%) 3,936 1.24 (0.51) 1.14 [0.88, 1.48] 4,944 (55.7%) 3,087 46.51 (14.12) 44.50 (37.00, 54.00) 5,793 (65.2%) 3,106 85.59 (40.41) 82.75 [61.00, 109.00] 5,774 (65.0%) 3,148 173.80 (47.86) 166.00 [142.00, 197.50] | 80.00 [47.00, 204.50] 8,707 [99.9%) 534 550.42 (9.028.78) 18.00 [13.50, 24.00] 8,182 [93.9%) 520 1.15 [0.52) 1.00 [0.84, 1.36] 8,196 [94.0%) 43.93 [15.31) 42.50 [35.00, 52.00] 8,215 [94.3%) 481 86.93 [43.78) 85.00 [62.00, 109.58] 8,235 [94.5%) 504 173.39 [53.59) 168.00 [143.00, 202.88] | 49.00 [15.10, 188.00] 8,705 [99.9%) 459 306.80 (6,067.08) 18.50 [14.00, 26.00] 8,257 [94.7%) 468 1.18 (0.61) 1.01 [0.84, 1.35] 8,248 [94.6%) 396 51.64 (174.45) 41.00 [34.00,52.00] 8,320 [95.5%) 376 85.05 [45.50] 84.50 [59.00, 111.38] 8,340 [95.7%] | N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) #VALUEI 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) 13,285 (75.5%) 3,500 45.40 (14.10) 43.79 (14.10) 14,096 (80.1%) 3,495 85.45 (41.81) 82.20 (41.81) 14,101 (80.1%) 3,552 172.79 (48.68) 166.28 (48.68) | #VALUEI 17,469 (99.3%) 4,298 52.43 (1981.24) #VALUEI 13,298 (75.6%) 4,404 1.23 (0.52) 1.13 (0.52) 13,192 (75.0%) 3,483 47.09 (60.26) 44.10 (60.26) 14,113 (80.2%) 3,482 85.53 (40.99) 82.94 (40.99) 14,114 (80.2%) 3,550 173.82 (49.00) 166.45 (49.00) | #VALUE! 0.03 0.01 #VALUE! 0.00 -0.08 -0.12 0.01 -0.04 -0.01 0.00 -0.02 0.00 -0.02 0.00 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only <5000 included)mean (sd)mean (sd)mean (sd)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only <5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only <5000 included)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only <5000 included)median [IQR]Missing; n (%)median [IQR]mean (sd)mean (sd)mean [IQR]mean [IQR] | 65.50 [32.60, 167.50] 8,805 [99.2%] 3,723 21.39 [9.92) 19.00 [15.00, 25.50] 5,157 [58.1%] 3,791 1.20 [0.50) 1.08 [0.87, 1.41] 5,089 [57.3%) 45.64 [13.89] 44.00 [36.00, 53.00] 5,881 [66.2%] 3,014 85.21 [41.48] 81.75 [60.00, 108.00] 5,866 [66.1%] | 8,764 (98.7%) 3,839 22.02 (10.30) 19.50 (15.00, 27.00) 5,041 (56.8%) 3,936 1.24 (0.51) 1.14 [0.88, 1.48] 4,944 (55.7%) 3,087 46.51 (14.12) 44.50 [37.00, 54.00] 5,793 (65.2%) 3,106 85.59 (40.41) 82.75 [61.00, 109.00] 5,774 (65.0%) 3,148 173.80 (47.86) | 80.00 [47.00, 204.50]<br>8,707 [99.9%)<br>550.42 (9,028.78)<br>18.00 [13.50, 24.00]<br>8,182 (93.9%)<br>520<br>1.15 (0.52)<br>1.00 [0.84, 1.36]<br>8,196 (94.0%)<br>501<br>43.93 [15.31)<br>42.50 [35.00, 52.00]<br>8,215 (94.3%)<br>481<br>86.93 (43.78)<br>85.00 [62.00, 109.58]<br>8,235 (94.5%) | 49.00 [15.10, 188.00]<br>8,705 [99.9%]<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 [94.7%]<br>468<br>1.18 (0.61)<br>1.01 [0.84, 1.35]<br>8,248 [94.6%]<br>396<br>51.64 (174.45)<br>41.00 [34.00, 52.00]<br>8,320 [95.5%]<br>376<br>85.05 [45.50]<br>84.50 [59.00, 111.38]<br>8,340 [95.7%] | N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) #VALUEI 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) 13,285 (75.5%) 3,500 45.40 (14.10) 43.79 (14.10) 14,096 (80.1%) 85.45 (41.81) 14,101 (80.1%) 3,552 172.79 (48.68) | #VALUEI 17,469 (99.3%) 4,298 52.43 (1981.24) #VALUEI 13,298 (75.6%) 4,404 1.23 (0.52) 1.13 (0.52) 1.3,192 (75.0%) 3,483 47.09 (60.26) 44.10 (60.26) 14,113 (80.2%) 3,482 85.53 (40.99) 82.94 (40.99) 14,114 (80.2%) 3,550 173.82 (49.00) | #VALUE! 0.03 0.01 #VALUE! 0.00 -0.08 -0.12 -0.01 -0.04 -0.01 -0.00 -0.02 -0.02 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-TDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) | 65.50 [32.60, 167.50] 8,805 [99.2%) 3,723 21.39 [9.92) 19.00 [15.00, 25.50] 5,157 [58.1%) 3,791 1.20 [0.50) 1.08 [0.87, 1.41] 5,089 [57.3%) 45.64 [13.89) 44.00 [36.00, 53.00] 5,881 (66.2%) 3,014 85.21 (41.48) 81.75 [60.00, 108.00] 5,866 (66.1%) 3,048 172.69 (47.81) 166.00 [141.00, 199.00] 5,832 (65.7%) | 8,764 (98.7%) 3,839 22.02 (10.30) 19.50 (15.00, 27.00] 5,041 (56.8%) 3,936 1.24 (0.51) 1.14 [0.88, 1.48] 4,944 (55.7%) 3,087 46.51 (14.12) 44.50 (37.00, 54.00) 5,793 (65.2%) 3,106 85.59 (40.41) 82.75 [61.00, 109.00] 5,774 (65.0%) 3,148 173.80 (47.86) 166.00 [142.00, 197.50] 5,732 (64.5%) | 80.00 [47.00, 204.50] 8,707 [99.9%) 534 550.42 (9,028.78) 18.00 [13.50, 24.00] 8,182 (93.9%) 520 1.15 (0.52) 1.00 [0.84, 1.36] 8,196 (94.0%) 501 43.93 (15.31) 42.50 [35.00, 52.00] 8,215 (94.3%) 481 86.93 (43.78) 85.00 [62.00, 109.58] 8,235 (94.5%) 173.39 (53.59) 168.00 [143.00, 202.88] 8,212 (94.2%) | 49.00 [15.10, 188.00]<br>8,705 [99.9%]<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 [94.7%]<br>468<br>1.18 (0.61)<br>1.01 [0.84, 1.35]<br>8,248 (94.6%)<br>396<br>51.64 (174.45)<br>41.00 [34.00, 52.00]<br>8,320 (95.5%)<br>376<br>85.05 (45.50)<br>84.50 [59.00, 111.38]<br>8,340 (95.7%)<br>402<br>173.95 (57.11)<br>170.00 [141.00, 205.00]<br>8,314 (95.4%) | N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) #VALUEI 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) 13,285 (75.5%) 3,500 45.40 (14.10) 43.79 (14.10) 14,096 (80.1%) 85.45 (41.81) 82.20 (41.81) 14,101 (80.1%) 3,552 172.79 (48.68) 166.28 (48.68) 14,044 (79.8%) | #VALUEI 17,469 (99.3%) 4,298 52.43 (1981.24) #VALUEI 13,298 (75.6%) 4,404 1.23 (0.52) 1.13 (0.52) 1.3,192 (75.0%) 3,483 47.09 (60.26) 44.10 (60.26) 14,113 (80.2%) 3,482 85.53 (40.99) 82.94 (40.99) 14,114 (80.2%) 3,550 173.82 (49.00) 166.45 (49.00) 14,046 (79.8%) | #VALUE! 0.03 0.01 #VALUE! 0.00 -0.08 -0.12 0.01 -0.04 -0.01 0.00 -0.02 0.00 -0.02 0.00 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only <5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only <5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only <5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only <5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only <5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Triglyceride level (mg/dl) mean (only <5000 included) | 65.50 [32.60, 167.50] 8,805 [99.2%) 3,723 21.39 [9.92) 19.00 [15.00, 25.50] 5,157 (58.1%) 3,791 1.20 (0.50) 1.08 [0.87, 1.41] 5,089 [57.3%) 2,999 45.64 [13.89) 44.00 [36.00, 53.00] 5,881 (66.2%) 3,014 85.21 [41.48) 81.75 [60.00, 108.00] 5,866 (66.1%) 3,048 172.69 [47.81] 166.00 [141.00, 199.00] 5,832 (65.7%) | 8,764 (98.7%) 3,839 22.02 (10.30) 19.50 (15.00, 27.00) 5,041 (56.8%) 3,936 1.24 (0.51) 1.14 [0.88, 1.48] 4,944 (55.7%) 3,087 46.51 (14.12) 44.50 [37.00, 54.00] 5,793 (65.2%) 3,106 85.59 (40.41) 82.75 [61.00, 109.00] 5,774 (65.0%) 3,148 173.80 (47.86) 166.00 [142.00, 197.50] 5,732 (64.5%) 3,135 | 80.00 [47.00, 204.50] 8,707 [99.9%) 534 550.42 [9,028.78) 18.00 [13.50, 24.00] 8,182 [93.9%) 520 1.15 [0.52) 1.00 [0.84, 1.36] 8,196 [94.0%) 501 43.93 [15.31) 42.50 [35.00, 52.00] 8,215 [94.3%) 481 86.93 [43.78) 85.00 [62.00, 109.58] 8,235 [94.5%) 504 173.39 [53.59) 168.00 [143.00, 202.88] 8,212 [94.2%) | 49.00 [15.10, 188.00]<br>8,705 [99.9%]<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 [94.7%]<br>468<br>1.18 (0.61)<br>1.01 [0.84, 1.35]<br>8,248 [94.6%]<br>396<br>51.64 (174.45)<br>41.00 [34.00,52.00]<br>8,320 [95.5%]<br>376<br>85.05 [45.50]<br>84.50 [59.00, 111.38]<br>8,340 [95.7%]<br>402<br>173.95 [57.11]<br>170.00 [141.00, 205.00]<br>8,314 [95.4%] | N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) #VALUEI 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) 13,285 (75.5%) 3,500 45.40 (14.10) 43.79 (14.10) 14,096 (80.1%) 85.45 (41.81) 82.20 (41.81) 14,101 (80.1%) 3,552 172.79 (48.68) 166.28 (48.68) 14,044 (79.8%) | #VALUEI 17,469 (99.3%) 4,298 52.43 (1981.24) #VALUEI 13,298 (75.6%) 4,404 1.23 (0.52) 1.13 (0.52) 13,192 (75.0%) 3,483 47.09 (60.26) 44.10 (60.26) 14,113 (80.2%) 3,482 85.53 (40.99) 82.94 (40.99) 14,114 (80.2%) 3,550 173.82 (49.00) 166.45 (49.00) 14,046 (79.8%) 3,532 | #VALUE! 0.03 0.01 #VALUE! 0.00 -0.08 -0.12 0.01 -0.04 -0.01 0.00 -0.02 0.00 -0.02 0.00 -0.02 0.00 0.00 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-TDL level (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only =<5000 included)mean (sd)median [IQR]Missing; n (%) | 65.50 [32.60, 167.50] 8,805 [99.2%) 3,723 21.39 [9.92) 19.00 [15.00, 25.50] 5,157 [58.1%) 3,791 1.20 [0.50) 1.08 [0.87, 1.41] 5,089 [57.3%) 45.64 [13.89) 44.00 [36.00, 53.00] 5,881 (66.2%) 3,014 85.21 (41.48) 81.75 [60.00, 108.00] 5,866 (66.1%) 3,048 172.69 (47.81) 166.00 [141.00, 199.00] 5,832 (65.7%) | 8,764 (98.7%) 3,839 22.02 (10.30) 19.50 (15.00, 27.00] 5,041 (56.8%) 3,936 1.24 (0.51) 1.14 [0.88, 1.48] 4,944 (55.7%) 3,087 46.51 (14.12) 44.50 (37.00, 54.00) 5,793 (65.2%) 3,106 85.59 (40.41) 82.75 [61.00, 109.00] 5,774 (65.0%) 3,148 173.80 (47.86) 166.00 [142.00, 197.50] 5,732 (64.5%) | 80.00 [47.00, 204.50] 8,707 [99.9%) 534 550.42 (9,028.78) 18.00 [13.50, 24.00] 8,182 (93.9%) 520 1.15 (0.52) 1.00 [0.84, 1.36] 8,196 (94.0%) 501 43.93 (15.31) 42.50 [35.00, 52.00] 8,215 (94.3%) 481 86.93 (43.78) 85.00 [62.00, 109.58] 8,235 (94.5%) 173.39 (53.59) 168.00 [143.00, 202.88] 8,212 (94.2%) | 49.00 [15.10, 188.00]<br>8,705 [99.9%]<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 [94.7%]<br>468<br>1.18 (0.61)<br>1.01 [0.84, 1.35]<br>8,248 (94.6%)<br>396<br>51.64 (174.45)<br>41.00 [34.00, 52.00]<br>8,320 (95.5%)<br>376<br>85.05 (45.50)<br>84.50 [59.00, 111.38]<br>8,340 (95.7%)<br>402<br>173.95 (57.11)<br>170.00 [141.00, 205.00]<br>8,314 (95.4%) | N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) #VALUEI 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) 13,285 (75.5%) 3,500 45.40 (14.10) 43.79 (14.10) 14,096 (80.1%) 85.45 (41.81) 82.20 (41.81) 14,101 (80.1%) 3,552 172.79 (48.68) 166.28 (48.68) 14,044 (79.8%) | #VALUEI 17,469 (99.3%) 4,298 52.43 (1981.24) #VALUEI 13,298 (75.6%) 4,404 1.23 (0.52) 1.13 (0.52) 1.3,192 (75.0%) 3,483 47.09 (60.26) 44.10 (60.26) 14,113 (80.2%) 3,482 85.53 (40.99) 82.94 (40.99) 14,114 (80.2%) 3,550 173.82 (49.00) 166.45 (49.00) 14,046 (79.8%) | #VALUE! 0.03 0.01 #VALUE! 0.00 -0.08 -0.12 0.01 -0.04 -0.01 0.00 -0.02 0.00 -0.02 0.00 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)mean (sd)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only <5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only <5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only <5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only <5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only <5000 included)mean (sd)median [IQR]Missing; n (%) Lab result number-Triglyceride level (mg/dl) mean (only <5000 included) | 65.50 [32.60, 167.50] 8,805 [99.2%) 3,723 21.39 [9.92) 19.00 [15.00, 25.50] 5,157 (58.1%) 3,791 1.20 (0.50) 1.08 [0.87, 1.41] 5,089 [57.3%) 2,999 45.64 [13.89) 44.00 [36.00, 53.00] 5,881 (66.2%) 3,014 85.21 [41.48) 81.75 [60.00, 108.00] 5,866 (66.1%) 3,048 172.69 [47.81] 166.00 [141.00, 199.00] 5,832 (65.7%) | 8,764 (98.7%) 3,839 22.02 (10.30) 19.50 [15.00, 27.00] 5,041 (56.8%) 3,936 1.24 (0.51) 1.14 [0.88, 1.48] 4,944 (55.7%) 3,087 46.51 (14.12) 44.50 (37.00, 54.00) 5,793 (65.2%) 3,106 85.59 (40.41) 82.75 [61.00, 109.00] 5,774 (65.0%) 3,148 173.80 (47.86) 166.00 [142.00, 197.50] 5,732 (64.5%) 3,135 189.61 (172.97) | 80.00 [47.00, 204.50] 8,707 [99.9%) 534 550.42 [9,028.78) 18.00 [13.50, 24.00] 8,182 [93.9%) 520 1.15 [0.52) 1.00 [0.84, 1.36] 8,196 [94.0%) 501 43.93 [15.31) 42.50 [35.00, 52.00] 8,215 [94.3%) 481 86.93 [43.78) 85.00 [62.00, 109.58] 8,235 [94.5%) 504 173.39 [53.59) 168.00 [143.00, 202.88] 8,212 [94.2%) | 49.00 [15.10, 188.00]<br>8,705 [99.9%]<br>459<br>306.80 (6,067.08)<br>18.50 [14.00, 26.00]<br>8,257 [94.7%]<br>468<br>1.18 (0.61)<br>1.01 [0.84, 1.35]<br>8,248 [94.6%]<br>396<br>51.64 (174.45)<br>41.00 [34.00,52.00]<br>8,320 [95.5%]<br>376<br>85.05 [45.50]<br>84.50 [59.00, 111.38]<br>8,340 [95.7%]<br>402<br>173.95 [57.11]<br>170.00 [141.00, 205.00]<br>8,314 [95.4%] | N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) #VALUEI 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) 13,285 (75.5%) 3,500 45.40 (14.10) 43.79 (14.10) 14,096 (80.1%) 85.45 (41.81) 82.20 (41.81) 14,101 (80.1%) 3,552 172.79 (48.68) 166.28 (48.68) 14,044 (79.8%) | #VALUEI 17,469 (99.3%) 4,298 52.43 (1981.24) #VALUEI 13,298 (75.6%) 4,404 1.23 (0.52) 1.13 (0.52) 13,192 (75.0%) 3,483 47.09 (60.26) 44.10 (60.26) 14,113 (80.2%) 3,482 85.53 (40.99) 82.94 (40.99) 14,114 (80.2%) 3,550 173.82 (49.00) 166.45 (49.00) 14,046 (79.8%) 3,532 | #VALUE! 0.03 0.01 #VALUE! 0.00 -0.08 -0.12 0.01 -0.04 -0.01 0.00 -0.02 0.00 -0.02 0.00 -0.02 0.00 0.00 |
| Missing; n (%) Lab result number-BUN (mg/dl) meanmean (sd)median [IQR]Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included)median [IQR]Missing; n (%) Lab result number-HDL level (mg/dl) mean (only <5000 included)mean (sd)mean (sd)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only<br><5000 included)median [IQR]Missing; n (%) Lab result number-LDL level (mg/dl) mean (only<br><5000 included)median [IQR]Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean (only<br><br>Lab result number-Triglyceride level (mg/dl) mean (only<br>median [IQR]Missing; n (%) Lab result number-Triglyceride level (mg/dl) mean (only<br>Lab result number-Triglyceride level (mg/dl) mean (only | 65.50 [32.60, 167.50] 8,805 [99.2%) 3,723 21.39 [9.92) 19.00 [15.00, 25.50] 5,157 (58.1%) 3,791 1.20 [0.50] 1.08 [0.87, 1.41] 5,089 (57.3%) 2,999 45.64 (13.89) 44.00 [36.00, 53.00] 5,881 (66.2%) 3,014 85.21 (41.48) 81.75 [60.00, 108.00] 5,866 (66.1%) 3,048 172.69 (47.81) 166.00 [141.00, 199.00] 5,832 (65.7%) 3,015 193.31 [156.70) | 8,764 (98.7%) 3,839 22.02 (10.30) 19.50 [15.00, 27.00] 5,041 (56.8%) 3,936 1.24 (0.51) 1.14 [0.88, 1.48] 4,944 (55.7%) 3,087 46.51 (14.12) 44.50 (37.00, 54.00) 5,793 (65.2%) 3,106 85.59 (40.41) 82.75 [61.00, 109.00] 5,774 (65.0%) 3,148 173.80 (47.86) 166.00 [142.00, 197.50] 5,732 (64.5%) 3,135 189.61 (172.97) | 80.00 [47.00, 204.50] 8,707 [99.9%) 534 550.42 [9.028.78) 18.00 [13.50, 24.00] 8,182 [93.9%) 520 1.15 [0.52) 1.00 [0.84, 1.36] 8,196 [94.0%) 501 43.93 [15.31] 42.50 [35.00, 52.00] 8,215 [94.3%) 481 86.93 (43.78) 85.00 [62.00, 109.58] 8,235 [94.5%) 504 173.39 [53.59) 168.00 [143.00, 202.88] 8,212 [94.2%) | 49.00 [15.10, 188.00] 8,705 [99.9%) 459 306.80 (6,067.08) 18.50 [14.00, 26.00] 8,257 [94.7%) 468 1.18 (0.61) 1.01 [0.84, 1.35] 8,248 [94.6%) 396 51.64 (174.45) 41.00 [34.00, 52.00] 8,320 [95.5%) 376 85.05 (45.50) 84.50 [59.00, 111.38] 8,340 (95.7%) 402 173.95 [57.11) 170.00 [141.00, 205.00] 8,314 (95.4%) 397 212.71 (232.81) | N/A | N/A | 17,512 (99.5%) 4,257 87.75 (3195.92) #VALUEI 13,339 (75.8%) 4,311 1.19 (0.50) 1.07 (0.50) 13,285 (75.5%) 3,500 45.40 (14.10) 43.79 (14.10) 14,096 (80.1%) 3,495 85.45 (41.81) 82.20 (41.81) 14,101 (80.1%) 3,552 172.79 (48.68) 166.28 (48.68) 14,044 (79.8%) 3,514 193.66 (159.37) | #VALUEI 17,469 (99.3%) 4,298 52.43 (1981.24) #VALUEI 13,298 (75.6%) 4,404 1.23 (0.52) 1.13 (0.52) 13,192 (75.0%) 3,483 47.09 (60.26) 44.10 (60.26) 14,113 (80.2%) 3,482 85.53 (40.99) 82.94 (40.99) 14,114 (80.2%) 3,550 173.82 (49.00) 166.45 (49.00) 14,046 (79.8%) 3,532 192.21 (180.70) | #VALUE! 0.03 0.01 #VALUE! 0.00 -0.08 -0.12 0.01 -0.04 -0.01 0.00 -0.02 0.00 -0.02 0.00 0.00 0.00 0 |

| Lab result number- Hemoglobin mean (only >0 | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| included) | 2,720 | 2,902 | 370 | 352 | N/A | N/A | 3,090 | 3,254 | |
| mean (sd) | 13.16 (1.75) | 13.17 (1.73) | 377.00 (7,000.31) | 444.91 (8,100.93) | N/A | N/A | 56.73 (2420.26) | 59.87 (2661.83) | 0.00 |
| median [IQR] | 13.20 [11.90, 14.40] | 13.20 [11.95, 14.40] | 13.30 [12.00, 14.70] | 13.30 [12.00, 14.54] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Missing; n (%) | 6,160 (69.4%) | 5,978 (67.3%) | 8,346 (95.8%) | 8,364 (96.0%) | N/A | N/A | 14,506 (82.4%) | 14,342 (81.5%) | 0.02 |
| Lab result number- Serum sodium mean (only > 90 | | | | | | | | | |
| and < 190 included) | 3,702 | 3,832 | 514 | 457 | N/A | N/A | 4,216 | 4,289 | |
| mean (sd) | 139.51 (2.85) | 139.59 (2.84) | 139.02 (3.31) | 139.09 (2.65) | N/A | N/A | 139.45 (2.91) | 139.54 (2.82) | -0.03 |
| median [IQR] | 140.00 [138.00, 141.33] | 140.00 [138.00, 141.50] | 139.00 [137.50, 141.00] | 139.33 [137.00, 141.00] | N/A | N/A | 139.88 (2.91) | 139.93 (2.82) | -0.02 |
| Missing; n (%) | 5,178 (58.3%) | 5,048 (56.8%) | 8,202 (94.1%) | 8,259 (94.8%) | N/A | N/A | 13,380 (76.0%) | 13,307 (75.6%) | 0.01 |
| Lab result number- Albumin mean (only >0 and <=10 | | | | | | | | | |
| included) | 3,422 | 3,605 | 447 | 397 | N/A | N/A | 3,869 | 4,002 | |
| mean (sd) | 4.20 (0.35) | 4.21 (0.36) | 4.04 (0.76) | 4.09 (0.71) | N/A | N/A | 4.18 (0.42) | 4.20 (0.41) | -0.05 |
| median [IQR] | 4.20 [4.00, 4.40] | 4.20 [4.00, 4.45] | 4.15 [4.00, 4.40] | 4.20 [4.00, 4.40] | N/A | N/A | 4.19 (0.42) | 4.20 (0.41) | -0.02 |
| Missing; n (%) | 5,458 (61.5%) | 5,275 (59.4%) | 8,269 (94.9%) | 8,319 (95.4%) | N/A | N/A | 13,727 (78.0%) | 13,594 (77.3%) | 0.02 |
| Lab result number- Glucose (fasting or random) mean<br>(only 10-1000 included) | 3.684 | 3,829 | 509 | 456 | N/A | N/A | 4.193 | 4.285 | |
| mean (sd) | 171.75 (75.07) | 164.58 (71.69) | 171.74 (71.84) | 166.42 (76.33) | N/A<br>N/A | N/A<br>N/A | 171.75 (74.69) | 164.78 (72.21) | 0.09 |
| median [IQR] | 171.73 (73.07) | 146.00 [118.50, 187.00] | 152.50 [124.25, 198.50] | 145.00 [121.12, 188.00] | N/A<br>N/A | N/A<br>N/A | 152.94 (74.69) | 145.89 (72.21) | 0.10 |
| Missing; n (%) | 5,196 (58.5%) | 5,051 (56.9%) | 8,207 (94.2%) | 8,260 (94.8%) | N/A | N/A | 13,403 (76.2%) | 13,311 (75.6%) | 0.01 |
| Lab result number- Potassium mean (only 1-7 | 3,130 (38.376) | 3,031 (30.376) | 8,207 (34.278) | 8,200 (34.8%) | N/A | N/A | 13,403 (70.270) | 13,311 (73.0%) | 0.01 |
| included) | 3,791 | 3,927 | 523 | 449 | N/A | N/A | 4,314 | 4,376 | |
| mean (sd) | 4.49 (0.46) | 4.49 (0.46) | 4.34 (0.47) | 4.37 (0.50) | N/A | N/A | 4.47 (0.46) | 4.48 (0.46) | -0.02 |
| median [IQR] | 4.50 [4.20, 4.80] | 4.50 [4.20, 4.80] | 4.30 [4.00, 4.70] | 4.40 [4.07, 4.70] | N/A | N/A | 4.48 (0.46) | 4.49 (0.46) | -0.02 |
| Missing; n (%) | 5,089 (57.3%) | 4,953 (55.8%) | 8,193 (94.0%) | 8,267 (94.8%) | N/A | N/A | 13,282 (75.5%) | 13,220 (75.1%) | 0.01 |
| Comorbidity Scores | . , , | . , , | | , | • | · | . , , | | |
| CCI (180 days)- ICD9 and ICD10 | | | | | | | | | |
| mean (sd) | 3.36 (2.08) | 3.35 (2.10) | 2.46 (1.88) | 2.45 (1.86) | 3.77 (2.14) | 3.77 (2.11) | 3.47 (2.09) | 3.47 (2.07) | 0.00 |
| median [IQR] | 3.00 [2.00, 5.00] | 3.00 [2.00, 5.00] | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | 4.00 [2.00, 5.00] | 4.00 [2.00, 5.00] | 3.48 (2.09) | 3.48 (2.07) | 0.00 |
| Frailty Score: Qualitative Version 365 days as | | | | | | | | | |
| Categories, v1 | | | | | | | | | |
| 0; n (%) | 4,324 (48.7%) | 4,263 (48.0%) | 2,619 (30.0%) | 2,596 (29.8%) | 9,977 (29.9%) | 9,686 (29.1%) | 16,920 (33.2%) | 16,545 (32.5%) | 0.01 |
| 1 to 2; n (%) | 2,752 (31.0%) | 2,873 (32.4%) | 3,661 (42.0%) | 3,717 (42.6%) | 10,036 (30.1%) | 10,218 (30.7%) | 16,449 (32.3%) | 16,808 (33.0%) | -0.01 |
| 3 or more; n (%) | 1,804 (20.3%) | 1,744 (19.6%) | 2,436 (27.9%) | 2,403 (27.6%) | 13,306 (39.9%) | 13,415 (40.3%) | 17,546 (34.5%) | 17,562 (34.5%) | 0.00 |
| Frailty Score: Empirical Version 365 days as | | | | | | | | | |
| Categories, | | | | | | | | | |
| < 0.12908; n (%) | 1,119 (12.6%) | 1,228 (13.8%) | 1,240 (14.2%) | 1,338 (15.4%) | 1,500 (4.5%) | 1,563 (4.7%) | 3,859 (7.6%) | 4,129 (8.1%) | -0.02 |
| 0.12908 - 0.1631167; n (%) | 2,577 (29.0%) | 2,521 (28.4%) | 2,640 (30.3%) | 2,578 (29.6%) | 5,589 (16.8%) | 5,398 (16.2%) | 10,806 (21.2%) | 10,497 (20.6%) | 0.01 |
| >= 0.1631167; n (%) | 5,184 (58.4%) | 5,131 (57.8%) | 4,836 (55.5%) | 4,800 (55.1%) | 26,230 (78.7%) | 26,358 (79.1%) | 36,250 (71.2%) | 36,289 (71.3%) | 0.00 |
| Non-Frailty; n (%) | 4,985 (56.1%) | 5,157 (58.1%) | 4,680 (53.7%) | 4,703 (54.0%) | 1,469 (4.4%) | 1,398 (4.2%) | 11,134 (21.9%) | 11,258 (22.1%) | 0.00 |
| Family Construction (Constitution Version 205 days of | | | | | | | | | |
| Frailty Score (mean): Qualitative Version 365 days, v1 | 1.34 (1.92) | 1 22 (1 00) | 1.80 (1.89) | 1.79 (1.89) | 2.26 (2.42) | 2.36 (2.39) | 2.09 (2.26) | 2.00 (2.22) | 0.00 |
| mean (sd)median [IQR] | 1.00 [0.00, 2.00] | 1.33 (1.90)<br>1.00 [0.00, 2.00] | 1.00 [0.00, 3.00] | 1.00 [0.00, 3.00] | 2.36 (2.43)<br>2.00 [0.00, 4.00] | 2.00 [0.00, 4.00] | 1.65 (2.26) | 2.08 (2.23)<br>1.65 (2.23) | 0.00 |
| Frailty Score (mean): Empirical Version 365 days, | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 1.00 [0.00, 5.00] | 1.00 [0.00, 5.00] | 2.00 [0.00, 4.00] | 2.00 [0.00, 4.00] | 1.03 (2.20) | 1.03 (2.23) | 0.00 |
| mean (sd) | 0.19 (0.06) | 0.18 (0.06) | 0.17 (0.05) | 0.17 (0.05) | 0.21 (0.07) | 0.21 (0.07) | 0.20 (0.07) | 0.20 (0.07) | 0.00 |
| median [IQR] | 0.17 [0.14, 0.21] | 0.17 [0.14, 0.21] | 0.16 [0.14, 0.20] | 0.17 (0.03) | 0.20 [0.17, 0.25] | 0.20 [0.17, 0.25] | 0.19 (0.07) | 0.19 (0.07) | 0.00 |
| Healthcare Utilization | 0.17 [0.14, 0.21] | 0.17 [0.14, 0.21] | 0.10 [0.14, 0.20] | 0.10 [0.14, 0.15] | 0.20 [0.17, 0.25] | 0.20 [0.17, 0.25] | 0.13 (0.07) | 0.13 (0.07) | 0.00 |
| Any hospitalization; n (%) | 951 (10.7%) | 916 (10.3%) | 906 (10.4%) | 897 (10.3%) | 4,351 (13.1%) | 4,278 (12.8%) | 6,208 (12.2%) | 6,091 (12.0%) | 0.01 |
| Any hospitalization within prior 30 days; n (%) | 309 (3.5%) | 317 (3.6%) | 272 (3.1%) | 263 (3.0%) | 1,445 (4.3%) | 1,387 (4.2%) | 2,026 (4.0%) | 1,967 (3.9%) | 0.01 |
| Any hospitalization during prior 31-180 days; n (%) | 693 (7.8%) | 651 (7.3%) | 677 (7.8%) | 677 (7.8%) | 3,166 (9.5%) | 3,174 (9.5%) | 4,536 (8.9%) | 4,502 (8.8%) | 0.00 |
| Endocrinologist Visit; n (%) | 1,343 (15.1%) | 1,478 (16.6%) | 1,393 (16.0%) | 1,466 (16.8%) | 5,278 (15.8%) | 5,440 (16.3%) | 8,014 (15.7%) | 8,384 (16.5%) | -0.02 |
| Endocrinologist Visit (30 days prior); n (%) | 991 (11.2%) | 1,058 (11.9%) | 1,024 (11.7%) | 1,071 (12.3%) | 3,820 (11.5%) | 3,835 (11.5%) | 5,835 (11.5%) | 5,964 (11.7%) | -0.01 |
| Endocrinologist Visit (31 to 180 days prior); n (%) | 887 (10.0%) | 950 (10.7%) | 917 (10.5%) | 947 (10.9%) | 3,673 (11.0%) | 3,706 (11.1%) | 5,477 (10.8%) | 5,603 (11.0%) | -0.01 |
| Internal medicine/family medicine visits; n (%) | 7,278 (82.0%) | 7,050 (79.4%) | 7,636 (87.6%) | 7,551 (86.6%) | 28,049 (84.2%) | 27,792 (83.4%) | 42,963 (84.4%) | 42,393 (83.3%) | 0.03 |
| Internal medicine/family medicine visits (30 days | | | | | | | | | |
| prior); n (%) | 5,304 (59.7%) | 5,228 (58.9%) | 5,717 (65.6%) | 5,661 (64.9%) | 20,249 (60.8%) | 20,237 (60.7%) | 31,270 (61.4%) | 31,126 (61.1%) | 0.01 |
| Internal medicine/family medicine visits (31 to 180 | | | | | | | | | |
| days prior); n (%) | 6,220 (70.0%) | 6,222 (70.1%) | 6,651 (76.3%) | 6,585 (75.6%) | 24,952 (74.9%) | 25,013 (75.1%) | 37,823 (74.3%) | 37,820 (74.3%) | 0.00 |
| Cardiologist visit; n (%) | 3,365 (37.9%) | 3,383 (38.1%) | 2,819 (32.3%) | 2,869 (32.9%) | 14,336 (43.0%) | 14,230 (42.7%) | 20,520 (40.3%) | 20,482 (40.2%) | 0.00 |
| Number of Cardiologist visits (30 days prior); n (%) | 1,244 (14.0%) | 1,238 (13.9%) | 963 (11.0%) | 974 (11.2%) | 4,841 (14.5%) | 4,850 (14.6%) | 7,048 (13.8%) | 7,062 (13.9%) | 0.00 |
| Number of Cardiologist visits (31 to 180 days prior); | | | | | | | | | |
| n (%) | 2,851 (32.1%) | 2,880 (32.4%) | 2,408 (27.6%) | 2,477 (28.4%) | 12,553 (37.7%) | 12,531 (37.6%) | 17,812 (35.0%) | 17,888 (35.1%) | 0.00 |
| Electrocardiogram ; n (%) | 3,280 (36.9%) | 3,359 (37.8%) | 3,176 (36.4%) | 3,230 (37.1%) | 13,574 (40.7%) | 13,706 (41.1%) | 20,030 (39.3%) | 20,295 (39.9%) | -0.01 |
| Use of glucose test strips; n (%) | 423 (4.8%) | 427 (4.8%) | 410 (4.7%) | 399 (4.6%) | 1,375 (4.1%) | 1,338 (4.0%) | 2,208 (4.3%) | 2,164 (4.3%) | 0.00 |
| Dialysis; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| Naive new user ; n (%) | 2,349 (26.5%) | 2,521 (28.4%) | 2,348 (26.9%) | 2,409 (27.6%) | 7,673 (23.0%) | 8,355 (25.1%) | 12,370 (24.3%) | 13,285 (26.1%) | -0.04 |

| N antidiabetic drugs at index date | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| mean (sd) | 1.76 (0.70) | 1.75 (0.68) | 1.77 (0.72) | 1.77 (0.70) | 1.73 (0.70) | 1.73 (0.67) | 1.74 (0.70) | 1.74 (0.68) | 0.00 |
| median [IQR] | 2.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 2.00 (0.70) | 2.00 (0.68) | 0.00 |
| number of different/distinct medication | | | | | | | , , | , , | |
| prescriptions | | | | | | | | | |
| mean (sd) | 11.06 (5.30) | 11.07 (5.36) | 10.74 (5.13) | 10.66 (5.07) | 11.45 (5.09) | 11.45 (5.01) | 11.26 (5.13) | 11.25 (5.08) | 0.00 |
| median [IQR] | 10.00 [7.00, 14.00] | 10.00 [7.00, 14.00] | 10.00 [7.00, 13.00] | 10.00 [7.00, 14.00] | 11.00 [8.00, 14.00] | 11.00 [8.00, 14.00] | 10.65 (5.13) | 10.65 (5.08) | 0.00 |
| Number of Hospitalizations | | | | | , | | , | , | |
| mean (sd) | 0.13 (0.41) | 0.13 (0.41) | 0.12 (0.38) | 0.12 (0.39) | 0.17 (0.48) | 0.16 (0.48) | 0.15 (0.45) | 0.15 (0.45) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | [00.0,00.0] | 0.00 [0.00, 0.00] | 0.00 (0.45) | 0.00 (0.45) | 0.00 |
| Number of hospital days | (,) | (,, | (,, | (,, | (,) | (,, | () | , | |
| mean (sd) | 0.65 (2.51) | 0.67 (2.66) | 0.63 (2.74) | 0.66 (2.86) | 1.03 (3.87) | 1.02 (3.97) | 0.90 (3.49) | 0.90 (3.60) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (3.49) | 0.00 (3.60) | 0.00 |
| Number of Emergency Department (ED) visits | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.00, 0.00) | 0.00 (5.15) | 0.00 (5.00) | 0.00 |
| mean (sd) | 0.50 (1.18) | 0.49 (1.40) | 0.19 (1.07) | 0.19 (1.26) | 0.63 (1.43) | 0.63 (1.44) | 0.53 (1.33) | 0.53 (1.40) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (1.33) | 0.00 (1.40) | 0.00 |
| Number of Office visits | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (1.55) | 0.00 (1.40) | 0.00 |
| mean (sd) | 5.54 (4.50) | 5.53 (4.36) | 5.93 (5.53) | 5.86 (4.31) | 6.33 (4.88) | 6.36 (4.75) | 6.12 (4.93) | 6.13 (4.61) | 0.00 |
| median [IQR] | 4.00 [2.00, 7.00] | 5.00 [3.00, 7.00] | 5.00 [3.00, 8.00] | 5.00 [3.00, 8.00] | 5.00 [3.00, 9.00] | 5.00 [3.00, 9.00] | 4.83 (4.93) | 5.00 (4.61) | -0.04 |
| Number of Endocrinologist visits | 4.00 [2.00, 7.00] | 3.00 [3.00, 7.00] | 3.00 [3.00, 8.00] | 3.00 [3.00, 8.00] | 3.00 [3.00, 3.00] | 3.00 [3.00, 3.00] | 4.83 (4.93) | 3.00 (4.01) | -0.04 |
| mean (sd) | 0.69 (2.65) | 0.80 (2.89) | 0.72 (2.77) | 0.83 (3.11) | 0.94 (3.83) | 0.94 (3.69) | 0.86 (3.48) | 0.90 (3.47) | -0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (3.48) | 0.00 (3.47) | 0.00 |
| Number of internal medicine/family medicine visits | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (3.48) | 0.00 (3.47) | 0.00 |
| mean (sd) | 10.20 (14.44) | 9.35 (14.18) | 7.99 (10.52) | 7.84 (10.00) | 8.97 (12.50) | 8.98 (11.60) | 9.02 (12.55) | 8.85 (11.84) | 0.01 |
| | 6.00 [2.00, 13.00] | 5.00 [1.00, 12.00] | 5.00 [2.00, 10.00] | 5.00 [2.00, 10.00] | 5.00 [2.00, 12.00] | 6.00 [2.00, 12.00] | 5.17 (12.55) | 5.65 (11.84) | -0.04 |
| median [IQR]<br>Number of Cardiologist visits | 0.00 [2.00, 13.00] | 5.00 [1.00, 12.00] | 5.00 [2.00, 10.00] | 3.00 [2.00, 10.00] | 3.00 [2.00, 12.00] | 0.00 [2.00, 12.00] | 3.17 (12.33) | 5.05 (11.04) | -0.04 |
| | 1.05 (4.06) | 1.05 (4.52) | 1 46 (2 50) | 1 47 (2 42) | 2.25 (5.02) | 2.33 (5.16) | 2.04 (4.64) | 2.42 (4.00) | -0.02 |
| mean (sd) | 1.85 (4.06) | 1.95 (4.53) | 1.46 (3.59) | 1.47 (3.43) | 2.25 (5.02) | , , | 2.04 (4.64) | 2.12 (4.80) | 0.02 |
| median [IQR] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 (4.64) | 0.00 (4.80) | 0.00 |
| Number electrocardiograms received | 0.76 (1.40) | 0.76 (4.50) | 0.60 (1.20) | 0.67/1.22\ | 0.06 (4.53) | 0.00 (1.50) | 0.01/1.40 | 0.01 (1.46) | 0.00 |
| mean (sd) | 0.76 (1.49) | 0.76 (1.50) | 0.68 (1.29) | 0.67 (1.22) | 0.86 (1.52) | 0.86 (1.50) | 0.81 (1.48) | 0.81 (1.46) | |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (1.48) | 0.00 (1.46) | 0.00 |
| Number of HbA1c tests ordered | 4 24 (0 05) | 4 20 (0 0 4) | 0.00 (0.05) | 0.00 (0.03) | 4 47 (4 00) | 4 47 (0 04) | 4.25 (4.00) | 4.25 (0.02) | 0.00 |
| mean (sd) | 1.31 (0.95) | 1.30 (0.94) | 0.99 (0.95) | 0.98 (0.93) | 1.47 (1.03) | 1.47 (0.91) | 1.36 (1.00) | 1.36 (0.92) | 0.00 |
| median [IQR] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 (1.00) | 1.00 (0.92) | 0.00 |
| Number of glucose tests ordered | 0.00 (6.63) | 0.02/7.24) | 0.40 (2.42) | 0.40(4.26) | 0.55 (4.53) | 0.57 (4.24) | 0.50 (2.46) | 0.62 (2.27) | 0.04 |
| mean (sd) | 0.80 (6.63) | 0.93 (7.31) | 0.49 (2.13) | 0.49 (1.26) | 0.55 (1.52) | 0.57 (1.31) | 0.58 (3.16) | 0.62 (3.27) | -0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (3.16) | 0.00 (3.27) | 0.00 |
| Number of lipid tests ordered | | | | | | | | | |
| mean (sd) | 1.04 (1.03) | 1.03 (1.00) | 0.85 (1.36) | 0.86 (1.33) | 1.08 (0.95) | 1.08 (0.89) | 1.03 (1.05) | 1.03 (1.00) | 0.00 |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 1.00 (1.05) | 1.00 (1.00) | 0.00 |
| Number of creatinine tests ordered | | | | | | | | | |
| mean (sd) | 0.06 (0.33) | 0.07 (0.47) | 0.07 (0.44) | 0.07 (0.58) | 0.10 (0.47) | 0.09 (0.40) | 0.09 (0.44) | 0.08 (0.45) | 0.02 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.44) | 0.00 (0.45) | 0.00 |
| Number of BUN tests ordered | | | | | | | | | |
| mean (sd) | 0.04 (0.27) | 0.04 (0.38) | 0.04 (0.38) | 0.05 (0.58) | 0.06 (0.39) | 0.06 (0.32) | 0.05 (0.37) | 0.05 (0.39) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.37) | 0.00 (0.39) | 0.00 |
| Number of tests for microalbuminuria | | | | | | | | | |
| mean (sd) | 0.89 (1.29) | 0.87 (1.32) | 0.58 (1.12) | 0.57 (1.04) | 0.56 (0.85) | 0.56 (0.84) | 0.62 (0.99) | 0.62 (0.98) | 0.00 |
| median [IQR] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (0.99) | 0.00 (0.98) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd | | | | | | | | | |
| digit level | 7.42 (0.00) | 7.25 (0.77) | 2.02 /5.22 | 2.05 (5.55) | 7.70 (0) | 7.00 (0.00) | 6 07 (0 75) | C 00 (0 75) | 0.55 |
| mean (sd) | 7.43 (8.69) | 7.35 (8.77) | 2.83 (5.33) | 2.85 (5.39) | 7.78 (9.41) | 7.69 (9.43) | 6.87 (8.72) | 6.80 (8.75) | 0.01 |
| median [IQR] | 5.00 [0.00, 11.00] | 5.00 [0.00, 11.00] | 0.00 [0.00, 4.00] | 0.00 [0.00, 4.00] | 5.00 [0.00, 12.00] | 5.00 [0.00, 12.00] | 4.14 (8.72) | 4.14 (8.75) | 0.00 |
| Use of thiazide; n (%) | 1,042 (11.7%) | 1,075 (12.1%) | 1,002 (11.5%) | 1,005 (11.5%) | 4,626 (13.9%) | 4,591 (13.8%) | 6,670 (13.1%) | 6,671 (13.1%) | 0.00 |
| Use of beta blockers; n (%) | 4,537 (51.1%) | 4,527 (51.0%) | 4,436 (50.9%) | 4,413 (50.6%) | 19,108 (57.3%) | 19,031 (57.1%) | 28,081 (55.2%) | 27,971 (54.9%) | 0.01 |
| Use of calcium channel blockers; n (%) | 2,943 (33.1%) | 3,037 (34.2%) | 2,769 (31.8%) | 2,780 (31.9%) | 13,117 (39.4%) | 12,995 (39.0%) | 18,829 (37.0%) | 18,812 (36.9%) | 0.00 |
| 222 2. Garciani Granici Diotecio, ii (70) | 2,545 (55.170) | 3,037 (37.270) | 2,, 33 (31.070) | 2,730 (31.370) | 13,117 (33.770) | 12,555 (55.670) | 10,023 (37.070) | 10,011 (30.370) | 5.50 |